## **CCTG 595**

# A Multicenter, Randomized Study of *T*ext messaging to improve *A*dherence to *P*rEP *In R*isky MSM (TAPIR)



A Multicenter Trial of the California Collaborative Treatment Group (CCTG)

Sponsored by:

The California HIV/AIDS Research Program (CHRP)

Protocol Co-chairs: Sheldon Morris, MD, MPH
David J. Moore, PhD

**Protocol Version 5.0** 

Original: November 1<sup>st</sup>, 2012 Amended: August 10<sup>th</sup>, 2015

# **TABLE OF CONTENTS**

| PROTOCOL TEAM ROSTER | pg 4 |
|----------------------------------------------------------------|-------|
| Study Co-Chairs | pg 4 |
| Study Vice-Chairs | _ |
| Co-Investigators | pg 4 |
| Clinical Trials Specialist | |
| Statistician | pg 6 |
| Study Monitor and Data Unit | pg 6 |
| Lab Technician | pg 7 |
| LIST OF ABBREVIATIONS | |
| SCHEMA | pg 9 |
| Design | pg 9 |
| Duration | pg 9 |
| Sample Size | pg 9 |
| Study Population | pg 9 |
| Stratification | pg 9 |
| Intervention | pg 10 |
| Regimen | pg 10 |
| Outcomes | |
| 1.0 STUDY OBJECTIVES AND HYPOTHESES | pg 11 |
| 1.1 Study Primary Objectives | pg 11 |
| 1.2 Study Secondary Objectives | pg 11 |
| 1.3 Exploratory Objectives | pg 12 |
| 2.0 INTRODUCTION | 17 |
| 2.1 Study Background | pg 11 |
| 2.2 Study Rationale | pg 14 |
| 3.0 STUDY DESIGN | pg 15 |
| 3.1 Study Design | pg 15 |
| 3.2 iTAB Adherence Intervention | pg 14 |
| 3.3 Qualitative Plasma Concentrations as an Adherence Marker | pg 16 |
| 4.0 SELECTION AND ENROLLMENT OF SUBJECTS | pg 17 |
| 4.1 Study Inclusion Criteria | pg 17 |
| 4.2 Study Exclusion Criteria | pg 17 |
| 4.3 Enrollment Procedures | 4.0 |
| 5.0 STUDY TREATMENT | |
| 5.1 Regimens, Administration, and Duration | pg 18 |
| 5.2 Study Product Formulation | pg 20 |
| 5.3 Pharmacy: Product Supply, Distribution, and Accountability | pg 20 |
| 5.4 Concomitant Medications | pg 20 |
| 5.5 Adherence Assessment | pg 20 |
| 6.0 CLINICAL AND LABORATORY EVALUATION | pg 22 |
| 6.1 Table of Schedule of Events | pg 22 |

| 6.2 Definitions for Schedule of Events and Timing of Evaluations | _ pg 23 |
|---|---|
| 6.3 Special Instructions and Definitions of Evaluations | _ pg 26 |
| 7.0 TOXICITY MANAGEMENT | _ pg 30 |
| 7.1 General Management for Grade 1-4 Events | _ pg 30 |
| 7.2 Management for Specific Adverse Events | _ pg 31 |
| 8.0 CRITERIA FOR EARLY DISCONTINUATION | |
| 8.1 Criteria for Discontinuation from Study | _ pg 33 |
| 9.0 STATISTICAL CONSIDERATIONS | _ pg 34 |
| 9.1 Primary Endpoints | |
| 9.2 Secondary Endpoints | _pg 34 |
| 9.3 Randomization and Stratification | _ pg 35 |
| 9.4 Study Power and Sample Size Justification | _ pg 35 |
| 9.5 Monitoring | _ pg 35 |
| 9.6 Analyses | |
| 10.0 PHARMACOLOGY PLAN | _ pg 38 |
| 10.1 Sample Assay Methods | _ pg 38 |
| 11.0 DATA COLLECTION AND MONITORING AND ADVERSE EVENT REPORTING $\_$ | _pg 38 |
| 11.1 Records to be Kept | _ pg 38 |
| 11.2 Role of Data Management | _ pg 38 |
| 11.3 Clinical Site Monitoring and Record Availability | _ pg 38 |
| 11.4 Serious Adverse Experiences (SAE) Reporting | |
| 12.0 HUMAN SUBJECTS | _ pg 39 |
| 12.1 Institutional Review Board (IRB) and Informed Consent | _ pg 39 |
| 12.2 Subject Confidentiality | _ pg 39 |
| 12.3 Study Discontinuation | _ pg 39 |
| 13.0 PUBLICATION AND RESEARCH FINDINGS | _ pg 40 |
| 14.0 BIOHAZARD CONTAINMENT | _ pg 40 |
| 15.0 REFERENCES | _ pg 40 |
| 16.0 APPENDICES_ | _ pg 42 |
| APPENDIX I: SAMPLE OF INFORMED CONSENT | _ pg 42 |
| APPENDIX II: QUESTIONNAIRES | _ pg 50 |
| APPENDIX III: VITAMIN D SUB-STUDY PROTOCOL | _ pg 86 |
| APPENDIX IV: VITAMIN D SUB-STUDY SAMPLE OF INFORMED CONSENT | _ pg 99 |
| APPENDIX V: MULTIVITAMIN SUPPLEMENT COMPARISONS | pg 104 |
| APPENDIX VI: DIFTARY CALCILIM AND VITAMIN D INTAKE CALCILIATOR | ng 106 |

#### **PROTOCOL TEAM ROSTER**

#### **Study Co-Chairs**

Sheldon Morris, MD, MPH David J. Moore, PhD

Associate Professor of Medicine Associate Professor of Psychiatry University of California, San Diego University of California, San Diego

Antiviral Research Center HIV Neurobehavioral Research Programs

220 Dickinson St., Suite A220 Dickinson St., Suite BSan Diego, CA 92103San Diego, CA 92103Phone619.543.8080Phone619.543.5093

Fax 619.543.5066 Fax 619.543.1235 E-mail shmorris@ucsd.edu E-mail djmoore@ucsd.edu

## **Co-Investigators**

Michael Dubé, M.D. Eric Daar, M.D.

Professor of Medicine Chief, Division of HIV Medicine
Keck School of Medicine Harbor-UCLA Medical Center

University of Southern California Professor of Medicine

1300 N. Mission Road, Room 349 David Geffen School of Medicine
Los Angeles, CA 90033 University of California, Los Angeles

 Phone
 323.343.8288
 1124 W. Carson St., N-24

 Fax
 323.226.2083
 Torrance, CA 90502

 E-mail
 mdube@usc.edu
 Phone
 310.222.2467

 Fax
 310.533.0447

E-mail edaar@labiomed.org

Jill Blumenthal, MD Katya Calvo, MD

HIV Research Fellow Health Sciences Assistant Professor
University of California, San Diego David Geffen School of Medicine at UCLA

Antiviral Research Center Harbor-UCLA Medical Center

220 Dickinson St., Suite A 1124 West Carson Street
San Diego, CA 92103 N-24

Phone 619.543.8080 Torrance, CA 90502 Fax 619.543.5094 Phone: 310.222.2159

E-mail jblumenthal@ad.ucsd.edu Fax: 310.533.0447

E-mail krcalvo@labiomed.org

Martin Sattah, MD Deborah Collins, PA-C

Clinical Assistant Professor Preventative Health Clinical Services Director
LAC/USC Medical Center Long Beach Department of Health and Human

Dept. of Internal Medicine/ Division of Services

Infectious Diseases 2525 Grand Avenue, Suite 106

1300 North Mission Road Long Beach, CA 90815 Los Angeles, CA 90033 Phone: 562.570.4379 Phone: 323.343.8255 Fax:

Fax: 323.226.3571 E-mail deborah.collins@longbeach.gov

E-mail sattah@usc.edu

# **Clinical Trials Specialist**

Eric E. Ellorin
Staff Research Associate
University of California, San Diego
Antiviral Research Center
220 Dickinson St., Suite A
San Diego, CA 92103

Phone 619.543.8080 Fax 619.543.5072

E-mail eellorin@ucsd.edu

# Statistician

E-mail

Sonia Jain, PhD
Associate Professor, Division of Biostatistics and Bioinformatics
Director, CCTG Biostatistics Core
Co-Director, Biostatistics Research Center (BRC)
University of California, San Diego
9500 Gilman Dr., MC 0717
La Jolla, CA 92093-0717
Phone 858.822.2388

# **Study Monitor and Data Unit**

sojain@ucsd.edu

Edward Seefried, RN
Medical Monitor, Study Coordinator, CCTG Data Unit
University of California, San Diego
Antiviral Research Center
220 Dickinson St., Suite A
San Diego, CA 92103
Phone 619.543.8080
Fax 619.543.5072

E-mail eseefried@ucsd.edu

#### **Lab Technician**

DeeDee Pacheco
Phlebotomist and Lab Manager
University of California, San Diego
Antiviral Research Center

220 Dickinson St., Suite A San Diego, CA 92103

Phone 619.543.8080 Fax 619.543.5067

E-mail dmpacheco@ucsd.edu

#### LIST OF ABBREVIATIONS

AE Adverse Event

ALERT Active Linkage, Engagement, and Retention to Treatment

ARV Antiretroviral Therapy

CCTG California Collaborative Treatment Group

CD4 CD4 Lymphocytes CRF Case Report Form

CT Chlamydia

DSMB Data Safety and Monitoring Board

GC Gonorrhea

HAART Highly Active Antiretroviral Therapy
HIV-1 Human Immunodeficiency Virus – 1

iTAB Individualized Texting for Adherence Building

**Modified Intention to Treat** mITT MSM Men who have Sex with Men NAAT **Nucleic Acid Amplification Test** PLWH Persons Living With HIV/AIDS PrEP Pre-Exposure Prophylaxis RPR Rapid Plasmin Reagin Statistical Analysis Plan SAP Serious Adverse Event SAE

SoC Standard of Care

STI Sexually Transmitted Infection

TPPA Treponema Pallidum Particle Agglutination Assay

VAS Visual Analog Scale

VDRL Venereal Disease Research Laboratory

#### **SCHEMA**

Design: CCTG 595 is a controlled, open-label, two-arm, randomized (1:1) clinical

demonstration project to determine if the use of a text-message based adherence intervention (iTAB) improves retention and adherence to PrEP

compared to standard of care (SoC) PrEP delivery.

Duration: Each subject will be followed for up to 48 weeks after enrollment of the

last subject to a maximum of 96 weeks. The primary endpoint will be

measured at 48 weeks.

<u>Sample Size:</u> A total of 400 subjects will be randomized, 200 per arm.

Study Population: Eligible subjects will include HIV-uninfected men who have sex with men

(MSM) and male to female (M to F) transgender individuals who have sex with men at least 18 years of age and who have a recent history of high-

risk transmission behavior.



Stratification: The randomization will be stratified based on clinic site.

Intervention:

All subjects will start PrEP with TDF + FTC fixed dose combination given once daily. Subjects will be randomized (1:1) to either the iTAB text messaging adherence reminder intervention with SoC or the SoC alone arm. Subjects placed into the iTAB intervention arm will receive a personalized, automated texting system to maintain adherence and retention. Both groups will receive access to PrEP in accordance with standardized comprehensive methods of prescribing, risk reduction counseling, adherence counseling, and clinical assessments that include safety monitoring, as well as HIV and STD screening.

Regimen:

TDF 300 mg + FTC 200 mg fixed dose combination will be given orally once daily starting at the baseline visit (month 0) and continued throughout the study.

Outcomes:

The CCTG 595 primary outcome is defined as a composite endpoint of remaining on PrEP and having adherence > 90% over 48 weeks of follow-up. The adherence endpoint will be derived from the 4 day ACTG adherence assessment from each of the visits from week 4, 12, 24, 36, and 48. 'Adherent' will be defined as self-reported TDF/ FTC adherence of 90% or greater (at least 18 of 20 days). If a subject misses an adherence assessment within the window of a scheduled visit or discontinues study prior to week 48, then the missed visits will be counted no adherence for the time of that visit. All randomized subjects that were dispensed PrEP at baseline will be included in the modified intent-to-treat analysis.

#### 1.0 STUDY OBJECTIVES AND HYPOTHESES

## 1.1 Study Primary Objective:

CCTG 595 will compare adherence to fixed dose TDF/FTC, between subjects randomized to receive SoC plus text message reminders versus SoC, when used for pre-exposure prophylaxis among MSM at high risk for HIV acquisition.

# 1.1.1 Hypothesis I

MSM and transgender M to F having sex with men with high risk of HIV acquisition randomized to the iTAB intervention will have higher self-reported adherence to TDF/FTC for PrEP over 48 weeks ('adherent' defined with a composite endpoint of continued retention on PrEP and > 90% adherence to TDF/FTC at 48 weeks) compared to MSM that have comprehensive SoC alone.

# 1.1.2 Hypothesis II

MSM and transgender M to F having sex with men with high risk of HIV acquisition randomized to the iTAB intervention will have higher adherence to TDF/FTC for PrEP over 48 weeks, as measured by having five of five detectable qualitative FTC plasma concentrations at scheduled visits compared to MSM that have comprehensive standard of care alone.

# 1.2 Study Secondary Objectives:

- 1.2.1 To compare adherence to TDF/FTC in the iTAB versus SoC in the subjects that remain on PrEP (at 48 weeks and up to 96 weeks of follow up) by the continuous measure of percent days adherent by the cumulative 4 day ACTG and the visual analog scale (VAS) recall in an 'as treated' analysis.
- 1.2.2 To compare adherence to TDF/FTC in the iTab versus SoC groups for the duration of the study (up to 96 weeks). Adherence will be compared using the same outcomes as hypothesis I (self-reported to be on drug and 90% adherent) and II (100% detectable FTC at each scheduled visit) as modified intent to treat analysis.
- 1.2.3 To determine factors associated with poor adherence/lost to PrEP in study participants (outcomes of < 90% adherent on drug at 48 weeks by ACTG 4 day recall or discontinuation of drug). Factors associated with poor adherence to TDF/FTC will include demographics, ongoing

substance use, untreated mental illness, socioeconomic status, low health/HIV and system literacy, fear of disclosure and non-English language.

- 1.2.4 To determine the factors associated with discontinuation of TDF/FTC at any time point including change in perceived and actual risk of HIV acquisition, demographics, ongoing substance use, untreated mental illness, socioeconomic status, low health/HIV and system literacy, fear of disclosure and non-English language.
- 1.2.5 To determine the rate of HIV seroconversion in PrEP users and compare the iTAB to SOC arms for number of new infections as a proportion at 48 weeks and end of study.
- 1.2.6 To measure acquisition of other sexually transmitted infections (STIs); the proportion of subjects with any new STI at any site will be compared between the iTAB to SOC arms at 48 weeks and through the end of the study.
- 1.2.7 To evaluate changes in risk behavior after initiation of PrEP (risk compensation) comparing baseline to subsequent visits for number of HIV positive/unknown status partners and any unprotected anal intercourse with an HIV positive/ unknown status partner.
- 1.2.8 To evaluate the safety and tolerability of daily TDF/FTC given for PrEP including discontinuation for any adverse event, serious adverse events and adverse events (grade 2 or higher).

# 1.3 Exploratory Objectives:

1.3.1 To describe changes over time of self-reported adherence in real time by texting.

# 2.0 INTRODUCTION

## 2.1 Study Background

Widespread deployment of PrEP will require operational research to study how best to integrate services into clinical care settings and to target them to various at-risk populations [1-3]. Randomized controlled trials of PrEP have shown a statistically significant reduction in acquisition of HIV among at-risk individuals in a research setting but provide little insight into how it could be practically applied. Implementing PrEP strategies will necessitate: 1) creation of an organizational framework to deliver services; 2) delineation of patient populations where PrEP should be targeted and would be most effective; 3) identification and removal of structural barriers to PrEP delivery (such as co-ordination of services between organizations, and establishing infrastructure to deliver services) and 4) establishing related services such as patient education, drug adherence counseling and reminder systems for medication adherence.

Sustainable programs for PrEP delivery may utilize either new clinical care systems or existing care providers such as treatment clinics, community care clinics, public health facilities or HIV testing sites. Adding PrEP to clinical HIV care may be the most efficient method considering the requirements for PrEP: 1) prescription of antiretroviral agents; 2) monitoring for adverse events and HIV acquisition; 3) interventions for risk reduction and drug adherence and 4) provision of comprehensive care for sexually transmitted infections, mental health and substance use [4].

This study will evaluate the integration of PrEP into clinical practice by identifying at-risk individuals at HIV testing sites, linking them to treatment clinics, and initiating and maintaining PrEP. This model for PrEP utilizes providers that are experienced with ARV drugs, adherence counseling, and care of high-risk patients. The CCTG clinical sites have successfully integrated other prevention interventions into their care delivery for previous studies and serve populations for which PrEP will be most needed [5].

HIV care clinics in California are familiar with the target population for PREP because the patient population is largely MSM who continue HIV transmission-associated behaviors. Epidemiological studies have found that MSM at the highest risk for acquiring HIV are those who have HIV positive partners, a sexually transmitted disease, multiple sexual partners, use methamphetamine, and attend specific venues such as bath houses and internet "hook-up" sites [6-8]. In the iPREX study, HIV acquisition among a diverse population of high-risk MSM was reduced by 44%, leading to current CDC guidance on PrEP which targets MSM who have "sustained" risk of HIV acquisition, normal renal function and negative HIV by EIA and no symptoms of acute HIV infection [9, 10].

Implementing PrEP for MSM will require education of the high risk groups since initial studies found only 47% had some knowledge of PrEP and only 4% were using PrEP [11]. Uptake

of PrEP is anticipated to be good in some high risk groups. Partners of HIV-infected individuals may be most motivated. In one study 80% of discordant heterosexual couples accepted PrEP during reproductive planning [12]. A similar study found that 74% of MSM, who received PrEP education, would consider taking it if available [13]. Therefore, increasing the community awareness and education of PrEP should increase interest, especially if barriers to referral for PrEP are minimized, and counseling and education are provided.

Once linked and engaged in PrEP, candidates will require a systematic approach to maintain follow-up and adherence to medication. The literature generally shows that adherence levels of 95-100% are needed to ensure optimal treatment effectiveness for the treatment of HIV [14]. Similarly, PrEP efficacy in iPREX was shown to be diminished with reductions in adherence [9]. In a nested case-control study, TDF and FTC drug levels were detectable in only 9% of individuals that seroconverted to HIV compared to 51% of the controls that did not acquire HIV [9]. Adherence is commonly defined as ≥ 90% of prescribed doses taken, but no single definition has achieved consensus across the literature and various definitions have be associated with worsened HIV disease outcome[15]. In iPREX, 90% adherence by self-report at 49% of visits was found to increase efficacy from 44% to 75% in HIV acquisition reduction. Barriers to adherence have been widely studied in HIV-infected individuals and summarized by Mills et al. [16]. From studies in developed countries the factors associated with adherence can be summarized as: 1) individual psycho-social factors (sense of stigma, feeling hopeless, having addiction diagnosis, mistrust of medical system and medications, problems with memory, poor understanding, low self-worth, finances, homelessness); 2) beliefs on medication (real or perceived adverse events, complicated regimens, uncertainly of effect); 3) daily schedules (irregular routines, coordinating adherence with social supports); and 4) issues of social cohesion (lack of trust in providers, social isolation, negative publicity in community, negative feedback from social network) [16]. Facilitators of adherence relevant to PrEP include 1) increasing self-worth and prioritizing health over addiction; 2) having 'faith' in the treatment and understanding adherence importance; 3) having daily routines and using reminder systems and 4) trusting providers, disclosing to social supports and feeling supported by social network. Maximizing adherence for PrEP will therefore require developing good relationships and providing ongoing heath education, counseling and reinforcement on HIV and PrEP. A promising method of reinforcing ART adherence is text messaging. In one study in a group of poorly adherent HIV-infected individuals, an increase in adherence from 42% to over 70% was observed in those receiving texting [17]. In this proposal, a comprehensive approach to routine clinical care will be expanded to provide the necessary elements for safely implementing PrEP. HIV prevention and PrEP education will figure prominently in the interactions with community and participants including reinforcement of the adherence message coupled with risk reduction counseling at each clinic visit. In the randomized component of the study, the ALERT worker will use text reminders as a strategy for enhancing PrEP adherence.

#### 2.2 Study Rationale

TDF/FTC has been approved by the FDA as an agent for PrEP. As noted previously, there is no research on how PrEP will be delivered in the community setting. CCTG 595, will implement PrEP at three sites (UCSD, UCLA/Long Beach Health Department, USC) to explore the operationalization of PrEP by the community providers of HIV testing and HIV care. Critical to the implementation of PrEP will be to maintain adherence to drug. CCTG 595 will perform a randomized controlled study of the iTAB texting intervention for TDF/FTC adherence for PrEP. This intervention is meant to be a simple automated method to reinforce adherence.

#### 3.0 STUDY DESIGN

# 3.1 Study Design

CCTG 595 is a comparative, interventional study that uses text messaging to improve adherence of PrEP in MSM and transgender that are at high risk of acquiring HIV. We will conduct an open-label, randomized, controlled clinical trial to evaluate an intervention strategy that uses a developed texting adherence method, the iTAB system, to improve adherence and retention compared to standard of care which will not have iTAB (see study schema). The RCT will occur in the context of implementation of PrEP at three large, diverse, urban HIV care clinics in the CCTG network at UCLA-Harbor, USC and UCSD and a fourth site at the Long Beach Public Health Department. These sites are collaborating with local testing sites to provide an integrated program that identifies individuals at highest risk for HIV acquisition and link them into preventive care that will provide the assessment, dispensing and monitoring of PrEP. A uniform system of HIV testing, risk assessment, health education and behavioral/adherence counseling will be developed for use at consortium sites.

Study enrollment criteria is based on the CDC guidance for PrEP use among MSM and transgender with ongoing risk for HIV infection. All subjects will be confirmed to be uninfected with no contraindication to TDF/FTC. Subjects will be randomized at baseline to iTAB versus SoC. Randomization will be stratified by CCTG site. Study visits will include screening, baseline, week 4 and 12 initial visits and then visits every 12 weeks. Visits for iTAB and SoC arms will both include routine HIV testing and counseling, STI testing, adherence counseling, and medical monitoring. Each visit will include a computer-assisted survey for self-reported adherence assessment and risk behaviors. Drug level monitoring will be performed for FTC qualitative levels in retrospect on banked samples and additional banked specimens will be available for future use and TDF measurement. Adherence by self-reported measures and FTC levels will be used for the main and secondary analyses of the study. Additional outcomes for the study will include changes in risk behavior and determinants of PrEP adherence. Outcomes will be assessed at 48 weeks and for the cumulative follow up of all participants. The study will continue for 48 weeks after randomization of the last participant (up to 96 weeks for any subject).

In order to have adequate representation of African Americans in the study population,

enrollment of non-African Americans will be capped at 85% of 400 subjects (340) to achieve at least 15% African Americans. If 340 non-African American subjects are enrolled, then enrollment for this subgroup will stop and the study will remain open only for African Americans.

## 3.2 iTAB Adherence Intervention

This proposal will perform a study of potential methods to improve adherence and retention by evaluating standard procedures versus the use of the iTAB platform. All subjects will receive SoC that will include health education, clinical assessments, laboratory safety monitoring, STI and HIV screening, HIV risk reduction counseling, assessment of psycho-social barriers, adherence counseling, and completion of a computer based survey.

Subjects will be randomized to 1) SoC clinic visits as outlined in section 6.0 and 2) SoC visits plus support using text messaging through the iTAB system. Subjects assigned to the iTAB intervention will have visits with the study coordinator to introduce the iTAB texting system, discuss contact information to assist in recovering the subject if they miss appointments and provide training on iTAB framework for texting supportive reminder messages and tracking adherence. The study will provide subject reimbursement to pay for unlimited text message use and in cases where a subject does not have a phone, the appropriate cell phone will be provided.

Daily dosing reminders will be sent for the first 6 weeks and then continue with reminders for the duration of the study. Both reminder timing and message content can be individualized. The study coordinator will work with the participant to select and refine 10 personal reminders from a list of pre-determined reminders that cover various themes shown to be effective in improving adherence (e.g., social support, loss frame, health gain, etc.) as developed through focus groups and targeted group feedback. These messages can be modified and the patient can choose to create their own reminders if they prefer. The coordinator will work with each participant individually to assure that adherence reminders are sent at times consistent with when the patient typically takes his medication. These reminder times can vary for different days of the week to accommodate for changes in schedule (e.g., 8 M-F, and 10 AM on Sat/Sun). Once the time is identified, the text reminder system is automated. Patients will confirm medication taking via text responses to the personalized reminders. If a participant does not respond on three consecutive occasions, a high alert message (chosen by the participant) will be sent. If the subject does not respond to this message, the study coordinator would initiate phone calls to contact the subject and explore barriers. The coordinator will continue to call the participant every 4 days until the participant re-engages with the iTAB system.

## 3.3 FTC Qualitative Plasma Concentration as an Adherence Marker

Adherence to prescribed treatment can be difficult to assess. One objective way to measure recent adherence is to measure plasma drug concentrations. FTC concentrations in plasma remain detectable throughout the dosing interval. Specifically, trough concentrations of FTC are approximately 60 - 70 ng/mL, and range from 10 - 300 ng/mL between subjects [23, 24]. Peak concentrations are approximately 1300 - 1800 ng/mL, and range from 600 to 2500 ng/mL. While many factors contribute to variability in plasma concentrations, such as drug-drug interactions and genetic differences in absorption and excretion, completely undetectable plasma concentrations of FTC are physiologically implausible for patients who are adherent with their regimen. Even with the sources of variability noted above, undetectable concentrations (< 1 ng/mL) would be 60 to over 1000 times less than the expected concentration depending on the time post-dose, and can be justifiably assumed to represent missed doses rather than pharmacokinetic variability. We plan for 400 subjects and in total will have 3467 levels (an average of 8.6 per person). Samples will be stored at each study visit (weeks 4, 12 and every 12 weeks thereafter).

#### 4.0 SELECTION AND ENROLLMENT OF SUBJECTS

## 4.1 Main Study Inclusion Criteria

- 4.1.1 Man or transgender M to F who has sex with men.
- 4.1.2 Age 18 years or older.
- 4.1.3 Subjects must have substantial ongoing risk of acquisition of HIV as evident by one or more of the following:
  - Has at least one HIV infected sexual partner for ≥4 weeks.
  - No condom use during anal intercourse with ≥3 male sex partners who are HIV-positive or of unknown HIV status during the last 3 months
  - No condom use during anal sex with ≥1 male partner and STI diagnosis during the last 3 months
- 4.1.4 Negative for HIV infection by rapid HIV test and confirmed negative by NAT or other sensitive method such as antibody- antigen test.
- 4.1.5 Acceptable laboratory values in the past 30 days:
  - Calculated creatinine clearance of at least 60 mL/min by the Cockcroft-Gault formula (eCcr (male) in mL/min = [(140 – age in years) x (lean body weight in kg)] / (72 x serum creatinine in mg/dL)
  - Alanine aminotransferase (ALT) and/ or aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN)</li>

- Hemoglobin > 9 g/dL
- Absolute neutrophil count > 750/ mm<sup>3</sup>
- Platelets > 75,000/ mm<sup>3</sup>

# 4.2 Main Study Exclusion Criteria

- 4.2.1 Unable to give informed consent.
- 4.2.2 Active hepatitis B (positive hepatitis B surface antigen (HBSAg) or HBSAg negative/ HB core antibody positive/ HBV PCR positive)
- 4.2.3 Has substantial medical condition, that in the opinion of the investigator would preclude participation, as defined by
  - cardiovascular condition that may lead to an increased risk of complication if placed on study drugs.
  - gastrointestinal condition that would impair absorption of study drugs.
  - neurological or psychiatric condition that would significantly impair the ability to adhere to PrEP.
  - calculated GFR < 60 mL/min</li>
  - alcohol or drug abuse or dependence that would significantly impair the ability to adhere to PrEP (only for those with severe impairment).
  - Other medical condition that would unacceptably increase the risk of harm from study drug or significantly impair the ability to adhere to PrEP.
- 4.2.4 Suspected sensitivity or allergy to the study drug or any of its components.
- 4.2.5 Currently using an essential product or medication that interacts with the study drug such as the following:
  - ART (including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents)
  - Agents with known nephrotoxic potential:
    - o aminoglycoside antibiotics (including gentamicin)
    - o IV amphotericin B
    - o cidofovir
    - cisplatin
    - foscarnet
    - IV pentamidine
    - o IV vancomycin

- o oral or IV gancyclovir
- o other agents with significant nephrotoxic potential
- Drugs that slow renal excretion
  - o Probenecid
- Immune system modulators
  - Systemic chemotherapeutic agents (i.e. cancer treatment medications)
  - Ongoing systemic corticosteroids (with the exception of short courses of tapering steroid doses for asthma or other selflimited condition).
  - o Interleukin-2 (IL-2)
  - Interferon (alpha, beta, or gamma)
- Other agent known to have a significant interaction with TDF or FTC
- 4.2.6 Proteinuria 2+ or greater by urine dipstick
- 4.2.7 Signs or symptoms suggestive of acute HIV infection
- 4.2.8 Any other reason or condition that in the opinion of the investigator would interfere with participation, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

# 4.3 Enrollment Procedures

- 4.3.1 Prior to implementation of this protocol, sites must have the protocol and consent form approved by their local institution review board (IRB). Sites must be registered with and approved by the CCTG Data Center. Site registration must occur before any subjects can be enrolled in this study.
- 4.3.2 Once a candidate for study entry has been identified, details will be carefully discussed with the subject. The subject will be asked to read and sign the consent form that was approved by both the local IRB and the CCTG Data Center.
- 4.3.3 A patient identification number (PID) will be assigned to each patient screened for the study. PIDs will include site code and be formatted to be compatible with the BIT data core. PIDs will not be reassigned even if the subject fails to enter the study. The PID must be included on every CRF and subject specimen during the study. Each site must maintain a master list of PIDs in a central location. The patient registration and inclusion/exclusion CRF must be completed on the online system.

#### 5.0 STUDY TREATMENT

# 5.1 Regimens, Administration, and Duration

## 5.1.1 Regimens

Subjects will be randomized 1:1 to one of the two treatment arms:

ARM A: FTC/TDF 200/300 mg fixed dose combination once daily + iTAB ARM B: FTC/TDF 200/300 mg fixed dose combination once daily

 Use of the FTC/TDF fixed dose combination is not allowed if the CrCl is <50 mL/min, which should be confirmed within 7 days. TDF/ FTC should be discontinued if confirmed.

# 5.1.2 Administering and Dispensing

Emtricitabine/tenofovir disoproxil fumarate fixed-dose combination containing 200 mg of emtricitabine and 300 mg tenofovir disoproxil fumarate will be administered orally as one tablet once daily with or without food.

Enough study product should be dispensed to last until the subject's next scheduled visit.

#### 5.1.3 Duration

Subjects will participate in this study until 48 weeks beyond the enrollment of the last subject with a maximum duration of 96 weeks for any subject. Subjects may receive study treatment until their last study visit.

Subjects will receive study treatment for the duration of the study unless they meet criteria for discontinuation.

## 5.2 Study Product Formulation

Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF, Truvada®): 200 mg/300 mg coformulated tablet. Store at 25°C (77°F); excursions permitted to 15°-30°C (59°-86°F) [see USP Controlled Room Temperature].

# 5.3 Pharmacy: Product Supply, Distribution, and Accountability

# 5.3.1 Study Product Supply/Distribution

Emtricitabine/tenofovir disoproxil fumarate will be supplied by Gilead Sciences through the UCSD/AVRC Research Pharmacy and distributed to all sites.

The site pharmacist can obtain study product for this protocol by following the instructions in the CCTG-595 Pharmacy Manual.

# 5.3.2 Study Product Accountability

The site pharmacist is required to maintain complete records of all study product received from the UCSD /AVRC Research Pharmacy. All unused study product must be returned to the sponsor (or as otherwise directed by the sponsor) after the study is completed or terminated. The procedures to be followed are provided in the CCTG-595 Pharmacy Manual.

## **5.4 Concomitant Medications**

Whenever a concomitant medication or study agent is initiated or a dose changed, site investigators must review the concomitant medications and study agent's most recent package inserts, Investigator's Brochures to obtain the most current information on drug interactions, contraindications, and precautions.

5.4.1 Prohibited Medications (Refer to Section 4.2 for addition information on prohibited medications).

All the contract to and also are

| 5.4.1.1 | All investigational drugs |
|---|---|
| 5.4.1.2 | All HIV vaccines |
| 5.4.1.3 | Any immunomodulators |
| 5.4.1.4 | Systemic cytotoxic chemotherapy |
| 5.4.1.5 | All other antiretroviral medications (excluding FTC/TDF given as PEP or PrEP) |
| 5.4.1.6 | Drugs with known nephrotoxicity |

Subjects must have discontinued prohibited medications at least 30 days prior to entry.

# 5.5 Adherence Assessment

Throughout the study, the documentation of adherence to study drug is essential. The adherence questionnaire will be completed during each study visit. This will include the ACTG 4-day adherence questionnaire as well as the VAS over the previous 4 week period, except for the week 4 visit where adherence will be assessed since starting medication.

# **6.0 CLINICAL AND LABORATORY EVALUATION**

# 6.1 Schedule of Evaluation

| Schedule of Evaluations | G | Study Weeks of Follow-up | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | | | | | | | | | | |
| | Within<br>30<br>days | 0 | 4 | 12 | 24<br>or<br>72 | 36<br>or<br>60<br>or<br>84 | 48<br>or<br>96 | End of<br>Study or<br>premature<br>D/C | Post-<br>study,<br>3-<br>month | Suspected<br>HIV/STI<br>infection <sup>4</sup> | Interim<br>for<br>Missed<br>Visit <sup>5</sup> |
| Visit Window | | | | ± | 14 da | ys | | | | | |
| Informed Consent | X | | | | | | | | | | |
| Medical/Medication<br>History | X | | | | | | | | | | |
| Documentation of HIV<br>status by rapid HIV test<br>plus NAT or Ag/Ab<br>combo assay | X | | | | | | | | | | |
| Randomization | | X | | | | | | | | | |
| Pre/Post Assessments <sup>1</sup> | | X | | | | | | X | | | |
| iPAD self–administered<br>survey <sup>2</sup> | | X | X | X | X | X | X | X | | X | X |
| Risk reduction<br>Counseling | | X | X | X | X | X | X | X | | X | X |
| Review PrEP adherence (ACTG 4 day and VAS) | | | X | X | X | X | X | X | | X | X |
| Clinical Hx of STI and PREP use | | X | X | X | X | X | X | X | | X | X |
| Assessment of adverse events | | X | X | X | X | X | X | X | | X | X |
| Targeted exam (as clinically indicated) | X | X | X | X | X | X | X | X | | X | X |
| Concomitant medications | | X | X | X | X | X | X | X | | X | X |
| Dispense TDF/FTC (if HIV rapid test negative) | | X | X | X | X | X | X | | | | X |
| Calcium and vitamin D intake | | | | | | X <sup>6</sup> | | | | | |
| Phone call follow-up | | | | | | | | | X | | |

| Schedule of Evaluations | | | Study Weeks of Follow-up | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | | | | | | | | | | |
| | Within<br>30<br>days | 0 | 4 | 12 | 24<br>or<br>72 | 36<br>or<br>60<br>or<br>84 | 48<br>or<br>96 | End of<br>Study or<br>premature<br>D/C | Post-<br>study,<br>3-<br>month | Suspected<br>HIV/STI<br>infection <sup>4</sup> | Interim<br>for<br>Missed<br>Visit <sup>5</sup> |
| Laboratory | | | | | | | | | | | |
| CBC/Chemistry | X | | | | | | | | | | |
| Calculated GFR (serum Cr) | X | | X | X | X | X | X | X | | | X |
| Urine Dipstick | X | | X | X | X | X | X | X | | | X |
| Rapid HIV Test | | X | X | X | X | X | X | X | | X | X |
| STI testing- throat,<br>rectum, urine; blood<br>RPR | | X | | | X | | X | X | | X | X |
| Rectal swab (x2) | | X | | | $X^7$ | | $X^7$ | | | | |
| HBsAg,/HBsAB/HBcAB | X | | | | | | | | | | |
| If HBsAg-/HBsAB-<br>/HBcAb+,<br>Hepatitis B DNA PCR | X | | | | | | | | | | |
| HIV RNA, CD4, HIV genotype, banked PBMC | | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | | $X^3$ | $X^3$ |
| Plasma banked specimen | | X | X | X | X | X | X | X | | $X^3$ | X |
| Banked clotted blood | | X | | | | | | | | | |
| Dried blood spot | | | | X | X | X | X | X | | $X^3$ | X |
| Urine for storage | | X | X | X | X | X | X | X | | X | X |

<sup>&</sup>lt;sup>1</sup> Pre: attitudes toward safe sex, disclosure, access to care, social support, texting ability, Kalichman sexual compulsivity; Post: satisfaction with iTAB; Pre/Post: HIV literacy, stigma and disclosure, AUDIT, DAST-10 <sup>2</sup>includes: risk behavior, adherence assessments, intention to adhere, PHO9, SCID substance use screen

# 6.2 Definitions for Schedule of Events and Timing of Evaluations

#### 6.2.1 Screening Assessments

Occur prior to the subject taking any study medications, treatments, or interventions

Patient Registration: A patient identification number (PID) will be assigned to each patient screened for the study. PIDs should not be reassigned even if the patient fails to enter the study. The PID must be included on every CRF and patient blood sample. Each site must maintain a master list of PIDs in a central location. The patient registration and inclusion/exclusion CRF must be completed on the online system.

<sup>&</sup>lt;sup>3</sup> Perform if HIV+

<sup>&</sup>lt;sup>4</sup> Any time history or symptoms suggest potential HIV or STI, check with study MD for appropriate test <sup>5</sup> Subjects may have an interim visit if past window of scheduled visit, next visit should be back to regular schedule

<sup>&</sup>lt;sup>6</sup> To be performed at week 36 only

<sup>&</sup>lt;sup>7</sup> Performed only once on or after Week 48 coinciding with STI screening (Week 48, 72, or 96)

All subjects interested in screening for the PrEP project will sign an informed consent document that had been approved by local IRB at the site. Screening procedures (see schedule of evaluations) will include: determination of inclusion and exclusion criteria; confirmation of HIV status and screen for acute HIV symptoms. HIV serology will be performed as part of screening, including rapid HIV test and NAT or equivalent (antigen antibody test). Laboratory screening will include CBC, chemistry values, GFR (Cockroft-Galt) LFT and HBsAg. If a subject qualifies and signs consent the window to complete the baseline assessment and start PrEP will be two weeks.

## 6.2.2 Entry Evaluations (day 0)

Randomization: subjects that meet all the inclusion and exclusion criteria will be randomized at their day 0 entry visit. Subjects will be randomized to receive standard of care or the iTAB adherence intervention, stratified by site. Subjects randomized to the iTAB intervention will set up the customized text message stems and enter the timing of the text message reminders; the information will be entered in the online iTAB system by the study coordinator.

At baseline all subjects will receive HIV transmission risk reduction counseling by a health educator and detailed information about the use of PrEP, including the risks, potential adverse events and the critical importance of drug adherence.

# 6.2.3 On-Study Evaluations

After counseling, laboratory testing and randomization, participants will receive sufficient TDF/FTC study medication to last until the next scheduled visit (either 4 or 12 weeks) through the investigational pharmacy. Medication renewals will not be available if a subject misses a scheduled appointment. An informational pamphlet on TDF/FTC will be provided that will summarize the label package insert information for patients (in English or Spanish) with changes made to tailor the information for someone that is not HIV infected. Participants will be directed to take one pill once a day at a convenient routine time. If there are missed doses, participants will be told to take the next scheduled dose on time and not to take any additional pills to catch up. Bottles with any remaining missed doses will be returned to the pharmacy at the time of medication renewal and the number of untaken doses will be recorded. At each clinic visit, TDF/FTC medication adherence will be

reviewed by the clinician, adverse events will be queried and adherence and barriers to adherence will be discussed. All subjects will receive episodic adherence counseling within the confines of routine clinic visit. Each clinic visit will also include blood draw for calculated GFR (serum creatinine) and plasma FTC drug levels, and HIV testing. STI testing including NAT screening for GC and chlamydia from throat and rectal swabs and from urine and RPR from blood will be done at week 0 and every 24 weeks thereafter.

#### Adherence and Behavioral Assessments

We will measure adherence using the ACTG medication adherence questionnaire [25]. At each follow-up visit, the ACTG four-day questionnaire will be administered using the web-based data capture system. The instrument tracks the number of doses skipped over the past four days and reasons why medications may have been skipped. In addition, we will ask their ability to adhere by Likert scale and use the Visual Analog Scale (VAS), which appears as an ordinal scale representing the percent of medication taken relative to that which has been prescribed over the past 4 weeks. Subjects are presented with a line anchored at 0% and 100% and are asked to mark a line on the scale indicating their own PrEP adherence [26].

In the standard study visit, the coordinator will perform HIV testing and blood work, review test results, provide TDF/FTC prescriptions, discuss medication use, adherence, risk reduction and troubleshoot any barriers. The standard behavioral survey will include assessment of TDF/FTC adherence, HIV transmission risk behaviors, substance use, depression scores and other risk behavior details (e.g. sexual partnerships, sexual acts, condom use).

# Laboratory Safety Assessments

At follow-up clinic visits, all participants will have a blood drawn for creatinine clearance estimates. A rapid test for HIV will be performed. HIV test results will be provided during the clinic visit. If there are grade 3-4 adverse events (thought to be related to study medication- see toxicity section) or HIV seroconversion is detected, the participant will be called to discontinue TDF/FTC and to come to the clinic as soon as feasible. Any positive rapid test will be confirmed by Western Blot and HIV RNA; CD4 cell count and an HIV genotype for drug resistance will be done. Newly diagnosed HIV subjects will be counseled and be linked to HIV clinical care within the existing clinic or to another provider

designated by the participant. All PrEP-related clinic visits, laboratory testing and TDF/FTC medication will be provided by the study without charge to the subject.

FTC Qualitative Plasma Concentration as an Adherence Marker:

Plasma will be drawn at every visit starting at week 4 for FTC concentrations. Samples will not be run in real time and will not be available for clinical use.

# Chlamydia, gonorrhea and syphilis testing

Subjects will have day 0 and every 24-week assessment to include urine and swabs from the rectum and throat for NAT testing for Chlamydia and gonorrhea. Blood will be drawn for RPR. In between visits, subjects will be told to come to the study nurse if they experience symptoms of an STI. They will also be asked if they were tested elsewhere between visits. All new STI cases will be referred to their provider or the Department of Health for treatment. They will be given a card to have filled out documenting treatment given, which they will be asked to bring back to their next study visit. All new STI cases will also be counseled on the need for partner therapy and will suggest that they receive assessment and treatment or partner delivered therapy. STI testing can also occur as an interim visit for high-risk exposure or symptoms suggestive of new STI.

# Sexual Risk Counseling

Standard of care HIV risk reduction counseling will be providing to all participants consistent with pre- and post-test counseling for persons receiving community HIV testing. The study will provide streamlined inperson risk reduction counseling at each visit that will use the RESPECT paradigm of focusing on a single risk behavior as identified by the subject. The goal of brief and targeted counseling is to help the individual to identify his most significant risky behavior and to implement concrete actions to decrease the specific risk behavior until the next study visit. Participants will undergo this process at each visit.

## 6.3 Special Instructions and Definitions of Evaluations

# 6.3.1 Documentation of HIV infected status at screening

The lack of HIV-1 infection will be documented by any licensed screening antibody (rapid test plus NAT or Ab/Ag) test. A positive HIV test will be confirmed by a second EIA, Western Blot, or HIV RNA viral load.

# 6.3.2 Medical and Laboratory History

At screening, a medical history will be obtained and will be recorded in the source documents. The medical history should include any previous illnesses that might be consistent with acute HIV infection, history of STI and other routine medical conditions.

## 6.3.3 Medication History

At screening, a medication history (only of those taken within the last 30 days prior to entry) with actual or estimated start and stop dates will be obtained and recorded in the source documents and the concomitant medication CRF, including:

- All prescription medications.
- Non-prescription medications.
- Alternative therapies and/or dietary supplements.
- Allergies to any medications and their formulations must be documented.

#### 6.3.4 Concomitant Medications

During study visits all antibiotics and other concomitant medications taken since the last visit will be recorded in the source documentation and entered into the concomitant medication log CRF.

# 6.3.5 Study Drug Modifications

No modifications of PrEP regimen will be allowed on this study. TDF/FTC may be temporarily held for adverse events as per section 7. TDF/FTC should be discontinued if any criteria for stopping are met (see discontinuation section). Discontinuation will be documented on the TDF/FTC discontinuation CRF.

#### 6.3.6 Clinical Assessments

# Targeted Physical Exam

A targeted physical examination will be based on any signs or symptoms previously identified that the subject has experienced within 30 days of entry or since the last visit. This examination will be performed at all visits when indicated. Documentation must include any symptoms consistent

with acute HIV infection.

Height and Weight

Height and weight will be measured at study entry.

Signs and Symptoms

All signs, symptoms, toxicities and deaths will be documented in the subject's record. At entry, all signs/symptoms experienced within 30 days of entry will be recorded on the CRFs. For all other visits including a suspected HIV infection visit, all Grade > 1 signs and symptoms will be recorded on the CRFs that have occurred since the last visit. Any signs or symptoms that lead to a change in treatment, regardless of Grade, will be recorded on the CRF. The source document will include date of onset and date of resolution, but the CRF will only record prevalence of a given adverse event since the previous study visit.

Refer to the ACTG Table for Grading Adult Adverse Experiences.

## Diagnoses

The following should be recorded on the CRFs: HIV and STI diagnoses, malignancies, new medical conditions and death. The source document must include date of diagnosis and date of resolution.

## 6.3.7 Clinical Assessments for Detected STI

At all visits ask if the participants if they have had an STI in the interim, current symptoms.

# 6.3.8 Laboratory Evaluations

Record all designated laboratory values on the CRFs throughout the course of the study. All baseline values, regardless of toxicity, for specific laboratories will also be recorded on the laboratory CRF including: WBC, neutrophil count, hemoglobin, platelets, creatinine with estimated GFR (Cockcroft-Galt formula), glucose, AST/ALT, alkaline phosphotase and total bilirubin. All values of creatinine with estimated GFR (Cockcroft-Galt Formula) will be recorded in the CRF and performed as per the SOE.

Any laboratory toxicities that lead to a change in treatment, regardless of Grade, will be recorded on the adverse event CRF.

Refer to the Division of AIDS Table for Grading Adult Adverse Experiences.

# 6.3.9 Urinalysis

A dipstick urine test will be done at screening and every visit after day 0. Protein, glucose and leukocyte esterase will be recorded in the CRF.

# 6.3.10 T-cell counts and Virology tests

## Plasma HIV-1 RNA

An HIV-1 RNA viral load will be performed at the site's local laboratory within 7 days of a new positive antibody test or NAT.

An HIV drug resistance test should be performed with detectable viral load of greater than 500 copies/mL.

CD4 T-cell enumeration will be performed to obtain absolute CD4+/CD8+ count and percentages within 7 days of new HIV diagnosis.

# 6.3.11 Stored Plasma and other specimens

Stored plasma will be collected at day 0, at all visits and with any new HIV diagnosis.

\*Specimens will be stored at the site's local laboratory and batched shipped to the central laboratory (UCSD) after completion of the study.

#### 6.3.12 *Pharmacokinetic Studies*

At each visit, record the time and date of the last 3 doses of TDF/FTC medication in the CRF. Dried blood spots will be stored at -80 at each visit beginning at Week 12 for possible future use for plasma and intracellular TFV and FTC pharmacology.

#### 6.3.13 *Questionnaires*

At each visit, the subject should complete the self-reported questionnaires.

## 6.3.14 Rectal swabs

At day 0 and at one additional time point on or after Week 48, all subjects will have a rectal swab stored for possible future studies of the gut microbiome. These tests will be done in retrospect and not available for the subjects.

- 6.3.15 At day 0, all subjects will have blood stored for future use to examine host DNA. Subjects will sign a consent that informs them of the storage of material for possible host genomic testing.
- Participants will be asked to recall food items eaten over the last 3 days at the week 36 visit. The calculator used in the ACTG 5280 study, which is adopted from the USDA database, will be used to quantify vitamin D and calcium intake (see Appendix VI).

# 6.4 Schedule of Evaluations for Subjects On-Study, Off-Medications

6.4.1 At any point, subjects may elect to stop study medications but remain on study. Subjects that stay on study but stop medications will not be allowed to resume again.

Subjects will follow the same schedule as defined in Section 6.1 until the end of study. Study medications will not be dispensed at clinic visits, and evaluations related to counseling or monitoring of medications (including urine dipstick and serum creatinine) will not be performed. These include Adherence and Risk-reduction counseling and collection of dried blood spots. If the subject was randomized to the iTab arm, their account will be switched to "inactive."

STI and HIV rapid test screenings and questionnaires will still be administered as the schedule dictates.

# 6.5 End of Study Visit and Post-study 3-month Follow-up

6.5.1 At the End of Study (EOS) visit, subjects will be asked to complete additional questionnaires in addition to completing regular procedures. These surveys will assess subjects' experiences over the course of the study including changes in their medical insurance status, access to other health services, changes in their perceptions of PrEP and of their own health, and their opinions on the intervention.

Upon completion, subjects will not be dispensed PrEP and will be discontinued from the study.

Subjects that express the desire to continue PrEP after completing the study will be provided information regarding access and payment strategies.

6.5.2 Subjects that complete CCTG 595 will be approached EOS and asked to join a supplement-funded extension, consisting of a one-time phone call follow-up scheduled for 3 months post-study. The purpose of this extension is to examine sexual risk compensation and the impact of transition after cessation of study-provided PrEP.

Written consent will be obtained at EOS; subjects that have already completed their EOS visit will be contacted and verbal consent will be obtained over the phone.

At 3 months post-study, subjects will be contacted over the phone and asked questions regarding their current HIV status, their ability to access and maintain their PrEP regimen after EOS, and their ability to obtain health insurance coverage. If subject is off PrEP and/or has no health insurance, the subject will be asked for their reasons and possible barriers. Subjects will also be asked an abbreviated number of questions from surveys similar to those done during the main study, including measures assessing risk compensation, perceptions of PrEP efficacy, and adherence (if on PrEP).

#### 7.0 TOXICITY MANAGEMENT

The management of medication related toxicities should be undertaken by the local investigators, with guidance available from the protocol team, protocol pharmacist and pharmaceutical sponsor, to ensure the optimal safety and efficacy for the individual subject.

# 7.1 General Management for Grade 1-4 Events

#### 7.1.1 Grade 1 or 2

Subjects who develop a Grade 1 or 2 adverse event or toxicity may continue TDF/FTC without alteration of the dosage, except as noted below. Persistent grade 1 or 2 toxicity should be discussed with the protocol team. Those subjects experiencing Grades 1 or 2 adverse events which results in discontinuation of the TDF/FTC should continue to be followed on study, but off study medication.

#### 7.1.2 Grade 3

Management of Grade 3 toxicities should be discussed with the protocol team via email. Please refer to the subsequent sections for management of specific events.

In the event that a subject develops a **symptomatic** Grade 3 reaction considered to be TDF/FTC-related, the study drug should be discontinued and the subject should be followed weekly until resolution of the adverse event. Once Grade 3 is resolved the subject should be followed on-study, but off study medication. For subjects with asymptomatic Grade 3 toxicity or laboratory abnormalities, the protocol team should be consulted for possible re-introduction of TDF/ FTC.

#### 7.1.3 Grade 4

Subjects who develop a Grade 4 adverse event or toxicity judged to be TDF/ FTC-related will have the study drug permanently discontinued. For other Grade 4 events, if the toxicity or laboratory elevation is thought not to be due to TDF/FTC, TDF/FTC may be continued and laboratories repeated within 2 weeks (for example for asymptomatic elevation of CPK or triglycerides). If it is not possible for the investigator to discern another causative agent/ condition or if TDF/FTC could be the causative agent, then TDF/FTC must be discontinued. Subjects experiencing Grade 4 adverse events requiring permanent discontinuation of TDF/FTC therapy should be followed weekly until resolution of the adverse event. Once Grade 4 is resolved the subject should be followed on-study, but off study medication.

## 7.2 Management for Specific Adverse Events

#### 7.2.1 Rash

Grade 1 or 2

TDF/FTC may be continued without interruption. Subjects with a Grade 1 or 2 rash may be treated symptomatically with permitted antipyretic, antihistamine and/or non-steroidal anti-inflammatory medications, but should be monitored closely by the local investigator.

Grade 3 or 4

Grade 3 or 4 rash necessitates that TDF/FTC be held unless the rash is determined to be unrelated to TDF/FTC. The rash should be followed closely for resolution and the subject followed on-study, off study medication.

# 7.2.2 Nausea and Vomiting

Grade 1 or 2

TDF/FTC may be continued without interruption. Subjects with Grade 1 and 2 nausea or vomiting may be treated symptomatically with permitted oral antiemetic therapies or antiemetic suppositories. Subjects will be instructed to take medications with food.

Grade 3 or 4

Subjects with Grade 3 TDF/FTC-related nausea and vomiting should interrupt TDF/FTC until the toxicity grade returns to Grade < 2 or to baseline and be treated symptomatically. After discussion with the protocol team and if the subject is willing, the TDF/FTC may be resumed when symptoms have resolved. If Grade 3 nausea and vomiting recurs upon the resumption of TDF/FTC despite symptomatic treatment, TDF/FTC should be discontinued. Grade 4 nausea or vomiting will lead to permanent discontinuation of drug. Once resolved, the subject should be followed on-study, but off study drug.

# 7.2.3 Diarrhea

Grade 1 or 2

TDF/FTC may be continued without interruption. Subjects with diarrhea of any toxicity grade may be treated symptomatically with permitted antimotility agents.

Grade 3 or 4

For grade 3 diarrhea that is unresponsive to antimotility agents and for which an alternative etiology (e.g., infectious diarrhea) is not established, TDF/FTC should be interrupted until resolution of diarrhea to Grade  $\leq 2$  or baseline. If Grade  $\geq 3$  diarrhea recurs upon the resumption of study medications, TDF/FTC should be permanently discontinued. Grade 4 will lead to permanent discontinuation of study medication.

# 7.2.4 Hyperglycemia

Fasting hyperglycemia of > 110 to 125 mg/dL is considered evidence of impaired glucose tolerance. A fasting blood glucose level above 126 mg/dL is highly suggestive of diabetes mellitus. Subjects with fasting hyperglycemia may continue TDF/FTC at the discretion of the investigator but should be discussed with the protocol team via email. A confirmatory fasting glucose will be obtained within 4 weeks and prior to the institution of medical therapy. Hyperglycemia may be treated with oral hypoglycemic agents or insulin according to standard guidelines. Abnormal glucose levels will be monitored closely, and further laboratory repeats will be at the discretion of the site PI.

# 7.2.5 AST/ALT Elevations

Grade 1 or 2

TDF/FTC may be continued. Tests should be repeated and reassessed within 2 weeks if AST/ALT results are > grade 2

## Grade 3

All grade 3 or 4 elevations of AST/ALT should be discussed immediately with the protocol team via email. TDF/FTC may be continued for Grade 3 AST/ALT elevations at the discretion of the site investigator after discussion with the protocol team. Careful assessments should be done to rule out the use of alcohol, non-study medication-related drug toxicity, or viral hepatitis as the cause of the Grade 3 elevation.

#### Grade 4

TDF/FTC will be permanently discontinued for AST or ALT Grade 4 elevations, and the protocol team will be notified. The subject should have repeated AST or ALT evaluations until the levels have returned to < grade 2 or baseline. Once the AE is resolved, the subject should be

followed on-study, but off study medication.

#### 7.2.6 Creatinine Elevations

TDF/FTC will be discontinued if the creatinine clearance is confirmed to be < 50 mL/min. Subjects should be followed as medically indicated until the creatinine returns to baseline. The protocol team will be notified within 48 hours of any permanent therapy discontinuations due to change in creatinine clearance.

If the serum creatinine increases more than 0.3 from baseline, the level should be repeated in 2 weeks. Elevations in creatinine will be monitored closely, and further laboratory repeats will be at the discretion of the site PI.

# 7.2.7 Anemia/Neutropenia

Subjects with Grade 3 anemia or neutropenia attributed to TDF/FTC should have all study treatment interrupted until the abnormality returns to Grade  $\leq 2$ . Therapy may be resumed after the anemia or neutropenia has returned to Grade  $\leq 2$ . If Grade 3 anemia or neutropenia recurs, TDF/FTC will be discontinued, and the protocol team will be notified.

Grade 4 anemia or neutropenia will result in permanent discontinuation of study medication if it is due to TDF/ FTC.

#### 8.0 CRITERIA FOR TREATMENT DISCONTINUATION

Diagnosis of HIV infection.

# 8.1 Criteria for Discontinuation from Study

8.1.1

- Request by the subject to withdraw.
  Request of the primary care provider if s/he thinks the study is no longer in the best interest of the subject.
- 8.1.4 Clinical reasons believed life threatening by the study physician, even if not addressed in the toxicity management of the protocol, and can no longer continue in follow up.
- 8.1.5 Subject judged by the investigator to be at significant risk of failing to

- comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.
- 8.1.6 At the discretion of the CCTG, FDA, CHRP or pharmaceutical sponsors.
- 8.1.7 Misses two consecutive scheduled visits prior to 48 weeks.
- 8.1.8 Misses one scheduled visit after 48 weeks.

## 9.0 STATISTICAL CONSIDERATIONS

A formal Statistical Analysis Plan (SAP) will be drafted and finalized prior to database lock. The SAP will contain a more detailed and/or comprehensive presentation of statistical methods, attention to any changes of substance to planned analysis procedures relative to those indicated in the protocol, and is the final authority for all statistical analyses. The following section briefly describes the planned statistical analyses. In case the language in this section differs from the language in the SAP, the SAP takes precedence.

# 9.1 Primary Endpoints

Adherent to PrEP through 48 weeks is defined as a composite endpoint of continuing on study (made all scheduled visits within window in the 48 week period) and on study medication and greater than or equal to 90% adherent to medication defined by self-report of  $\geq$  18 of 20 doses of medication on the 5 ACTG adherence questionnaires at weeks 4, 12, 24, 36 and 48. Missing adherence forms will be imputed as no doses taken.

# 9.2 Secondary Endpoints

- 9.2.1 Adherent to PrEP by FTC measurement at 48 weeks and at the end of study follow-up is defined by attending all scheduled visits and having detectable FTC.
- 9.2.2 Adherent to PrEP in continuous follow up is aggregate percentage of selfreported ACTG days of adherence where missed schedule visits are counted as 0/4 days.
- 9.2.3 Poor adherence is considered those with <90% self-reported adherence by ACTG 4 day survey or if discontinued drug. Subgroup analysis should explore the endpoint for discontinuation for reasons other than quit drug for lack of risk or confirmed adverse event.
- 9.2.4 Safety and tolerability defined as: i) discontinuation of TDF/ FTC for any

toxicity; ii) grade 2 or higher adverse event or laboratory toxicity; iii) serious adverse event; iv) death

#### 9.3 Randomization and Stratification

We will conduct an open-label, randomized, controlled, two-arm, clinical strategy trial for PrEP adherence. Subjects will be randomized (1:1) to one of two arms: the **Standard of Care** (SoC) or the **iTAB** enhanced adherence arm. Randomization will be stratified by clinic site. A total of 400 subjects (200 per arm) will be randomized and followed in the study for 48 weeks after enrollment of the last subject.

Once eligibility and consent are confirmed, randomization will occur using the web-based CFAR BIT data management system.

# 9.4 Study Power and Sample Size Justification

The primary objective for this study is to compare the proportion of subjects that reach the composite endpoint, defined as: continued retention and adherence to PrEP. Sample size calculations were based on a two-sided, two- sample binomial test to compare the differences in composite endpoint proportions between the intervention arm and the standard of care arm. Since attrition is a component of the composite endpoint, attrition rates are not used as an adjustment in the power calculations. Assuming 200 subjects per group in each of the two groups (for a total of 400 subjects) and alpha set to 0.05, we have 94% power to detect a difference of 15%, assuming that 30% with a composite endpoint rate in standard of care and that 15% with endpoint in the intervention arm. We have 84% power to detect as small a difference of 13% between the two groups (i.e., 30% versus 17%).

# 9.5 Monitoring

The study team will review all adverse events during PrEP therapy by cumulative reports, both arms combined in aggregate, on a monthly basis. Adverse events will be graded using the ACTG toxicity grading scale and recorded using standard CCTG AE electronic data capture. The study investigators will monitor safety events in aggregate on monthly team calls. An independent Data Safety and Monitoring Board (DSMB) will not be used for this study.

# 9.6 Analyses

# 9.6.1 Statistical Analysis Plan

In general, analyses will incorporate the modified intent-to-treat (mITT) principle, namely, all randomized participants dispensed study medication will be included in the analysis. The primary analysis compares the iTAB enhanced proportion of adherence to the SOC arm.
For all secondary analyses of interest, no adjustments for multiple comparisons will be made and a p-value of 0.05 will be considered statistically significant. Demographic and baseline measurement variables will be summarized via standard descriptive statistics. There will be no interim analyses for futility or efficacy conducted.

## 9.6.2 Analysis of Primary Outcome

The primary analysis will use a two-sample binomial test for proportions to determine if the intervention arm will produce an improved composite endpoint rate compared to the standard of care arm. Fisher's exact test will be used along with a 95% confidence interval. As a sensitivity analysis, the two components of the composite primary endpoint will be analyzed separately (retained on PrEP and Adherence > 90%). A Fisher's exact test will be used to compare rates of study discontinuation between the active intervention arm versus standard of care arm.

## 9.6.3 Analysis of FTC Plasma Concentrations

With repeated qualitative FTC assays in each subject over time, adherence will be defined using a continuous and categorical metric. The percent adherence, calculated as number of detectable samples divided by total number of samples measured, will be compared between intervention and control using a two- sample t-test (or an appropriate non-parametric alternative if parametric assumptions fail). For strict mITT analyses, subjects that are missing a FTC concentration at any time point (whether due to missed visit or TDF/ FTC discontinuation) will be defined as having an undetectable FTC concentration while per protocol analyses will consider only available data (i.e., no imputation for missing values). A categorical metric of good adherence (> 90% of concentrations detectable) will be compared between intervention and control with the Fisher's exact test.

## 9.6.4 Analysis of additional Secondary outcomes

The incidence rate of STI will be compared between SOC and ALERT- iTAB intervention arms using Fisher's exact test as will the rate of HIV seroconversion between groups (the rate of new HIV is expected to be low). In order to evaluate hypothesis 3c (factors associated with the composite primary endpoint of on therapy and adherence > 90%), multivariable logistic regression models will also be used. A subgroup analysis by treatment arm will be conducted, looking at each arm separately. Descriptive analysis will be performed within each subgroup

to compare adherent versus non-adherent subjects. The models will include the following potential covariates: demographics, ongoing substance use, untreated mental illness, socioeconomic status, HIV risk transmission behaviors, low health/ HIV and system literacy, fear of disclosure and non-English. Further, any covariates (including stratification factors) that are simultaneously unbalanced at baseline (univariate p <0.10) and associated with the outcome (univariate p<0.15) will be included in the model as observed confounders. Sub-group analyses based on race/ ethnicity, gender, primary language, socioeconomic status by randomization arm will also be conducted. Secondary endpoints for adherence will be analyzed analogously to the primary endpoint.

9.6.5 Safety and tolerability of daily TDF/FTC given for PrEP including discontinuation for any adverse event, serious adverse events and adverse events (grade 2 or higher) will be compared between study arms. Descriptive statistics will be used to characterize safety events. Fisher's exact test will be used to compare discontinuation rates due to safety and incidence rates of adverse events and serious adverse events. The time to TDF/ FTC discontinuation for adverse events will be compared between groups using the log-rank test and plotted using Kaplan-Meier curves. Similar analysis will be done for the time to discontinuation for any reason (including drop-out or subject electing to stop PrEP due to lack of perceived risk for HIV).

## 10.0 PHARMACOLOGY PLAN

## 10.1 Sample Assay Methods

FTC concentrations will be measured in the Pediatric Clinical Pharmacology Laboratory of the University of California, San Diego by a validated, Liquid Chromatography-Mass Spectrometry (LC-MS) method. The laboratory is registered with the ACTG Quality Assurance/Quality Control proficiency testing program [27] and successfully completes proficiency testing for the accuracy and precision of the FTC assay every 6 months. Inter-assay variability is less than 6% for low, middle and high controls. The lower limit of detection of FTC is approximately 1 ng/mL (the lower limit of quantitation is 11.8 ng/mL). For qualitative assays, unknown samples will be measured in the presence of internal standard to determine if the FTC ion peak is present (≥ 1 ng/mL) or absent (< 1 ng/mL). Stored plasma samples will be bulk testing of qualitative presence of FTC at the end of follow-up. Additional pharmacology analyses will be done in retrospect and the specific analysis will be included in the SAP prior to data log and sample testing.

#### 11.0 DATA COLLECTION AND MONITORING AND ADVERSE EVENT REPORTING

### 11.1 Records to be Kept

Case report forms (CRFs) will be provided for each subject. Subjects must not be identified by name on any CRFs. Subjects will be identified by the PID provided by the CCTG Data Unit upon registration and the linkage to the PID will be kept in paper copy only in a locked cabinet in a secure office at the study sites available only to the site investigators.

Subject self-reported surveys that are performed electronically will be automatically stored in the electronic database secured by the CFAR BIT group for the CCTG.

## 11.2 Role of Data Management

- 11.2.1 Instructions concerning the recording of study data on CRFs will be provided by the CCTG Data Unit.
- 11.2.2 It is the responsibility of the CCTG Data Unit to assure the quality of computerized data for this study.

## 11.3 Clinical Site Monitoring and Record Availability

- 11.3.1 Site monitors provided by the CCTG will visit participating clinical research sites to review the individual subject records including consent forms, CRFs, supporting data, laboratory specimen records, and medical records (e.g., physician progress notes, nursing notes, individual hospital charts), to ensure protection of study subjects, compliance with the protocol and accuracy and completeness of records. The monitors also will inspect sites's regulatory files to ensure that regulatory requirements are being followed.
- 11.3.2 The investigator will make study documents (e.g., consent forms and CRFs) and pertinent hospital or clinic records readily available for inspection by the local IRB or the site monitors.

## 11.4 Serious Adverse Experience (SAE) Reporting

Serious adverse events are not expected in this study. All SAEs must be documented on the SAE Reporting Form within 5 working days of site awareness of the event and submitted to the CCTG Data Unit.

#### 12.0 HUMAN SUBJECTS

## 12.1 Institutional Review Board (IRB) Review and Informed Consent

This protocol and the informed consent document and any subsequent modifications will be reviewed and approved by the IRB or ethics committee responsible for the oversight of the study. A signed consent form will be obtained from the subject. The consent form will describe the purpose of the study, the procedures to be followed and the risks and benefits of participation. A copy of the consent form will be given to the subject.

## 12.2 Subject Confidentiality

All laboratory specimens, evaluation forms, reports, and other records that leave the site will be stripped of any patient identifiers (name, birthdate, medical record number) and only identified by the coded PID in order to maintain subject confidentiality. All records will be kept locked. All computer entry and networking programs will be done with coded numbers only and analyzed centrally without any possibility of linking subject identity with subject data. Clinical information will not be released without written permission of the subject, except as necessary for monitoring by IRB and governmental agencies.

## 12.3 Study Discontinuation

The study may be discontinued at any time by the IRB or other government agencies as part of their duties to ensure that research subjects are protected.

#### 13.0 PUBLICATION OF RESEARCH FINDINGS

Publication of the results of this trial will be governed by CCTG policies. Any presentation, abstract or manuscript will be made available for review by pharmaceutical supporters prior to submission.

#### 14.0 BIOHAZARD CONTAINMENT

As the transmission of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood and blood products; appropriate blood and secretion precautions will be employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the Centers for Disease Control and Prevention and the National Institutes of Health.

All infectious specimens will be transported using packaging mandated in the Federal Code of Regulations, CDC 42 CFR Part 72. Please also refer to individual carrier guidelines, e.g., FedEx, Airborne, for specific instructions.

#### **15.0 REFERENCES**

- K. HSeal, et al.; A randomized controlled trial of monetary incentives vs. outreach to enhance adherence to the hepatitis B vaccine series among injection drug users; Drug Alcohol Depend; 2003
- J. M. FitzGerald, et al.; Use of incentives to increase compliance for TB screening in a population of intravenous drug users. Vancouver Injection Drug Use Study Group; Int J Tuberc Lung Dis; 1999
- 3. D. B. Marlowe, et al.; Day treatment for cocaine dependence: incremental utility over outpatient counseling and voucher incentives; Addict Behav; 2003
- 4. L. W. Kimbrough, et al.; Accessing social networks with high rates of undiagnosed HIV infection: The social networks demonstration project; Am J Public Health; 2009
- 5. J. L. Richardson, et al.; Using patient risk indicators to plan prevention strategies in the clinical care setting; Journal of acquired immune deficiency syndromes; 2004
- 6. M. R. Golden, et al.; Peer referral for HIV case-finding among men who have sex with men; AIDS; 2006
- 7. S. R. Morris, et al.; Evaluation of an HIV nucleic acid testing program with automated Internet and voicemail systems to deliver results; Ann Intern Med; 2010
- 8. A. S. Klovdahl, et al.; Social networks and infectious disease: the Colorado Springs Study; Soc Sci Med; 1994
- 9. R. M. Grant, et al.; Preexposure chemoprophylaxis for HIV prevention in men who have sex with men; N Engl J Med; 2010
- 10. Interim guidance: preexposure prophylaxis for the prevention of HIV infection in men who have sex with men; MMWR Morb Mortal Wkly Rep; 2011
- 11. N. A. Christakis, et al.; Social network sensors for early detection of contagious outbreaks; PLoS One; 2010
- 12. S. F. University of California; http://clinicaltrials.gov/ct2/show/NCT01377857;
- 13. M. J. Mimiaga, et al.; Preexposure antiretroviral prophylaxis attitudes in high-risk Boston area men who report having sex with men: limited knowledge and experience but potential for increased utilization after education; Journal of acquired immune deficiency syndromes; 2009
- 14. D. R. Bangsberg; Preventing HIV antiretroviral resistance through better monitoring of treatment adherence; The Journal of infectious diseases; 2008
- 15. B. Singh, et al.; Alterations in head and neck cancer occurring in HIV-infected patients-results of a pilot, longitudinal, prospective study; Acta Oncol; 1999
- 16. E. J. Mills, et al.; Adherence to HAART: a systematic review of developed and developing nation patient-reported barriers and facilitators; PLoS Med; 2006
- 17. A. Ammassari, et al.; Timed Short Messaging Service Improves Adherence and Virological Outcomes in HIV-1-Infected Patients With Suboptimal Adherence to Antiretroviral Therapy; Journal of acquired immune deficiency syndromes; 2011
- 18. K. Voigt; Incentives, health promotion and equality; Health Econ Policy Law; 2010
- N. M. Petry; Contingency management treatments: controversies and challenges;
   Addiction; 2010

- 20. J. Lorvick, et al.; Incentives and accessibility: a pilot study to promote adherence to TB prophylaxis in a high-risk community; J Urban Health; 1999
- 21. D. C. Perlman, et al.; Impact of monetary incentives on adherence to referral for screening chest x-rays after syringe exchange-based tuberculin skin testing; J Urban Health; 2003
- 22. Hepatitis B vaccination for injection drug users--Pierce County, Washington, 2000; MMWR Morb Mortal Wkly Rep; 2001
- 23. F. Huang, et al.; Concomitant administration of BILR 355/r with emtricitabine/tenofovir disoproxil fumarate increases exposure to emtricitabine and tenofovir: a randomized, open-label, prospective study; Basic Clin Pharmacol Toxicol; 2011
- 24. D. A. Parks, et al.; Steady-state amprenavir, tenofovir, and emtricitabine pharmacokinetics before and after reducing ritonavir boosting of a fosamprenavir/tenofovir/emtricitabine regimen from 200 mg to 100 mg once daily (TELEX II); HIV Clin Trials; 2009
- 25. M. A. Chesney, et al.; Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committee of the Adult AIDS Clinical Trials Group (AACTG); AIDS Care; 2000
- 26. K. R. Amico, et al.; Visual analog scale of ART adherence: association with 3-day self-report and adherence barriers; J Acquir Immune Defic Syndr; 2006
- 27. D. T. Holland, et al.; Quality assurance program for clinical measurement of antiretrovirals: AIDS clinical trials group proficiency testing program for pediatric and adult pharmacology laboratories; Antimicrob Agents Chemother; 2004

#### **16.0 APPENDICES**

**APPENDIX I: SAMPLE OF INFORMED CONSENT** 

# UNIVERSITY OF CALIFORNIA - SAN DIEGO CONSENT TO ACT AS A RESEARCH SUBJECT

**TITLE**: CCTG 595: A Multicenter, Randomized Study of Text messaging to improve Adherence to PrEP during In Risky MSM (TAPIR)

Drs. Sheldon Morris, Constance Benson, Maile Karris, Scott Letendre, Susan Little,, Jill Blumenthal, Richard Haubrich, David Moore, and their associates are conducting a research

study sponsored by the California Collaborative Treatment Group (CCTG) to determine if using text-message based adherence interventions can improve retention and adherence to Pre-exposure Prophylaxis (PrEP) in HIV-negative men who have sex with men (MSM) and male to female transgenders who are at high-risk for HIV acquisition.

Before you can decide whether or not to volunteer for this study, we would like to let you know about the study's purpose, how it may or may not help you, any risks to you, and what is expected of you. This process is called informed consent.

The FDA recently approved a fixed dose combination of tenofovir disoproxil fumarate/ emtricitabine (TDF/FTC) to reduce the risk of HIV infection in uninfected individuals who are at high risk of HIV infection and who may engage in sexual activity with HIV-infected partners. From other studies, we know that the use of PrEP in HIV negative individuals has been shown to reduce acquisition of HIV among at-risk individuals. We also know that the more a person takes the PrEP medication (called adherence), the more effective it is.

The purpose of this study is to evaluate a promising method of reinforcing PrEP adherence using text message. In this study, we will hope to learn if text message reminders increase PrEP adherence.

You have been asked to participate in this study because you are HIV-negative and are sexually active with men and are at ongoing risk for acquiring HIV.

#### **DURATION OF THE STUDY**

The study will enroll about 400 people at all participating sites. We plan to enroll about 250 subjects at UCSD. If you participate in the study, you have up to 11 visits at the UCSD Antiviral Research Center (AVRC) for at least 1 year and up to a maximum of 2 years.

## **PROCEDURES**

If you agree to participate in this study, the following will happen:

To see if it is okay for you to participate in this study, you will first come to the clinic for a study visit known as a "screening" visit. At your first visit, this consent form will be reviewed with you and you will be asked to sign it.

Once you sign this form and agree to participate, we will confirm your HIV status, screen for symptoms of recent HIV infection and perform a medical/medication history. You will also be asked to complete a survey on a computer. Because you will be asked questions about your sexual, and drug using history and practices, the computer you will use to complete this survey will be in a private location in the clinic.

Approximately 2-3 tablespoons of blood will be drawn for laboratory tests including blood count, chemistry values, liver function and kidney tests, HIV test and Hepatitis B will be obtained.

Your Screening visit will take about 1 to 2 hours.

Entry Visit:

The information gathered at your screening study visit will determine if you are able to take part in this study. If you qualify for the study, you will return to the clinic for your "entry visit". At your entry visit, you will have the following procedures done:

- A medical and medication history will be taken. This will include any recent or previous drug history and anti-HIV drugs you have taken.
- **◆** Sample will be obtained for the following tests:
  - Screening for sexually transmitted infections (STIs). In addition to the urine and blood sample, a throat and rectal swab will need to be done in order to screen for STIs. These collected samples and swabs will be tested to see if you have gonorrhea, Chlamydia, or syphilis. These samples will be taken at entry and every 24 weeks after your entry visit.

The test in your throat will be done by inserting a cotton swab (Q-Tip) into your mouth and gently turning it to collect the sample.

The test in your rectum will be done by carefully inserting a cotton swab and gently turning it to collect the sample.

If your tests show that you have an STI, our study staff will refer you to your medical provider for treatment. If you do not have a provider, you will be referred to the public health clinic where treatment will be provided at a small fee or free to those who cannot afford this fee. According to California state law, study staff are required to give the public health department the names, contact information and treatment records of people who have a positive test result for chlamydia, gonorrhea or syphilis.

- Blood to be stored for future study-related tests including the amount of PrEP medicine in your blood.
- An additional sample from your throat and rectum may be taken for future study related tests.
- Approximately 2-3 tablespoons of blood will be drawn at the entry visit.

At this entry visit, you will be randomized (assigned by chance, like flipping a coin) into one of the following two groups. You have an equal chance of being assigned to either group.

- Group 1: PrEP daily, HIV/STI screening, adherence and risk behavior counseling, and safety monitoring
- Group 2: PrEP daily, HIV/STI screening, adherence and risk behavior counseling, and safety monitoring as well as iTAB text adherence reminders

The PrEP medicine is TDF/FTC combination pill. At this study, visit Groups 1 and 2 will complete a survey that is done on a computer in a location that is private so no one can see the answers to any questions you type into the computer. The survey will ask specific question about your sex life and recreational drug use. Groups 1 and 2 will receive detailed information about the use of PrEP, including the risks, potential adverse events and the importance of drug adherence. You will be provided with enough TDF/FTC to last until your next visit. You will be instructed to take one pill once a day at a convenient routine time.

Group 2 will be introduced to the iTAB (Individualized Texting for Adherence Building) system by a study worker who will help you select and refine 10 personal reminders from a list of predetermined reminders. The study worker will help you to set adherence reminders that are sent at times consistent with when you typically take medications. You will be provided with information about how the iTAB texting system works. If you are in Group 2 and do not have a cell phone, you will be provided with one at this time.

This study visit will take about 1 - 2 hours.

Clinic Study Visits (Month 1, 3, 6, 9, 12 and every 3 months thereafter)

You will come to the clinic at 1 month and then every 3 months (3, 6, 9, 12 and every 3 months) for a study visit. At these study visits, you will have the following procedures done:

- ◆ A urine sample and approximately 2-3 tablespoons of blood will be drawn for the following tests:
  - ◆ Laboratory tests including kidney tests and HIV testing. You will find out the results of the HIV test during each visit.
  - Screening for sexually transmitted infections (STIs). In addition to the urine and blood sample a throat and rectal swabs will need to be done in order to screen for STIs. These collected samples and swabs will be tested to see if you have gonorrhea, Chlamydia, or syphilis. Samples will be collected as described above. Screening for STI will be done every 6 months after your entry visit.
  - Blood to be stored for future study related tests including blood levels of PrEP medications.
  - ◆ An additional sample from your throat and rectum may be taken for future study related tests.

At your study visits, you will complete a survey done on a computer that is in a location that is private so no one can see the answers to any questions you type into the computer. The survey will ask specific question about your sex life, recreational drug use, how well you took your PrEP medication and questions about your mood. You will receive risk assessment and adherence counseling. Study medication use and adverse events will be reviewed by study personnel.

Each study visit will take about 1 hour.

## Additional Study Visits

If at anytime during the study you think you might have gotten an STI because someone you had sex with tells you they were diagnosed with one or you are having symptoms that you think are those of a STI or acute HIV infection you need to tell your study staff immediately so you can get an appointment to be checked. If you come for an additional visit because you think you have an STI, tests for STI will be done (blood and urine sample and rectal or throat swabs). An HIV test will be done if you think you were exposed to HIV or if you have symptoms of HIV.

If you have a positive test for HIV during the study, additional blood tests will be done to find out the amount of HIV virus in your blood, to check the HIV strain for drug resistance and to look at your immune system (T-cell count). You will be referred for HIV care.

## Contact for Future Studies:

There may be other studies that are being conducted at the AVRC for which you may qualify. You may be asked to participate in one or more of these additional studies. Are you willing to be contacted for future research studies by our staff?

| NC |
|----|

#### RISKS/DISCOMFORTS:

Participation in this study may involve some added risks or discomforts. These include:

Study drug side effects

You may experience side effects from the study medication which include but are not limited to nausea, vomiting, diarrhea, abdominal pain, rash, dizziness, body weakness, fever, weight loss, allergic reaction, elevations in liver tests and impairment in kidney function. Any side effect will be carefully evaluated and managed according to standard guidelines and may require discontinuation of the study drug.

A small number of people in this study may have these side effects or other side effects that we do not know about. However, we will screen your kidney function and overall health before you join the study. This will reduce the chances of having any side effects.

*Text messaging adherence reminders* 

You may feel increased stigma or intrusions of privacy or confidentiality when receiving text message reminders to take your medication.

Drug Resistance

In previous studies, it was found that a few people became HIV infected despite taking the study drug. Should you become HIV infected during the course of the study, there is a very small chance that you may develop resistance to the study drug while participating in the study.

Risks of drawing blood

You may experience temporary discomfort from the blood draws. The needlesticks may cause local pain, bleeding, bruising and swelling, as well as lightheadedness, dizziness and rarely, blockage of the vein, fainting and/or a local infection.

Sexually Transmitted Infections (STIs)

You may experience some anxiety or embarrassment when being tested for sexually transmitted infections. If you are found to have a sexually transmitted disease, an appropriate referral for

treatment will be made to one of several free public health clinics in your area.

Since this is an investigational study, there may be other unknown risks that are unforeseen or at this time cannot be predicted. You will be told of any significant new risks. If you have questions concerning the study, ask the study staff.

Sample Storage

As a result of your participation in this study, you are now being asked to take part in an optional part of the study involving the collection of blood and swabs for genetics testing and storage. It is up to you to decide whether to participate.

We would like your permission to store some of your blood and swab samples for future DNA research. As scientific discoveries are made, valuable research can be done in the future on samples collected today. Therefore, we ask your permission to store your DNA sample to allow for research to be done in the future.

If you agree, some of your blood, swabs, and oral specimens that are left over after all required study testing is done may be stored for future use for approved research. Your left over blood may be stored for an indefinite length of time. Because research using your left over blood will be done in the future, you will not be told the results of the research done on these samples. You may cancel your permission to store and use your left over blood at any time and still remain in this study.

| obtained not be lis | dicate below whether or not you agree to have your blood and swabs stored, which was as part of this study. All samples will be identified by a number only (your name will ted on the sample) _You agree that your left over samples can be used for future HIV/AIDS-related |
|---|---|
| (Initials) | research. |
| (Initials) | You do not agree that your left over samples can be used for future HIV/AIDS-related research. |
| (Initials) | You agree that your left over samples can be used for future DNA-related research. |
| (Initials) | You do not agree that your left over samples can be used for future DNA-related research |

## STORED SAMPLES

Some of your blood, swabs, and oral specimens obtained as part of this study will be stored

indefinitely and may be used for approved HIV/AIDS-related research in the future. You will not be identified by name in any testing and your confidentiality will be maintained. Specimens will be identified only by an identification number (your name will not be listed on the sample). All of the individuals receiving these specimens will be scientific partners in this study. Your blood, swabs, and oral specimens and the DNA that it contains may also be used in additional research to be conducted by the University of California personnel collaborating in the research. This blood, swabs, and/or oral specimens and its derivatives may have significant therapeutic or commercial value. You consent to such uses.

The University has policies and procedures to ensure your confidentiality. We will use our best efforts to ensure that your identity and test results will not become known outside the research program, which if released, could affect your employment and ability to obtain insurance. If you decide later that you do not want the specimens collected from you to be used for future research, you may tell this to Dr. Morris, who will use his best efforts to stop any additional studies. However, in some cases, such as if the material within your samples are found to be generally useful, it may be difficult or impossible, to stop such future research once the materials have been widely shared with other researchers. Dr. Morris, his associates, or his successors in these studies will keep your DNA specimen or the information derived from it indefinitely.

#### **BENEFITS**

There may or may not be a direct benefit to you from the procedures done as part of this study. However, information learned from this study may help the study doctor/staff learn more about different ways to help high-risk HIV negative reduce their risk of acquiring HIV.

#### **NEW FINDINGS**

You will be told of any new information learned during the course of the study that might cause you to change your mind about staying in the study. At the end of the study, you will be told when study results may be available and how to learn about them.

# REASONS FOR WITHDRAWAL FROM THE STUDY DRUGS AND/OR STUDY WITHOUT YOUR CONSENT:

You may be removed from the study without your consent for the following reasons:

- The study is canceled by the California Collaborative Treatment Group (CCTG) the sponsors, the UCSD AVRC study doctor, or the UCSD Institutional Review Board (IRB). An IRB is a committee that watches over the safety and rights of research subjects;
- You are unable to keep appointments as required by the study, including missing 2 consecutive visits before 48 weeks, 1 visit after 48 weeks or discontinuing study drug at 48 weeks or more
- ◆ You do not start the study treatment.
- ◆ You experience a high level drug toxicity
- You acquire HIV or viral hepatitis.

#### ALTERNATIVES TO PARTICIPATION

You may decide not to take part in this study. The alternatives to participating in this study is to receive counseling on HIV prevention and testing for sexually transmitted infections and HIV infection from your current primary care doctor. The study medication TDF/FTC could be obtained from your doctor.

#### COSTS TO YOU

There is no cost to you for the study-related medications, clinic visits, procedures, examinations, or laboratory tests in this study. The cost of any drugs you may need to treat other medical conditions, and any other medical costs for your treatment outside this study, will be the responsibility of you or your insurance company.

As compensation for your time and any inconvenience you may experience as a result of your participation in this study, you will receive \$10 after you complete your entry and your month 1, 3, 6, 9, 12 and every 3 months study visits. You will not receive compensation for visits that are not completed.

## **CONFIDENTIALITY**

Your research records will be confidential to the extent permitted by law. You will be identified by a code, and personal information from your records will not be released without your written permission. You will not be personally identified in any publication about this study. However, your records may be reviewed, under guidelines of the Federal Privacy Act, by Office for Human Research Protection (OHRP), study monitors, drug companies supplying the study drugs and their designees and the UCSD Institutional Review Board (IRB).

The University has policies and procedures to ensure your confidentiality. We will use our best efforts to ensure that your identity and test results will not become known outside the research program. Please talk with your study staff if you have any concern in this issue.

Because the University of California complies with the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA) and its privacy regulations, and all other applicable laws that protect your privacy, in addition to this informed consent form, you will be asked to read and sign the attached HIPAA Authorization Form prior to your participation in this research study.

The U.S. Department of Health and Human Services (DHHS) has issued a Confidentiality Certificate to this research project to help protect your identity. This certificate means that researchers cannot be forced to release any research data in which you are identified, even under court order or subpoena, without your written consent. If we learn something that would immediately endanger you or others, we may discuss it with you, if possible, or seek help from others to protect you or others. Having a Certificate of Confidentiality does not prevent you from releasing information about yourself and your participation in the study.

Even with the Certificate of Confidentiality, if the study staff learns of possible child abuse and/or neglect or a risk of harm to yourself or others, we will be required to tell the proper authorities.

A Certificate of Confidentiality does not represent an endorsement of the research study by the Department of Health and Human Services or the National Institutes of Health.

## RESEARCH-RELATED INJURY

**PROBLEMS OR QUESTIONS** 

If you are injured as a direct result of participation in this study, the University of California will provide any medical care you need to treat those injuries. Neither the sponsor of the study California Collaborative Treatment Group (CCTG), nor the University of California will provide any compensation to you if you are injured. You may call the UCSD Human Research Protection Program Office at (858) 455-5050 for more information about this, to inquire about your rights as a research subject, or to report research-related problems.

| Dr. [[Morris]] and/or has explained this study to you and answered your questions. If you ever have questions about this research study, or in case of research-related problems, you may reach [[ <b>Dr. Sheldon Morris at (619) 543-8080</b> ]] or an AVRC doctor on call at (619) 543-6737 after working hours or in an emergency. | |
|---|---|
| Participation in this study is entirely voluntary. You me time without jeopardy to the medical care you will receive which you are entitled. | |
| The study purpose, procedures, possible risks and ben<br>explained to you. You have been invited to ask any qu<br>and all your inquiries have been answered. You do<br>signing this form. | estions about the study that you may have, |
| You have received a copy of this document and a co<br>Rights" to keep. | ppy of the "Experimental Subject's Bill of |
| You agree to participate. | |
| Printed Subjects Name | |
| Subjects Signature | Date |
| Witness or Research Team Member Signature | Date |
| Signature of Person Obtaining Consent | Date |

## **16.0 APPENDICES**

# **APPENDIX II: QUESTIONNAIRES**

| Domain | Assay | Header in Survey | Page | # of Q's | Schedule |
|---|---|---|---|---|---|
| HIV Literacy | HIVKQ18 | HIV Knowledge | 2 | 20 | B, 48, EOS |
| Stigma and<br>Disclosure | USC Survey | Stigma and disclosure | 4 | 20 | B, 48, EOS |
| Risk Behavior | Sexual Risk Scale | Attitude to safe sex | 9 | 24 | В |
| Partner<br>Disclosure<br>Provider<br>Education | Milam Survey | Provider Education | 11 | 4 | В |
| | Anatomic Risk | | 12 | 3 | В |
| | Modified State Form | Sexual risk survey | 12 | 13 | All |

| Adherence | ACTG Adherence,<br>modified | PrEP Adherence | 15 | 13 | All except baseline |
|---|---|---|---|---|---|
| | Ira Wilson Adherence<br>Questions | 4 week medication recall | 19 | 5 | All except baseline |
| | Visual Analog Scale | Adherence scale | 20 | 4 | All except baseline |
| Intention to<br>Adhere | VAS Intention | | | | All visits |
| Depression | PHQ9 | Mood scale | 22 | 10 | All |
| Substance Use | AUDIT | Alcohol use | 23 | 10 | B, 48, EOS |
| | DAST-10 | Drug Use | 25 | 10 | B, 48, EOS |
| | SCID Screen | Drug Use | 26 | 16 | All |
| Access to Care | Modified USC | Access to care | 27 | 7 | В |
| Social Support | Modified USC | Social Support | 30 | 6 | В |
| Technology | Text Message Ability | Texting Knowledge | 33 | 8 | В |
| Sexual<br>Compulsivity | Kalichman; Scale 1 | Sexual Desire | 34 | 9 | B, EOS |
| | iTab/PrEP Feedback | | 35 | 15 | 48 |

| iPad Header: HIV Knowledge | Assay: HIVKQ18, BEHKA | # of Questions: 20 | Time: |
|---|---|---|---|

*Instructions*: Please select the most appropriate answer.

1. Coughing and sneezing DO NOT spread HIV or STD.

True False Don't Know

2. A person can get HIV or STD by sharing a glass of water with someone who has an STD or HIV.

True False Don't Know

3. Pulling out the penis before a man climaxes/cums keeps their partner from getting HIV or STD during sex.

True False Don't Know

4. Anyone can get HIV or STD if they have anal sex with a man.

True False Don't Know

5. Showering, or washing one's genitals/private parts, after sex keeps a person from getting HIV.

True False Don't Know

6. All pregnant women infected with HIV quickly show serious signs of being infected.

True False Don't Know

7. People who have been infected with HIV quickly show serious signs of being infected.

True False Don't Know

8. There is a vaccine that can stop adults from getting HIV.

True False Don't Know

9. People are likely to get HIV by deep kissing, putting their tongue in their partner's mouth, if their partner has HIV.

True False Don't Know

10. A woman cannot get HIV if she has sex during her period.

True False Don't Know

11. A condom that can help decrease a chance of getting HIV.

True False Don't Know

12. A natural skin condom works better against HIV than does a latex condom.

True False Don't Know

13. A person will NOT get HIV if she or he is taking antibiotics.

True False Don't Know

14. Having sex with more than one partner can increase a person's chance of being infected with an STD or HIV.

True False Don't Know

15. Taking a test for HIV less than one week after having sex will tell a person if he or she has HIV.

True False Don't Know

16. A person can get HIV or STD by sitting in a hot tub or swimming pool with someone who has HIV.

True False Don't Know

17. A person can get HIV from oral sex.

True False Don't Know

18. Using Vaseline or baby oil with condoms lowers the chance of getting HIV or STDs.

True False Don't Know

19. Is the goal of treatment to make the 'CD4 count" go up or down?

Up Down

20. Is the goal of treatment to make the "viral load" go up or down?

Up Down

| 'D 111 1 61' 1 D' 1 | | " ( O '' 30 | |
|---|---|---|---|
| iPad Header: Stigma and Disclosure | Assay: Bluthenthal | # of Questions: 20 | Time: |

*Instructions*: The next set of questions asks about some of your feelings and opinions about HIV/AIDS. Please indicate how much you agree or disagree with the following statements:

1. People who have HIV or AIDS should be isolated from the rest of society.

1 Strongly disagree

2 Disagree

| | 3 | Neither agree or disagree |
|---|---|---|
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 2. People who have HIV or AIDS should only date other | r HIV po | sitive people. |
| | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 3. People who have HIV or AIDS are not sexually desira | | Ci. L. II |
| | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 4. People who have HIV or AIDS are more sexually pror | _ | |
| 4. Feople with have fire of Albs are more sexually prof | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 5. The promiscuity of people who are gay is the reason | why HI | V/AIDS exists. |
| | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |

## 9 Prefer not to answer

In the next questions, we will ask you personal beliefs about privacy. For each of the following statements, mark the response that best indicates your experience. On the scale, 1 is Disagree Strongly and 7 is Agree Strongly. Please be as honest as possible in your responses.

| 15. I prefer to keep my sexual relationships rather p | rivate. | |
|---|---|---|
| | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 16. I keep careful controls over who knows about m | ıy sexual | relationships with men. |
| | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 17. My sexual behavior is nobody's business. | 4 | C |
| | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | 8 | Do not know |
| | 9 | Prefer not to answer |
| 18. If you are not careful who you ask about their H | | |
| zor ir you are not careful timo you ask about their ri | 1 | Strongly disagree |
| | 2 | Disagree |
| | 3 | Neither agree or disagree |
| | 4 | Agree |
| | 5 | Strongly agree |
| | J | 2 00.1 00.00 |
| | 8 | Do not know |

9

Prefer not to answer

| 19. I think very carefully before asl | king about someone's HIV | status | | | | |
|---|---|---|---|---|---|---|
| 19. I tillik very carefully before asi | ting about someone's riv | Strongly dis | agroo | | | |
| | 2 | Disagree | agicc | | | |
| | | • | | licaaraa | | |
| | 3 | Neither agr | ee or o | iisagree | | |
| | 4 | Agree | | | | |
| | 5 | Strongly ag | ree | | | |
| | 8 | Do not know | N | | | |
| | 9 | Prefer not t | o answ | ver | | |
| 20. My sexual orientation is a very | personal and private mat | ter. | | | | |
| | 1 | Strongly dis | agree | | | |
| | 2 | Disagree | | | | |
| | 3 | Neither agr | ee or d | disagree | | |
| | 4 | Agree | | | | |
| | 5 | Strongly ag | ee | | | |
| | 2 | 5 | | | | |
| | 8 | Do not know | | | | |
| | 9 | Prefer not t | o answ | ver | | |
| <i>iPad Header</i> : <b>Attitude to safe sex</b> | Assay: Sexual Risk Scale | # of ( | Duestio | ons: 24 | Time: | |
| iPaa Header: Attitude to safe sex | Assay: Sexual Risk Scale | # <i>0</i> J C | luestio | ons: 24 | Time: | |
| Instructions: Safer sex means sexual condoms is an example of safer sex to other sexual activity which might following items, please choose the | t. <u>Unsafe</u> , <u>risky</u> , or <u>unprotec</u><br>t increase the risk of AIDS v | cted sex refers<br>virus transmiss | to sex<br>ion. Fo | withou<br>or each c | t a cond | _ |
| | | Strongly<br>Disagree | Disagree | Undecided<br>/neutral | Agree | Strongly<br>Agree |

| _ | | | | | | |
|---|---|---|---|---|---|---|
| 1. | If my partner wanted me to have unprotected sex, I would probably "give in". | 1 | 2 | 3 | 4 | 5 |
| 2. | I may have had sex with someone who was at risk for HIV/AIDS. | 1 | 2 | 3 | 4 | 5 |
| 3. | If I were to have sex, I would take precautions to reduce my risk for HIV/AIDS. | 1 | 2 | 3 | 4 | 5 |
| 4. | I am at risk for HIV/AIDS. | 1 | 2 | 3 | 4 | 5 |
| 5. | I would try and use a condom when I had sex. | 1 | 2 | 3 | 4 | 5 |
| 6. | Condoms interfere with romance. | 1 | 2 | 3 | 4 | 5 |
| 7. | My friends talk a lot about "safer" sex. | 1 | 2 | 3 | 4 | 5 |
| 8. | If my partner wanted me to participate in "risky" sex and I said that we needed to be safer, we would probably end up having "unsafe" sex. | 1 | 2 | 3 | 4 | 5 |
| 9. | Generally, I am in favor of using condoms. | 1 | 2 | 3 | 4 | 5 |
| 10. | If a friend knew I might have sex on a date, he/she would ask if I were carrying a condom. | 1 | 2 | 3 | 4 | 5 |
| | | Strongly<br>Disagree | Disagree | Undecided<br>/neutral | Agree | Strongly<br>Agree |
| 11. | If I had a date, I would probably not drink alcohol or use drugs. | Strongly<br>Disagree | ν Disagree | Undecided<br>w<br>/neutral | A Agree | Strongly<br>Agree |
| 11.<br>12. | · | | | | | |
| | drugs. "Safer sex" reduces the mental pleasure of sex. If I thought that one of my friends had sex on a date, I would | 1 | 2 | 3 | 4 | 5 |
| 12. | "Safer sex" reduces the mental pleasure of sex. | 1 | 2 | 3 | 4 | 5 |
| 12.<br>13. | drugs. "Safer sex" reduces the mental pleasure of sex. If I thought that one of my friends had sex on a date, I would ask them if they used a condom. | 1 1 1 | 2 2 2 | 3 3 | 4 4 | 5<br>5<br>5 |
| 12.<br>13.<br>14. | drugs. "Safer sex" reduces the mental pleasure of sex. If I thought that one of my friends had sex on a date, I would ask them if they used a condom. The idea of using a condom doesn't appeal to me. | 1<br>1<br>1 | 2 2 2 | 3 3 3 | 4 4 4 | 5<br>5<br>5 |
| 12.<br>13.<br>14. | "Safer sex" reduces the mental pleasure of sex. If I thought that one of my friends had sex on a date, I would ask them if they used a condom. The idea of using a condom doesn't appeal to me. "Safer" sex is a habit for me. If my partner wanted me to participate in "risky" sex and I suggested a lower risk alternative, we would have the | 1<br>1<br>1<br>1 | 2 2 2 2 | 3<br>3<br>3<br>3 | 4 4 4 | 5<br>5<br>5<br>5 |
| 12.<br>13.<br>14.<br>15. | drugs. "Safer sex" reduces the mental pleasure of sex. If I thought that one of my friends had sex on a date, I would ask them if they used a condom. The idea of using a condom doesn't appeal to me. "Safer" sex is a habit for me. If my partner wanted me to participate in "risky" sex and I suggested a lower risk alternative, we would have the "safer" sex instead. The sensory aspects (smell, touch, etc.) of condoms make | 1<br>1<br>1<br>1<br>1 | 2<br>2<br>2<br>2<br>2 | 3<br>3<br>3<br>3 | 4 4 4 | 5<br>5<br>5<br>5 |
| 12.<br>13.<br>14.<br>15.<br>16. | "Safer sex" reduces the mental pleasure of sex. If I thought that one of my friends had sex on a date, I would ask them if they used a condom. The idea of using a condom doesn't appeal to me. "Safer" sex is a habit for me. If my partner wanted me to participate in "risky" sex and I suggested a lower risk alternative, we would have the "safer" sex instead. The sensory aspects (smell, touch, etc.) of condoms make them unpleasant. | 1<br>1<br>1<br>1<br>1 | 2<br>2<br>2<br>2<br>2<br>2 | 3<br>3<br>3<br>3 | 4 4 4 4 | 5<br>5<br>5<br>5<br>5 |

| | | Strongly<br>Disagree | Disagree | Undecided<br>/Neutral | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|---|
| 21. | When I socialize, I usually drink alcohol or use drugs. | 1 | 2 | 3 | 4 | 5 |
| 22. | If a sexual partner didn't want to use condoms, we would have sex without using condoms. | 1 | 2 | 3 | 4 | 5 |
| 23. | People can't get the same pleasure from "safer" sex as from unprotected sex. | 1 | 2 | 3 | 4 | 5 |
| 24. | Using condoms interrupts sex play. | 1 | 2 | 3 | 4 | 5 |

| iPad Header: Provider Education | Assay: Milam | # of Questions: 4 | Time: |
|---------------------------------|--------------|-------------------|-------|
|---------------------------------|--------------|-------------------|-------|

1. Thinking about all the visits you made to your health care provider(s) during the past 3 months, how often did you receive any information (got a brochure, saw a poster, spoke with someone) about preventing transmission of HIV infection (choose only one answer)?

0 = every visit

1 = most visits

2 = some visits

3 = none of my visits

7 = Don't Know

8 = Refuse to Answer

| <ol><li>In the last 6 months, how many times have you be<br/>scheduled visits for care that addressed HIV preven</li></ol> | | our hea | alth care provider f | or regular, |
|---|---|---|---|---|
| • | 0 times | : | | |
| | 1 time | , | | |
| | 2 times | | | |
| | 3 times | | | |
| | 4 or mo | | es. | |
| | Don't K | | | |
| | Refuse | | wer | |
| 3. Think about these visits. At how many of these v you using safer sex, such as condoms? | isits did | your o | care provider talk w | ith you about |
| 0 = | 0 visits | | | |
| 1 = | 1 visit | | | |
| 2 = | 2 visits | | | |
| 3 = | 3 visits | | | |
| 4 = | 4 or mo | ore visit | S | |
| 7 = | Don't K | now | | |
| 8 = | Refuse | to Ans | wer | |
| 4. Still thinking about these visits. At how many of to you about asking your sexual partners about their H | | | d your care provide | r talk with |
| 0 = | 0 visits | | | |
| 1 = | 1 visit | | | |
| 2 = | 2 visits | | | |
| 3 = | 3 visits | | | |
| 4 = | 4 or mo | ore visit | S | |
| 7 = | Don't K | (now | | |
| 8 = | Refuse | to Ans | wer | |
| | | | | 1 |
| iPad Header: Anatomic Baseline RIsks Assay: Morris | | | # of Questions: 3 | Time: |
| 1. Is your penis circumcised? | | | | |
| | 0 | No | | |
| | 1 | Yes | | |
| | _ | | | |
| | 8 | Do no | t know | |
| | 9 | Prefe | r not to answer | |
| 2. In the past month how frequently have you perforn | ned rect | al douc | hing or enema (clea | ning out your |
| rectum or colon)? | - 3- | | <b>5</b> - 1,000 | J 1, 1 |
| | 0 | Never | • | |
| | 1 | Karely | / (once or twice) | |

- 2 A few times (less than weekly)
- 3 Fairly regular (about weekly)
- 4 Many times (more than once a week)
- 8 Do not know
- 9 Prefer not to answer
- 3. For rectal douching or enemas in the past month what do you use? (check all that are apply)
  - Nothing in past month
  - 1 Soapy water enema
  - 2 Plain water enema
  - 3 Saline ('Fleet') enema
  - 4 Mineral oil enema
  - 5 Polyethylene glycol oral (e.g. Go-Lytely)
  - 6 Other enema type
  - 7 Other oral colonic cleanser
  - 8 Do not know
  - 9 Prefer not to answer

| iPad Header: Sexual Risk Survey | Assay: Modified State form | # of Questions:13 | Time: |
|---|---|---|---|

*Instructions*: The following questions ask more questions about the specific sexual activities that you have been participated in recently.

- 1. In the past 3 months, did you talk about safer sex with any of your sexual partners?
  - 5 Never
  - 6 Rarely
  - 7 Some of the time
  - 8 Most of the time
  - 9 All of the time
  - 10 Do not know

| | 11 F | Prefer not to answe | r |
|---|---|---|---|
| 2. How many of the sexual partners that you medicine to prevent HIV transmission? | had in the past 1 m | onth knew that yo | u were taking |
| · | 0 1 | lone knew | |
| | 1 9 | Some knew | |
| | 2 A | All knew | |
| | 8 [ | Oo not know | |
| | 9 F | Prefer not to answe | r |
| 3. In the past three month who did you have | sex with? (check al | I that are apply) | |
| | 0 1 | lo sex partners | |
| | 1 N | Men | |
| | 2 V | Vomen | |
| | | Male to female tran | _ |
| | 4 F | emale to male tran | sgender |
| | 8 F | Prefer not to answe | r |
| 4. How many male sexual partners have you h | nad in past 3 mont | <b>hs:</b> (if 0, skip | ) |
| With your male partners in the past 3 months 4a. Have Anal insertive (your penis in them) se How frequently did you use condoms during a past 3 months? | x? (Y/N) (if N, skip) | penis in them) sex | with men in the |
| 1 | | | |
| | 50 | | 100 |
| Never | Half of the time | | All the Time |
| 4b. Anal receptive (their penis in you) condom | use | | |
| 0 | 50 | | <br> <br>100 |
| | 50<br>Half of the time | | 100<br>All the Time |
| | Half of the time | | |
| Never 5. How many transgender sexual partners have the sexual partners | Half of the time ve you had in past in the past 3 months | 3 months: | |
| Never 5. How many transgender sexual partners have | Half of the time ve you had in past in the past 3 months | 3 months: | |
| Never 5. How many transgender sexual partners have the sexual partners | Half of the time ve you had in past in the past 3 months | 3 months: | |



8. We are interested in your condom use if you had anal sex with someone where you did not know their HIV status or that you knew their status was HIV positive.

| | ms (these) partners in the <u>past 3 months</u> v | vhen |
|---|---|---|
| 8a. having Anal insertive (your p | penis in them) sex | |
| I | | |
| 0 | 50 | 100 |
| Never | Half of the time | All the Time |
| 8b. when having anal receptive | (their penis in you) sex | |
| 1 | | |
| 0 | 50 | 100 |
| Never | Half of the time | All the Time |
| | Than or the time | 7 ( |
| 9. Other | | |
| 10. Did you inject drugs? | (yes) (no) | |
| 10a. If you inject, did yo | ou share needles? | |
| | (not applicable) | |
| | (never) | |
| | (sometimes)<br>(usually) | |
| | (always) | |
| | (aiways) | |
| | d you meet a sex partner through any of th | he following ways (check |
| none or all that apply) | - None | |
| | - Internet | |
| | - Mobile applications | |
| | - Bath house | |
| | - Bar | |
| | - Sex Party | |
| | - Other | |
| | - Other | |
| 12. Now we want you to think | about just the last month. How many male | e or transgender sex partners |
| did you have in the past one me | | |
| | now status because you discussed) | <del></del> |
| • | now status because you discussed) | |
| # of HIV unknown (you | did not discuss HIV status) | <del></del> |
| | r of sex acts you have with those partners | that were HIV positive or |
| unknown status: | | |
| # of unprotected anal re | eceptive (their penis in you) acts | |

| of unprotected anal insertive | (your penis in them) acts |
|-------------------------------|---------------------------|
| of unprotected oral sex acts | |

| iPad Header: PrEP Adherence | Assay: ACTG 4-da | y recall # | of Questions: | Time: |
|---|---|---|---|---|

*Instructions*: Most people with HIV have many pills to take at different times during the day. Many people find it hard to always remember pills:

- Some people get busy and forget to take their pills with them.
- Some people find it hard to take their pills according to all the instructions, such as "with food", "on an empty stomach", "every 8 hours", or "with plenty of fluids".
- Some people choose to skip pills to avoid side effects or to just not be taking pills that day.

We need to understand how people on PrEP are really doing with their pills. Please tell us what you are actually doing. Don't worry about telling us that you don't take all your pills. We need to know what is really happening, not what you think we "want to hear."

Complete frequency of drug

| 1. | How many times a day are supposed to take your PrEP medication? |
|----|-----------------------------------------------------------------|

| | 2. | How many pills you supposed to take when you take this drug? | |
|---|---|---|---|
| | | Are you currently taking any of your PrEP medication? | |
| Yes. | ••••• | SKIP TO QUESTION 6 | 1 |
| | | Why are you not taking your PrEP medication? (CIRCLE ALL THAT APPLY) | |
| | | ed to avoid the side effects | 1 |
| | | ving sex2 | |
| | _ | sex but do not think you are at risk | |
| Don | ı't k | believe in these medications | 4 |
| | | Over the last 4 days, have you not been able to take any of your PrEP medication? | |
| | | SKIP TO QUESTION 7 | |
| Yes. | | | 1 |
| | 6. | The next section of the questionnaire asks about the PrEP medication that you have able take taking over the <u>last four days</u> . When were not able to take your medication all that apply) | on (check |
| Yest | tero | day | 1 |
| Day | be | efore yesterday ((2 days ago) | 2 |
| 3 da | ays | ago | 3 |
| 4 da | ays | ago | 4 |
| | 7. | PrEP medication would best be taken at the same time every day. How closely did y | you take |
| | | the medication at about the same time over the last four days? | |
| Nev | er | | 0 |
| | | of the Time | |
| Abo | ut | Half of the Time | 2 |
| | | of the Time | |
| All | of th | he Time | 4 |
| | 8. | Some people find that they forget to take their pills on the weekend days. Were yo | u not able |
| | | to take any of your PrEP medication last weekend—last Saturday and Sunday? | |
| Yes. | ••••• | | 1 |
| | 9. | Including the four days you just described, when was the last time you were not ab your PrEP medication? | le to take |
| Nev | er ı | missed PrEP medication | 0 |
| | | han 3 Months Ago | |
| 1— | 3 M | Nonths Ago | 2 |

| 2—4 Months Ago | 3 |
|----------------------|---|
| 1—2 Weeks Ago | |
| Within the Past Week | |

Instructions: For participant to complete questions 12 and 13.

10. People may miss taking their medications for various reasons. Here is a list of possible reasons why you may miss taking your medications. How often have you missed taking your medications because you:

| | | Never | Rarely | Sometimes | Often |
|---|---|---|---|---|---|
| A. | Were away from home? | 1 | 2 | 3 | 4 |
| В. | Were busy with other things? | 1 | 2 | 3 | 4 |
| C. | Simply forgot? | 1 | 2 | 3 | 4 |
| D. | Had too many pills to take? | 1 | 2 | 3 | 4 |
| E. | Wanted to avoid side effects? | 1 | 2 | 3 | 4 |
| F. | Did not want others to notice you taking medication? | 1 | 2 | 3 | 4 |
| G. | Had a change in daily routine? | 1 | 2 | 3 | 4 |
| Н. | Felt like the drug was toxic/harmful? | 1 | 2 | 3 | 4 |
| I. | Fell asleep/slept through dose time? | 1 | 2 | 3 | 4 |
| J. | Felt sick/ill from side effects? | 1 | 2 | 3 | 4 |
| K. | Felt depressed/overwhelmed? | 1 | 2 | 3 | 4 |
| L. | Had problem taking pills at specified time (with meals, on empty stomach, etc.?) | 1 | 2 | 3 | 4 |
| M. | Lost medications? | 1 | 2 | 3 | 4 |
| N. | Could not obtain medications? | 1 | 2 | 3 | 4 |
| 0. | Did not have sex with a HIV positive person | 1 | 2 | 3 | 4 |
| P. | Did not have sex with anyone unknown status | 1 | 2 | 3 | 4 |
| Q. | Did not have sex with anyone | 1 | 2 | 3 | 4 |

11. In the last 30 days, how good a job did you do at taking Truvada for PrEP in the way you were supposed to?

- o Very poor
- o Poor
- o Fair

| 0 | Good |
|---|-----------|
| 0 | Verv good |

| | , | 0 |
|---|------|-------|
| О | Exce | llent |

| 12. In the last 30 days, how often did you take Truvada for PrEP in the way you were supposed to? | 12. In the | e last 30 days, | how often did | vou take 1 | Truvada for PrEF | in the way | you were sui | posed to? |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

- o Never
- o Rarely
- o Sometimes
- o Usually
- o Almost always
- o Always

# 13. In the last 30 days, how hard was it for you to take Truvada for PrEP in the way you are supposed to?

- o Extremely hard
- o Very hard
- o Somewhat hard
- o Not very hard
- o Not hard at all

| iPad Header: 4 week medication recall | Assay: Ira Wilson | # of Questions: | Time: |
|---|---|---|---|
| " da ricader. 4 week incalcation recan | Assay. II a Wilsoll | # of Questions. | THITC. |

*Instructions*: Please select the most appropriate answer.

- 1. Thinking about the past 4 weeks, on average, how would you rate your ability to take all of your PrEP medication as your doctor prescribed them?
- o Very poor
- o Poor
- o Fair
- o Good
- o Very good
- o Excellent
- 2. Thinking about the past 4 weeks, how often did you take all of your PrEP medication as your doctor prescribed them?
- o None of the time

o A little of the time o A good bit of the time o Most of the time o All of the time 3. Thinking about the past 4 weeks, what percent of the time were you able to take all your PrEP medications as your doctor prescribed them? 0 / 10 / 20 / 30 / 40 / 50 / 60 / 70 / 80 / 90 / 100 4. Place your finger on the bar and slide to the right to indicate your level of adherence over the past 4 weeks. Zero percent means you have taken no antiretroviral medications, 50% means you have taken half of your antiretroviral medications, 100% means you have taken every single dose of your antiretroviral medications during the past 4 weeks. 50 100 0 Half of the time All the Time Never 5. Thinking about the past 7 days, how many Truvada pills did you take? o All of my pills every day o Most of my pills o About one-half of my pills o Very few of my pills o None of my pills iPad Header: Adherence Scale Assay: VAS; Intention # of Questions: Time: Instructions: Please put a mark on the line below indicating what percentage of the time over the past 4 weeks you took your PrEP medication exactly as prescribed on the pill bottle. 100 All the time Never

Alarm/watch 1 Calendar

*Instructions*: Score

| "Post-it" reminder pad | 3 |
|---|---|
| Pill box | |
| iTAB texting reminders | |
| | app.)6 |
| | 7 |
| Other—explain: | 8 |
| | below indicating what percentage of the time over the $\frac{1}{1}$ cation exactly as prescribed on the pill bottle. |
| 1. | |
| 0 | 100 |
| Never | All the time |
| INSTRUCTIONS TO CLINICIAN: Score: | |
| • | below indicating what percentage of the time over the <u>next 4</u> PrEP medication exactly as prescribed on the pill bottle. |
| 1. | |
| 0 | 100 |
| Never | All the time |
| INSTRUCTIONS TO CLINICIAN: Score: | |

| 1 ( <i>)</i> A |
|------------------|

| iPad Header: Mood Scale | Assay: PHQ9 | # of Questions: | Time: |
|-------------------------|-------------|-----------------|-------|

*Instructions*: Over the last 2 weeks how often have you been bothered by any of the following problems?

| | | NOT<br>AT ALL | SEVERAL<br>DAYS | MORE<br>THAN HALF<br>THE DAYS | NEARLY<br>EVERY DAY |
|---|---|---|---|---|---|
| 1. | Little interest or pleasure in doing things | 0 | 1 | 2 | 3 |
| 2. | Feeling down, depressed, or hopeless | 0 | 1 | 2 | 3 |
| 3. | Trouble falling or staying asleep, or sleeping too much | 0 | 1 | 2 | 3 |
| 4. | Feeling tired or having little energy | 0 | 1 | 2 | 3 |
| 5. | Poor appetite or overeating | 0 | 1 | 2 | 3 |
| 6. | Feeling bad about yourself — or that you are a failure or have let yourself or your family down | 0 | 1 | 2 | 3 |
| 7. | Trouble concentrating on things, such as reading the newspaper or watching television | 0 | 1 | 2 | 3 |

| 8. | Moving or speaking so slowly that other people could have noticed? Or the opposite — being so fidgety or restless that you have been moving around a lot more than usual | 0 | 1 | 2 | 3 |
|---|---|---|---|---|---|
| 9. | Thoughts that you would be better off dead or of hurting yourself in some way | 0 | 1 | 2 | 3 |

| | | NOT<br>DIFFICULT<br>AT ALL | SOMEWH<br>AT<br>DIFFICULT | VERY<br>DIFFICULT | EXTREMELY<br>DIFFICULT |
|---|---|---|---|---|---|
| 10. | If you checked off any problems, how difficult have<br>these problems made it for you to do your work, take<br>care of things at home, or get along with other people | 0 | 1 | 2 | 3 |

| iPad Header: Alcohol Use | Assay: AUDIT | # of Questions: | Time: |
|--------------------------|--------------|-----------------|-------|
|--------------------------|--------------|-----------------|-------|

*Instructions*: These are some questions about your use of alcoholic beverages <u>during the past year</u>. By alcoholic beverages we mean beer, wine, or liquor (vodka, whiskey, brandy, etc.).

1. How often do you have a drink containing alcohol?

| Never | 0 |
|---|---|
| Never Monthly or less | 1 |
| 2 to 4 times a month | |
| 2 to 3 times a week | 3 |
| 4 or more times a week | 4 |
| 2. How many drinks of alcohol do you have in a typical day when you are drinking? | |
| 1 or 2 | 0 |
| 1 or 2 | |
| 5 or 6 | 2 |
| 7, 8 or 9 | 3 |
| 10 or more | 4 |
| 3. How often do you have six or more drinks on one occasion? | |
| Never | |
| Less than monthly | 1 |
| Monthly | 2 |
| Weekly | 3 |
| Daily or almost daily | 4 |
|---|---|
| 4. How often during the last year have you found | that you were unable to stop drinking once you |
| had started? | |
| Never | 0 |
| Less than monthly | |
| Monthly | |
| Weekly | |
| Daily or almost daily | |
| 5. How often during the last year have you failed | |
| because of drinking? | to do what was normany expected from you |
| Never | 0 |
| Less than monthly | 1 |
| Monthly | 2 |
| Weekly | 3 |
| Daily or almost daily | 4 |
| 6. How often during the last year have you neede after a heavy drinking session? | d a first drink in the morning to get yourself going |
| Never | 0 |
| Less than monthly | 1 |
| Monthly | 2 |
| Weekly | 3 |
| Daily or almost daily | 4 |
| 7. How often during the last year have you had a | feeling of guilt or remorse after drinking? |
| Never | 0 |
| Less than monthly | |
| Monthly | |
| Weekly | 3 |
| Daily or almost daily | 4 |
| 8. How often during the past year have you been | unable to remember what happened the night |
| before because you had been drinking? | - |
| Never | 0 |
| Less than | |
| monthly | 1 |
| Monthly | |
| Weekly | |
| Daily or almost | |
| daily | Δ |
| 9. Have you or someone else been injured as a re | |
| No | , - |
| Yes, but not in the last year | |
| • | |
| Yes, during the last year | |
| 10. 10. Has a relative, friend, doctor, or other healt suggested you cut down? | in worker been concerned about your drinking or |
| No | Λ |
| Yes, but not in the last year | |
| Yes, during the last year | |
| , 0 1 1 | |

| IPad Hedder: Drug Use | iPad Header: <b>Drug Use</b> | Assay: DAST-10 | # of Questions: | Time: |
|---|---|---|---|---|
|---|---|---|---|---|

*Instructions*: The following questions concern your use of any illicit drug (e.g. methamphetamine, marijuana, non-prescription opiate, cocaine) <u>during the past 12 months</u>. Carefully read each statement and decide if your answer is "Yes" or "No". Then, circle the appropriate response "0" for "No" or "1" for "Yes".

Please answer every question. If you have difficulty with a statement, then choose the response that is mostly right.

| | THESE QUESTIONS REFER TO THE PAST 12 MONTHS | NO | YES |
|---|---|---|---|
| 1. | Have you used drugs other than required for medical reasons? | 0 | 1 |
| 2. | Do you abuse more than one drug at a time? | 0 | 1 |
| 3. | Are you always able to stop using drugs when you want to? | 0 | 1 |
| 4. | Have you had "blackouts" or "flashbacks" as a result of drug use? | 0 | 1 |
| 5. | Do you ever feel bad or guilty about your drug use? | 0 | 1 |
| 6. | Does your spouse/partner (or parents) ever complain about your involvement with drugs? | 0 | 1 |
| 7. | Have you neglected your family because of your use of drugs? | 0 | 1 |
| 8. | Have you engaged in illegal activities in order to obtain drugs? | 0 | 1 |
| 9. | Have you ever experienced withdrawal symptoms (felt sick) when you stopped taking drugs? | 0 | 1 |
| 10. | Have you had medical problems as a result of your drug use (e.g., memory loss, hepatitis, convulsions, bleeding, HIV, etc.)? | 0 | 1 |



| iPad Header: <b>Drug Use</b> | Assay: SCID Screen | | # of Questions: | Time: |
|---|---|---|---|---|
| Instructions: Please select the most appr | opriate answer. | | | |
| 1. Alcohol | | No | Yes <u>≥</u> 5x | Yes <u>&lt;</u> 4x |
| 2. Tobacco (e.g., cigarettes, cigars, chew | , snuff) | No | Yes ≥ 5x | Yes ≤ 4x |
| 3. Marijuana | | No | Yes <u>&gt;</u> 5x | Yes <u>&lt;</u> 4x |
| 4. Cocaine / Crack | | No | Yes <u>&gt;</u> 5x | Yes <u>&lt;</u> 4x |
| 5. Methamphetamine (i.e., crystal meth | , ice glass) | No | Yes <u>&gt;</u> 5x | Yes <u>&lt;</u> 4x |
| 6. Other Stimulants (e.g., amphetamines | s, ritalin) | No | Yes <u>&gt;</u> 5x | Yes <u>&lt;</u> 4x |
| 7. Heroin | | No | Yes <u>&gt;</u> 5x | Yes <u>&lt;</u> 4x |
| 8. Other opioids (e.g., vicodin, oxycontin | ) | No | Yes ≥ 5x | Yes ≤ 4x |
| 9. Sedatives (e.g., rohypnol, GHB, Quaali | udes, etc.) | No | Yes ≥ 5x | Yes ≤ 4x |
| 10. Antianxiety drugs (e.g., valium, Xana | x, ativan) | No | Yes ≥ 5x | Yes ≤ 4x |
| 11. Hallucinogens (e.g., LSD, mushrooms | s, acid, etc.) | No | Yes ≥ 5x | Yes ≤ 4x |
| 12. Dissociative drugs (e.g., PCP, angel d | ust, ketamine) | No | Yes ≥ 5x | Yes ≤ 4x |
| 13. Inhalants (e.g., nitrous oxide, gasolin | e, glue, whippits, etc.) | No | Yes ≥ 5x | Yes ≤ 4x |
| 14. Poppers (e.g., amyl nitrate, butyl nitr | rate) | No | Yes ≥ 5x | Yes ≤ 4x |
| <b>15. Ecstasy</b> (i.e., MDMA, E, X) | | No | Yes <u>&gt;</u> 5x | Yes ≤ 4x |
| 16. Other: | | No | Yes <u>&gt;</u> 5x | Yes <u>&lt;</u> 4x |

| iPad Header: Access to care | Assay: Modified USC | # of Questions: | Time: |
|-----------------------------|---------------------|-----------------|-------|

*Instructions*: Please select the most appropriate answer. 1. When was the last time you went to a doctor? Less than 3 months ago 3—6 months ago 6-12 months ago More than a year ago 2. Has anyone helped you get into medical care? (check all that apply) 1 Nobody 2 Counselor, social worker, case manager, or other lay professional Doctor, nurse, or other health care professional 4 Partner (boyfriend/husband, girlfriend/wife) 5 Family member 6 Friend 0 Don't want to answer **Barriers to Medical Care** 3. Which of the following are barriers that make it difficult for you to make an appointment and see a **doctor?** (check all that apply) a. Don't know how h. My other health problems interfere I don't have transportation c. d. Takes too much time e. I forget f. Other things are more important I don't think it will improve my health g. h. Costs too much I am worried about what other people will think or that they will judge me i. j. I had a bad experience at an HIV clinic k. I don't trust the medical system ١. I prefer alternative treatments

4. If you have any prescription medication which of the following are barriers that make it difficult for you to take any of your MEDICATIONS? (check all that apply)

The clinic is too busy (no appointments available)

Worries about immigration status or deportation

a. Don't take any medications

m.

n.

- b. My other health problems interfere
- c. I don't have transportation
- d. Takes too much time
- e. I forget
- f. Other things are more important
- g. I don't think it will improve my health
- h. Costs too much
- i. I am worried about what other people will think or that they will judge me.
- j. I had a bad experience at an HIV clinic
- k. I don't trust the medical system
- I. I prefer alternative treatments
- m. The pharmacy is too busy
- n. Worries about immigration status or deportation
- o. Don't know how

# 5. Have you experienced any of the following fears or concerns when trying to receive health care? (check all that apply)

- a. Fears that people would find out about HIV risk behavior
- b. Worries that people would find out about your sexual orientation.
- c. Worries that family members or partners would be upset
- d. Worries that family members or partners would be upset
- e. Fears that children would be taken away
- f. Concerns that health care providers would ask uncomfortable questions
- g. Worries that providers would ask about drug abuse
- h. Worries that providers would ask about sexual practices
- i. Worries about being judged by hospital staff

## **Potential Facilitators to Care**

- **6. Which of the following would help you make and keep an appointment with a doctor?** (check all that apply).
  - a. Money, e.g. \$20 at each visit
  - b. Food, e.g. a bag of groceries at each visit
  - c. Long term housing
  - d. Free cell phone service
  - e. Transportation to medical care
  - f. I don't need any incentives
  - g. TEXT message reminders
  - h. Phone call reminders
  - i. Other: \_\_\_\_\_

| 7. Which of the fo | llowing would help you get and take your medications? (check all that apply) |
|---|---|
| a. | Don't take medications |
| b. | Money, e.g. \$20 at each visit |
| C. | Food, e.g. a bag of groceries at each visit |
| d. | Long term housing |
| e. | Free cell phone service |
| f. | Transportation to medical care |
| g. | I don't need any incentives |
| h. | TEXT message reminders |
| i. | Phone call reminders |
| j. | Other: |

*Instructions*: For the next set of questions, please think about the different types of support you may receive. Please indicate how much you agree or disagree with the following statements.

# of Questions:

Time:

1. There is no one I can talk to about the important decisions in my life. (Choose one)

Assay:

*iPad Header*: **Social Support** 

Strongly agree 1 2 Agree somewhat 3 Disagree somewhat 4 Strongly disagree 8 Prefer Not to Answer 2. I feel no one respects who I am. (Choose one) 1 Strongly agree 2 Agree somewhat 3 Disagree somewhat 4 Strongly disagree 8 Prefer Not to Answer 3. No one really understands my most private worries and fears. (Choose one) Strongly agree 1 2 Agree somewhat 3 Disagree somewhat 4 Strongly disagree 8 Prefer Not to Answer 4. There is no one I can depend on to lend me \$50 if I needed it for an emergency. (Choose one) 1 Strongly agree 2 Agree somewhat 3 Disagree somewhat 4 Strongly disagree 8 Prefer Not to Answer **5. I often feel isolated and alone.** (Choose one) 1 Strongly agree 2 Agree somewhat 3 Disagree somewhat 4 Strongly disagree 8 Prefer Not to Answer Cell Phone Questions at baseline 1. Do you have a cell phone? a. Yes b. No 2. Does your cell phone have the ability to send/receive text message? a. Yes b. No c. Not sure 2a. If yes, do you send text messages? a. Yes b. No ii. About how often?

| a. Hourly |
|---|
| b. Daily |
| c. Weekly |
| d. Monthly |
| e. Less than monthly |
| 2b. If yes, do you receive text messages? |
| a. Yes |
| b. No |
| ii. About how often? |
| a. Hourly |
| b. Daily |
| c. Weekly |
| d. Monthly |
| e. Less than monthly |
| 3. Does your cell phone have the ability to send/receive instant messages? (ex. Yahoo messenger, MSN messenger, or Google chat) |
| a. Yes |
| b. No |
| c. Not sure |
| 3a. If yes, do you send instant messages? |
| a. Yes |
| b. No |
| ii. About how often? |
| a. Hourly |
| b. Daily |
| c. Weekly |
| d. Monthly |
| e. Less than monthly |
| 3b. If yes, do you receive instant messages? |
| a. Yes |
| b. No |
| ii. About how often? |
| a. Hourly |
| b. Daily |
| c. Weekly |
| d. Monthly |
| e. Less than monthly |
| 4. Can your cell phone run applications (apps)? |
| a. Yes |
| b. No |
| c. Not sure |
| 4a. If yes, do you use them? |
| a. Yes |

| b. No |
|-------|

## 5. Can your cell phone access the internet?

- a. Yes
- b. No
- c. Not sure

## 5a. If yes, do you ever browse the internet or use search engines on your phone?

- a. Yes
- b. No

# 6. Does your cell phone have the ability to send/receive email?

- a. Yes
- b. No
- c. Not sure

## 6a. If yes, do you send emails on your phone?

- a. Yes
- b. No

## 6b. If yes, do you receive emails on your phone?

- a. Yes
- b. No

# 7. How long have you had the same cell phone number?

- a. 0-3 months
- b. 3-6 months
- c. 6 months 1 year
- d. 1-5 years
- e. More than 5 years

## 8. Has your cell phone service been disconnected in the last 6 months?

- a. Yes
- b. No

| iPad Header: Sexual Desire | Assay: Kalichman | # of ( | Questic | ns: | Time: | |
|---|---|---|---|---|---|---|
| | | | Ⅎ | Þ | щ | Ŧ |
| | | | T AI | SOMEWHA<br>LIKE ME | , | MUC |
| | | | T A<br>IKE | ME. | ΉE<br>Σ | VERY N |
| | | | ž | SO | Ö | VE<br>L |
| 1. I like wild "uninhibited" sexu | al encounters. | | 1 | 2 | 3 | 4 |

| 2. | The physical sensations are the most important thing about having sex. | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|
| 3. | I enjoy the sensations of intercourse without a condom. | 1 | 2 | 3 | 4 |
| 4. | My sexual partners probably think I am a "risk taker". | 1 | 2 | 3 | 4 |
| 5. | When it comes to sex, physical attraction is more important to me than how well I know the person. | 1 | 2 | 3 | 4 |
| 6. | I enjoy the company of "sensual" people. | 1 | 2 | 3 | 4 |
| 7. | I enjoy watching "X-rated" videos. | 1 | 2 | 3 | 4 |
| 8. | I have said things that were not exactly true to get a person to have sex with me. | 1 | 2 | 3 | 4 |
| 9. | I am interested in trying out new sexual experiences and sensations. | 1 | 2 | 3 | 4 |

| iPad Header: | Assay: iTAB PrEP Feedback | # of Questions: | Time: |
|--------------|---------------------------|-----------------|-------|
| | ,, | 0, 0000.0 | |

Scale #1-3

- (1) Extremely unsatisfied
- (2) Somewhat unsatisfied
- (3) Neither unsatisfied nor satisfied
- (4) Somewhat satisfied

| (5) Extremely satisfied |
|---|
| <ol> <li>How would you rate your overall satisfaction of participating in this study?</li> <li>How satisfied were you with the medication education that you received at your first study visit?</li> <li>Overall, how satisfied were you with the text messaging intervention?</li> </ol> |
| Scale #4-11 |
| (1) Not helpful |
| (2) A little helpful |
| (3) Somewhat helpful |
| (4) Very helpful |
| (5) Extremely helpful |
| <ul> <li>4. How helpful was participating in this study?</li> <li>5. How helpful was the medication education that you received at your first study visit?</li> <li>6. How helpful was the overall text messaging intervention for your medication adherence?</li> <li>7. How helpful were the text messages that reminded you to take your medications?</li> <li>8. How helpful were the text messages that praised you for taking your medications?</li> <li>9. How helpful were the text messages that asked you why you missed a medication dose?</li> <li>10. How helpful were the text messages that told you how adherent you were in the past week?</li> <li>11. How helpful were the text messages that told you how adherent you would be when you took your next dose?</li> </ul> |
| Scale #12-13 |
| (1) Not at all |
| (2) A little bit |
| (3) Moderately |
| (4) Quite a bit |
| (5) Very much |
| 12. Overall, this experience was pleasant. |
| 13. A text messaging intervention could be helpful to me in the future. |
| Scale #14-15 |
| (1) Strongly disagree |

- (2) Disagree
- (3) Neither disagree nor agree
- (4) Agree
- (5) Strongly agree
- 14. I would use a test messaging intervention like this again.
- 15. I would opt to continue receiving the text message intervention if offered.
- **16.** Place your finger on the bar and slide to the right to indicate how effective you think PrEP is in preventing HIV. Zero percent means PrEP will not prevent HIV infection and 100% means PrEP will always prevent HIV infection.



## **16.0 APPENDICES**

## **APPENDIX III: VITAMIN D SUB-STUDY PROTOCOL**

Effect of Vitamin D Supplementation on Bone Turnover Markers during Tenofovir-Emtricitibine Pre-Exposure Prophylaxis in Men Who Have Sex with Men

A Sub-study of CCTG 595

**California Collaborative Treatment Group (CCTG)** 

Protocol Chair: Michael P. Dube, MD

**USC Keck School of Medicine** 

Investigators: Turner Overton, MD

University of Alabama, Birmingham

Kathleen Mulligan, PhD

**UC San Francisco** 

Deepa D. Nanayakkara, MD, MS USC Keck School of Medicine

Sheldon Morris, MD

**UC San Diego** 

Katya Calvo Corado, MD

**Harbor-UCLA Medical Center** 

Biostatistician: Sonia Jain, PhD

**UC San Diego** 

Substudy Version 1.0 3 September 2014

# **CONTENTS**

| | Page |
|------------------------------------------|-------|
| GLOSSARY OF TERMS | pg 3 |
| SCHEMA | pg 5 |
| 1.0 STUDY OBJECTIVES AND HYPOTHESES | pg 11 |
| 2.0 INTRODUCTION | pg 12 |
| 3.0 STUDY DESIGN | pg 15 |
| 4.0 SELECTION AND ENROLLMENT OF SUBJECTS | pg 17 |
| 5.0 STUDY TREATMENT | pg 19 |
| 6.0 CLINICAL AND LABORATORY EVALUATION | pg 22 |
| 7.0 CLINICAL MANAGEMENT | pg 30 |
| 8.0 CRITERIA FOR DISCONTINUATION | pg 33 |
| 9.0 STATISTICAL CONSIDERATIONS | pg 34 |

# SITES PARTICIPATING IN THE STUDY

University of California at San Diego (UCSD) University of Southern California (USC) Harbor-University of California at Los Angeles (UCLA) Medical Center

**GLOSSARY OF TERMS** 

AE adverse event

AIDS acquired immune deficiency syndrome

ART antiretroviral therapy or treatment

ARV antiretroviral or antiretroviral drug

BMD bone mineral density

BTM bone turnover marker

CCTG California Collaborative Treatment Group

CDC Centers for Disease Control and Prevention

CrCl creatinine clearance

CRF case report form

CTX C-terminal telopeptide or carboxy-terminal collagen crosslinks

(a marker of bone resorption)

CVD cardiovascular disease

DAERS DAIDS Adverse Event Reporting System

DHHS Department of Health and Human Services (US)

EAE expedited adverse event

EC ethics committee

FDA Food and Drug Administration (US)

FTC emtricitabine

HAART highly active antiretroviral therapy

HIV human immunodeficiency virus

IRB institutional review board

ITT intent to treat

IU international unit

LFT liver function tests

MI myocardial infarction

MVI multivitamin

NHANES National Health and Nutrition Examination Survey

NIH National Institutes of Health

P1NP total procollagen type 1 N-terminal propeptide (a marker of

bone formation)

PEP post-exposure prophylaxis

PrEP pre-exposure prophylaxis

PTH parathyroid hormone

QD once daily

SAE serious adverse event

SID study identification number

SOE schedule of events

SOP standard operating procedure

TDF tenofovir disoproxil fumarate (Viread)

ULN upper limit of normal

WBC white blood cell count

WHO World Health Organization

#### SCHEMA

## CCTG 595 Vitamin D Sub-study

## Effect of Vitamin D Supplementation on Bone Turnover Markers during Tenofovir-Emtricitibine Pre-Exposure Prophylaxis in Men Who have Sex with Men

| <u>DESIGN</u> | CCTG 595 is an open-label clinical trial of the effect of text messaging |
|---|---|
| | intervention vs. standard of care on adherence to Truvada (tenofovir- |
| | emtricitibine) as PrEP in MSM at increased risk of HIV infection. |

This sub-study is a matched case-control study, in which cases prospectively take vitamin D3 4000 IU/day beginning at week 24 of PrEP.

DURATION Subjects will be followed for 6 months (24 weeks)

SAMPLE SIZE 50 eligible subjects will receive vitamin D and will be compared to 50

matched control subjects from CCTG 595 who are not participating in this

sub-study.

POPULATION HIV-negative men aged ≥18 years initiating CCTG 595, who are not taking

bisphosphonates and do not have a history of osteoporosis, fragility

fracture, or kidney stones, or use of tenofovir prior to entry into CCTG 595

REGIMEN Vitamin D3 4000 IU/day from week 24 through 48 of PrEP with Truvada

ENDPOINTS Primary endpoint will be changes in bone turnover markers from week 24

through week 48 in the vitamin D intervention group as compared to age-

and BMI-matched controls

ANALYSIS A sample size of 44 subjects per group will provide 80% power to detect a

20% change in P1NP means from week 24 through week 48 between matched cases and controls using a paired t-test with a two-sided  $\alpha$  = 0.05. To account for attrition, a sample size of 100 is proposed, including 50

vitamin D treated cases and 50 matched controls from CCTG 595.

## 1.0 HYPOTHESIS AND STUDY OBJECTIVES

## 1.1 Hypothesis

Supplementation with vitamin D 4000 IU/day will significantly blunt the increases in BTMs that occur after initiation of PrEP with Truvada.

## 1.2 Primary Objective

To compare the change in P1NP levels from week 24 through week 48 among subjects (cases) who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls.

## 1.3 Secondary Objectives

- 1.3.1 To compare the change in CTX levels from week 24 through week 48 among subjects who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls.
- 1.3.2 To compare the change in PTH level from week 24 through week 48 among subjects who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls.
- 1.3.3 To compare vitamin D levels at week 48 among subjects who receive vitamin D 4000 IU/day and matched unsupplemented controls.
- 1.3.4 To demonstrate the change in P1NP, CTX, PTH, and vitamin D levels from baseline to week 24 in both cases and controls.

## 2.0 INTRODUCTION

## 2.1 Background and Rationale

Current HIV treatment guidelines recommend combination antiretroviral therapy with three active ARVs and 7 of the 9 currently recommended initial combination regimens for ART-naïve patients include tenofovir disoproxil fumarate (TDF) 1. While treatment with TDF-containing antiretroviral treatment (ART) regimens have proven durable, tolerable, and effective. TDF has well described toxicities, including greater loss of bone mineral density (BMD) in the first 48 weeks after ART initiation and an increased risk for fragility fracture <sup>2-4</sup>. The FDA recently approved TDF given with emtricitabine (FTC) as a single daily fixed dose combination (FDC) pill (Truvada (TDF/FTC)) for Pre-Exposure Prophylaxis (PrEP) to prevent HIV acquisition for persons with increased risk for HIV infection. In studies evaluating the efficacy of TDF/FTC for PrEP, daily use has been shown to significantly reduce BMD <sup>5,6</sup> albeit to a lesser extent than that seen during initial treatment for HIV. Although TDF-containing PrEP has not yet been associated with increased fracture risk, reduced BMD is nonetheless a concern for patients and providers of PrEP. Thus, strategies are needed to attenuate or prevent BMD loss. particularly when TDF-containing PrEP will be given for prolonged periods of time. The mechanism by which TDF induces BMD loss is unclear but appears to be mediated

through a reduction in PTH levels and PTH-controlled calcium and phosphate metabolism <sup>7</sup>. Additional data from ATN 063 suggest that TDF induces a state of functional vitamin D deficiency <sup>8</sup>

Recently, Overton and colleagues reported a dramatic reduction in the magnitude of BMD loss during initial therapy of HIV infection with vitamin D (4000 IU/day) and calcium supplementation <sup>9</sup> when co-administered with efavirenz/TDF/FTC ART. The amount of BMD loss at the hip measured by DXA over 48 weeks with vitamin D-calcium was approximately half that seen with placebo (-1.5% vs. -3.2%, respectively, p< 0.001), and was reduced to levels that would be expected with ART that does not contain TDF. Notably, the median daily vitamin D intake was low for the cohort (120 IU/day) while calcium intake approached recommended daily intake (810mg). Thus, these data provide a strong rationale to study prophylactic administration of daily oral supplemental vitamin D in subjects receiving PrEP with Truvada.

In ACTG 5280, vitamin D-calcium supplementation prevented the increase in parathyroid hormone (PTH) and blunted the increase in bone turnover markers (BTMs), including P1NP (a marker of bone formation) and CTX (a marker of bone resorption). Importantly, there was a good correlation between changes in DXA-measured BMD over time and changes in BTMs, particularly with P1NP. The percentage change of P1NP at week 48 correlated with the percentage change in total hip BMD (r=-0.32, p=0.01) as well as the change in lumbar spine BMD (r=-0.37, p=0.002) [Overton ET, unpublished data]. Due to the difficulties and expense of performing DXA scans in a clinical trial, P1NP levels are proposed as the primary outcome measure for this pilot trial.

CCTG 595 is an open-label clinical trial of the effect of a text messaging intervention vs. standard of care on adherence to Truvada as PrEP in MSM at increased risk for HIV infection (ClinicalTrials.gov Identifier: NCT01761643). Approximately 1/3 of the planned 400 subjects have been enrolled as of April 2014. Study sites include University of California at San Diego, University of Southern California, and Harbor-UCLA Medical Center.

Rationale for use of vitamin D dose: The dose of vitamin D (4000 IU/day) in this protocol carries little risk for the study subjects. This dose was without adverse effects in a more ill population, namely the HIV-infected subjects in ACTG 5280 (see above). Generally, vitamin D supplementation is well tolerated and safe. Dosages up to 10,000 IU daily in healthy adults is considered safe and the current upper U.S. Dietary Reference Intake of 2,000 IU daily is considered to be well below the actual physiologic requirements <sup>10,11</sup>. The Institutes of Medicine guideline considers 4000 IU/day to be the safe upper limits for daily intake for adults <a href="http://www.iom.edu/Reports/2010/dietary-reference-intakes-for-calcium-and-vitamin-D/DRI-values.aspx">http://www.iom.edu/Reports/2010/dietary-reference-intakes-for-calcium-and-vitamin-D/DRI-values.aspx</a>. Several studies have focused specifically on the safety of chronic daily administration of 4000 IU <sup>12-14</sup>. In these studies, 228 adult subjects received 4000 IU/day vitamin D with excellent tolerability, no toxicity, and a concomitant increase in 25 (OH) vitamin D levels ranging from 39-51 ng/mL. No abnormalities in serum calcium or urinary calcium excretion were noted.

In this study supplemental calcium will not be used because: a) in ACTG 5280, calcium intake among untreated HIV-infected subjects was generally adequate <sup>9</sup>. It can be anticipated that the largely healthy HIV-uninfected subjects in CCTG 595 will have levels of intake that are higher than the diseased population in ACTG 5280. This suggests supplemental calcium will not be required for 4000 IU/d vitamin D's beneficial effects,

particularly in the CCTG 595 subjects; b) there is concern that multiple additional pills a day may influence adherence with the primary intervention used in CCTG 595.

#### 3.0 STUDY DESIGN

CCTG 595 is an open-label clinical trial of the effect of a text messaging intervention vs. standard of care on adherence to Truvada as PrEP in MSM at increased risk for HIV infection (ClinicalTrials.gov Identifier: NCT01761643). Eligible subjects for this matched case control substudy will receive vitamin D 4000 IU/day for 24 weeks, from week 24 through week 48. In CCTG 595, plasma from participants are being collected and stored at entry and every 12 weeks. These plasma samples will be used to measure P1NP, CTX, PTH, and vitamin D levels in both cases and controls at entry, week 24, and week 48.

#### 4.0 SELECTION AND ENROLLMENT OF SUBJECTS

#### 4.1 Inclusion Criteria

4.1.1 All subjects must meet CCTG 595 inclusion criteria.

#### 4.2 Exclusion Criteria

- 4.2.1 All subjects must meet CCTG 595 exclusion criteria.
- 4.2.2 Current or prior use of bisphosphonate therapy.
- 4.2.3 Current use of vitamin D supplements greater than 400 IU/day.
- 4.2.4 Current use of androgenic hormones or growth hormones.
- 4.2.5 History of nephrolithiasis (kidney stones).
- 4.2.6 History of fragility fracture.
- 4.2.7 No use of tenofovir prior to entry into CCTG 595

## 4.3 Study Enrollment Procedures

Once a candidate for study entry has been identified, details will be carefully discussed with the subject. The subject will be asked to read and sign the approved protocol consent form. Participation in this substudy is not required for continued participation in CCTG 595.

#### 5.0 STUDY TREATMENT

## 5.1 Study Product Formulation and Preparation

Vitamin D capsules will be supplied as 2000 IU capsules and will be taken as two capsules once daily. Store at 15°-30°C (59°-86°F). Do not expose to excessive heat or moisture.

#### 5.2 Concomitant Medications

All concomitant medications will be recorded on existing CRFs for CCTG 595, with particular attention to vitamin D content of dietary supplements. Use of >400 IU of vitamin D3 in any dietary supplement (such as a multivitamin) will be prohibited.

#### 6.0 CLINICAL AND LABORATORY EVALUATIONS

These will be performed as per the main study. All assays on subjects and controls will be performed on stored samples already being collected by the main study.

The only additional evaluation that will be performed will be calculating the average daily dietary intake of vitamin D and calcium from food. The participants will be asked to recall food items eaten over the last 3 days at the week 36 visit, and the calculator used in the ACTG 5280 study, which is adopted from the USDA database, will be used to quantify vitamin D and calcium intake.

## 7.0 CLINICAL MANAGEMENT

Instructions are provided only for toxicities related to study therapy (vitamin D). The grading system for drug toxicities is located in the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), located at the Division of AIDS Regulatory Support Center Web Site: <a href="http://RSC.tech-res.com/safetyandpharmacovigilance.">http://RSC.tech-res.com/safetyandpharmacovigilance.</a>

For toxicities attributed to vitamin D, investigators may discontinue therapy.

## 7.1 Toxicity

The general guidelines presented below apply to toxicities that are not specifically addressed in section 7.2.

## Grade 1 or 2

Subjects who develop a Grade 1 or 2 AE or toxicity may continue vitamin D without alteration of the dosage. For subjects experiencing Grade 1 or 2 AEs who choose to discontinue vitamin D, the site investigator should contact the protocol chair, and encourage the subject to complete other aspects of CCTG 595.

NOTE: If subjects discontinue study therapies due to experiencing Grade 1 or 2 AEs, this should be noted in the CRF as the reason for discontinuation.

#### Grade 3

If the investigator has evidence that the AE was NOT caused by vitamin D, dosing may continue. Subjects who develop a Grade 3 AE or toxicity thought to be related to vitamin D, should have vitamin D withheld. The subject should be reevaluated weekly until the AE returns to Grade ≤2 or baseline, at which time the study therapies may be reintroduced, at the discretion of the site investigator or according to standard practice.

If the same Grade 3 AE recurs within 4 weeks of restarting treatment, vitamin D must be permanently discontinued. However, if the same Grade 3 AE recurs after 4 weeks, the management scheme outlined above may be repeated.

Subjects experiencing a Grade 3 AE requiring permanent discontinuation of vitamin D should be followed weekly until resolution of the AE and should be encouraged to complete the follow-up protocol study evaluations.

#### Grade 4

Subjects who develop a Grade 4 symptomatic AE or toxicity will have vitamin D permanently discontinued. Subjects experiencing a Grade 4 AE requiring permanent discontinuation of vitamin D should be followed weekly until resolution of the AE and encouraged to complete the follow-up protocol study evaluations.

## 7.2 Specific Management

## 7.2.1 Kidney Stones

Subjects who develop signs and symptoms consistent with urinary tract obstruction should have further evaluation. Subjects with evidence of a new kidney stone on study will be taken off vitamin D but continue to be followed on study.

#### 8.0 CRITERIA FOR DISCONTINUATION

## 8.1 Permanent Treatment Discontinuation

- Drug-related toxicity
- Requirement for prohibited concomitant medications
- Subject develops a kidney stone (see section 7.3.1).
- Completion of treatment as defined in the protocol.
- Reguest by subject to discontinue treatment.
- Discontinuation of PrEP for any reason
- Clinical reasons believed serious by the physician, even if not addressed in the toxicity section of the protocol.

## 9.0 STATISTICAL CONSIDERATIONS

## 9.1 Sample size justification

In ACTG 5280, administration of vitamin D-calcium resulted in a significant reduction in

the magnitude of the rise in BTMs P1NP and CTX 9. Because of more consistent association with changes in BMD with P1NP, this will be used as the primary surrogate marker to reflect bone health. Data on TDF effects on P1NP levels in the absence of HIV infection (e.g. during PrEP) are not available. In A5280, at week 24 P1NP increased by 60% with placebo and 36% with vitamin D-calcium (p<0.001). If we anticipate that supplementation with vitamin D results in a decrease of similar magnitude from week 24 to week 48, then the expected intervention effect size is in the range of 24%. The SD of the change in P1NP at month 6 for the vitamin D-calcium group was 63%, but it is anticipated that the variability of P1NP levels in this study will be much less than that in HIV infected subjects undergoing a variety of pro- and anti-inflammatory changes after initiation of ART as in A5280. If we anticipate that in the absence of vitamin D supplementation that P1NP will increase by 20% and those receiving vitamin D will experience a reduction of this amount at week 48, then with an SD of the change in P1NP of 40%, a sample size of 44 cases and 44 controls will provide 80% power to detect a significant difference in the change in P1NP from week 24 to week 48 between cases and controls using a paired t-test with a two-sided α=0.05. In order to account for attrition, a sample size of 100 is proposed, consisting of 50 vitamin D treated cases and 50 matched controls.

## 9.2 Analyses

All analyses are ITT, unless specified otherwise. Evaluable subjects will be individuals who agree to participate in the vitamin D substudy. The primary endpoint analysis will use a paired t-test to compare the changes in P1NP levels from week 24 to 48 weeks between cases and matched controls. Secondary endpoint analyses will include comparison of changes in 25-OH vitamin D levels, PTH, and CTX and will be analyzed analogously to the primary endpoint. If parametric assumptions fail, the corresponding non-parametric test will be applied, in this case, the Wilcoxon signed rank test. Sensitivity analyses will include linear regression models that adjust for possible confounding covariates, such as dietary intake.

<u>Matching</u>: Concurrent controls who are not enrolled in the vitamin D substudy who are reporting supplementation with  $\leq$  400 IU of vitamin D/day will be matched 1:1 by randomization arm in the CCTG 595 main study (text messaging arm vs. standard of care), age ( $\pm$  5 years), race/ethnicity, season of study entry, and BMI ( $\pm$  3 kg/m<sup>2</sup>).

#### **REFERENCES**

- 1. DHHS Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. 2014; <a href="http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL.pdf">http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL.pdf</a>. Accessed May 1, 2014.
- 2. Bedimo R, Maalouf NM, Zhang S, Drechsler H, Tebas P. Osteoporotic fracture risk associated with cumulative exposure to tenofovir and other antiretroviral agents. *AIDS*. Apr 24 2012;26(7):825-831.
- 3. Gallant JE, DeJesus E, Arribas JR, et al. Tenofovir DF, emtricitabine, and efavirenz vs. zidovudine, lamivudine, and efavirenz for HIV. *New England Journal of Medicine*. Jan 19 2006;354(3):251-260.
- 4. McComsey GA, Kitch D, Daar ES, et al. Bone mineral density and fractures in antiretroviral-naive persons randomized to receive abacavir-lamivudine or tenofovir disoproxil fumarate-emtricitabine along with efavirenz or atazanavir-ritonavir: Aids Clinical Trials Group A5224s, a substudy of ACTG A5202. *J Infect Dis.* Jun 15 2011;203(12):1791-1801.
- 5. Liu AY, Vittinghoff E, Sellmeyer DE, et al. Bone mineral density in HIV-negative men participating in a tenofovir pre-exposure prophylaxis randomized clinical trial in San Francisco. *PLoS ONE [Electronic Resource]*. 2011;6(8):e23688.
- 6. Mulligan K, Glidden DV, Gonzales P, et al. Effects of emtricitabine/tenofovir on bone mineral density in seronegative men from 4 continents: DEXA results of the global iPrex study. *18th CROI*. Boston, MA2011:Abstract 94LB.
- 7. Havens PL, Stephensen CB, Hazra R, et al. Vitamin D3 decreases parathyroid hormone in HIV-infected youth being treated with tenofovir: a randomized, placebo-controlled trial. *Clinical Infectious Diseases*. Apr 2012;54(7):1013-1025.
- 8. Havens PL, Kiser JJ, Stephensen CB, et al. Association of higher plasma vitamin d binding protein and lower free calcitriol levels with tenofovir disoproxil fumarate use and plasma and intracellular tenofovir pharmacokinetics: cause of a functional vitamin D deficiency? *Antimicrobial Agents & Chemotherapy*. Nov 2013;57(11):5619-5628.
- 9. Overton ET, Chan ES, Brown TT, et al. High-Dose Vitamin D and Calcium Attenuates Bone Loss With ART Initiation: Results From ACTG A5280. Paper presented at: Conference on Retroviruses and Opportunistic Infections; March 2014, 2014; Boston, MA.
- 10. Vieth R, Bischoff-Ferrari H, Boucher BJ, et al. The urgent need to recommend an intake of vitamin D that is effective. *American Journal of Clinical Nutrition*. Mar 2007;85(3):649-650.
- 11. Mitka M. More evidence on low vitamin D levels fuels push to revise recommended intake. *JAMA*. Dec 16 2009;302(23):2527-2528.
- 12. Vieth R, Chan PC, MacFarlane GD. Efficacy and safety of vitamin D3 intake exceeding the lowest observed adverse effect level. *American Journal of Clinical Nutrition*. Feb 2001;73(2):288-294.
- 13. Vieth R, Kimball S, Hu A, Walfish PG. Randomized comparison of the effects of the vitamin D3 adequate intake versus 100 mcg (4000 IU) per day on biochemical responses and the wellbeing of patients. *Nutr J.* 2004;3:8-18.

| 14. | Hollis BW, Wagner CL. Vitamin D requirements during lactation: high-dose maternal supplementation as therapy to prevent hypovitaminosis D for both the mother and the nursing infant. <i>American Journal of Clinical Nutrition</i> . Dec 2004;80(6 Suppl):1752S-1758S. |
|---|---|
| | 16.0 APPENDICES |

#### APPENDIX IV: VITAMIN D SUB-STUDY SAMPLE OF INFORMED CONSENT

# CALIFORNIA COLLABORATIVE TREATMENT GROUP (CCTG)

## SAMPLE INFORMED CONSENT

## Study Title

CCTG 595 Substudy: Effect of Vitamin D Supplementation on Bone Turnover Markers during Tenofovir-Emtricitibine Pre-Exposure Prophylaxis in Men Who Have Sex with Men

## INTRODUCTION

You are being asked to take part in this research study because you are HIV-negative and are sexually active with men and are at ongoing risk for acquiring HIV. You are taking a medication (tenofovir-emtricitibine, also known as Truvada), to reduce risk of HIV infection but which may affect your bone health.

This study is sponsored by the California HIV Research Program and receives additional funding from Gilead Sciences, the makers of Truvada. The doctor in charge of this study at this site is: (insert name of Principal Investigator). Before you decide if you want to be a part of this study, we want you to know about the study.

This is a consent form. It gives you information about this study. The study staff will talk with you about this information. You are free to ask questions about this study at any time. If you agree to take part in this study, you will be asked to sign this consent form. You will get a copy to keep.

## WHY IS THIS STUDY BEING DONE?

The purpose of this study is to see if taking vitamin D will help prevent the bone loss that sometimes happens when people are taking PrEP with Truvada. The risks seen with this vitamin D treatment are the same that you would encounter when taking this dose of this vitamin outside of the study.

Vitamin D, which is a nutritional supplement important for bone health, will be provided by the study.

# WHAT DO I HAVE TO DO IF I AM IN THIS STUDY?

## Screening and Entry

If you would like to be in this sub-study, you will already be participating in CCTG 595

when you are asked to participate in this substudy after you have been taking Truvada for 24 weeks. Specifically for this study:

- You will be asked questions about your medical history and any medications and vitamin/mineral supplements you are taking or have taken within the last 30 days.
- You will be asked questions about your dietary intake.
- Blood already being drawn as part of the main study will be used to measure the amount of vitamin D as well markers of bone formation and breakdown (P1NP, CTX, and PTH) in your blood. The results of these tests will not be available until after the end of the study.

# If you do not enroll into the study:

If you decide not to take part in this study or if you do not meet the eligibility requirements, this will not affect your participation in the main CCTG 595 study.

## Study Visits

No additional study visits are required by this sub-study. Bottles of vitamin D at a dose of 4000 units per day (supplied as two 2000 unit capsules) will be dispensed to you at your regular week 24 visit and your week 36 visit. You will be asked to bring your bottles of study medications with you to each of your regular visits.

# If You Have to Stop Taking Vitamin D Early or You Have to Stop the Study Early

If you stop taking vitamin D or leave the vitamin D sub-study early due to side effects, you may be asked to come to the clinic for an additional study visit.

- You will have a brief physical exam.
- You will be asked about your health and any changes in your medicines since your last visit.

## HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

About 50 people will take part in this study.

## HOW LONG WILL I BE IN THIS STUDY?

You will be in this sub-study for about 24 weeks (about 6 months). This will be from your regular week 24 visit until your regular week 48 visit. After completion of this sub-study, you will continue with the main study.

## WHY WOULD THE DOCTOR TAKE ME OFF THIS STUDY EARLY?

The study doctor may need to take you off the study early without your permission if:

- You are not able to attend the study visits as required by the study.
- The study is stopped or canceled.
- You are not able to take vitamin D as required by the study.
- Your primary care physician no longer thinks that participating in the study is in your best interest.

The study doctor may also need to take you off vitamin D without your permission if:

- Continuing vitamin D may be harmful to you.
- You need a treatment that you may not take while on the study.
- You develop a fragility fracture. (A fragility fracture is a fracture that occurs after any fall from a standing height or less. Our bodies should be able to sustain a fall from this height, without a fracture, unless there is some underlying cause like osteoporosis. The spine, wrist, and hip are the most common sites for fragility fractures.)
- You develop a kidney stone.

If you must stop taking vitamin D before the study is over, the study doctor may ask you to continue to be part of the study and return for some study visits and procedures.

IF I HAVE TO PERMANENTLY STOP TAKING STUDY-PROVIDED VITAMIN D, OR ONCE I LEAVE THE STUDY, HOW WOULD DRUGS BE PROVIDED?

# **During the study:**

If you must permanently stop taking study-provided vitamin D before your study participation is over, the study staff will discuss other options that may be of benefit to you.

## After the study:

After you have completed your study participation, the study will not be able to continue to provide you with vitamin D that you received on the study. If continuing to take vitamin D or similar drugs/agents would be of benefit to you, the study staff will discuss how you may be able to obtain them.

## WHAT ARE THE RISKS OF THE STUDY?

## Risks of PrEP

The drug used in this study, Tenofovir-Emtricitibine, also known as Truvada, may have side effects, as listed in the CCTG 595 consent form.

## Risks of Vitamin D

- High calcium levels in the blood (muscle weakness, headache, indifference, loss of appetite, nausea/vomiting, bone pain, calcium deposits in the tissues of the body, kidney disease, high blood pressure, and irregular heartbeats)
- High calcium levels in urine (kidney stone disease and kidney failure)

NOTE: With the doses of vitamin D provided in the study, the risk of having high calcium in blood or urine is low.

If you have questions concerning side effects of vitamin D, please ask the medical staff at your site.

There is a risk of serious and/or life-threatening side effects when non-study medications are taken with any of the study drugs. For your safety, you must tell the study doctor or nurse about all medications you are taking before you start the study and also before starting any new medications while on the study. Also, you must tell the study doctor or nurse before enrolling in any other clinical trials while on this study.

## SIGNATURE PAGE

If you have read this consent form (or had it explained to you), all your questions have been answered and you agree to take part in this study, please sign your name below.

| Participant's Name (print) | Participant's Signature and Date |
|---|---|
| Participant's Legally Authorized<br>Representative (print)<br>(As appropriate) | Participant's Legally Authorized Representative's Signature and Date |
| Study Staff Conducting<br>Consent Discussion (print) | Study Staff's Signature and Date |
| Witness's Name (print)<br>(As appropriate) | Witness's Signature and Date |

Appendix V: Multivitamin Supplement Comparisons

| Appendix v: Multivitamin Supplement Comparisons | | | | | |
|---|---|---|---|---|---|
| | 1.4.10.11 | | | | |
| | Multivitamin Supplement | | | | |
| | Calcium and Vitamin D content | | | | |
| References | Drug Facts and Comparisons | | | | |
| | Dietary Supplements Database | | | | |
| | (http://dietarysupplements.nlm.nih.gov) | | | | |
| | | | Calcium/ | | |
| Manufacturer/ | | | serving | VitD/serving | |
| Brand | Product | servings | (mg) | (IU) | |
| | NA. Iki Vita main and NA. Iki NAin and | | | | |
| 24 at Cantum | Multi Vitamin and Multi Mineral | 2 toblete | 4500 | 400.00 | |
| 21st Century | Diabetes formula | 3 tablets | 1500 | 400.00 | |
| | CM Super Calaium 9 Magnasium | - | | | |
| 41 ifo | CM Super Calcium & Magnesium | 2 tablete | 2000 | 400.00 | |
| 4Life | Superiority Multiplex Vitamin & Mineral Formula | 3 tablets | 2000 | 400.00 | |
| | RiteStart Men | 2 tablets | 100<br>225 | 400.00 | |
| | RiteStart Wen RiteStart Women | 2 tablets<br>2 tablets | 1100 | 400.00<br>400.00 | |
| | Transfer Factor | 2 tablets | 200 | 400.00 | |
| | Farance Oliver as Buttone Bird | | | | |
| A1 | Emergen C Immune Defense Drink | 4 | 50 | 400.00 | |
| Alacer | Mix | 1 packet | 50 | 100.00 | |
| | EmerGen-C Kids Multi (various | 4 | 00 | 400.00 | |
| | flavors) | 1 packet | 63 | 400.00 | |
| Albantaana | Coloium I D | Otobloto | 1000 | 400.00 | |
| Albertsons | Calcium + D | 2 tablets | 1200 | 400.00 | |
| Alcon | L Cana MV Major | 4 tablets | 330 | 400.00 | |
| Alcon | I Caps MV Major | 4 lablets | 330 | 400.00 | |
| American | Chewy Bears Multi Vitamin with | + | | | |
| Health | Calcium 250mg | 2 bars | 250 | 400.00 | |
| Health | More Than a Multiple (with or without | 2 bais | 230 | 400.00 | |
| | iron) | 3 tablets | 500 | 400.00 | |
| | 11011) | 2 | 300 | 400.00 | |
| | Nutri-Mega | capsules | 400 | 400.00 | |
| | | 34754.00 | 100 | 100.00 | |
| Amerifit | Estoven Plus Multi-Vitamin | 1 capsule | 200 | 1000.00 | |
| | Estroven PM | 1 capsule | 60 | 800.00 | |
| | Estroven Maximum Strength | 1 capsule | 100 | 400.00 | |
| AmeriScience | | | | | |
| S | Childrens Chewable | 1 tablet | 20 | 400.00 | |
| | Mens Master-Multi | 2 packets | 540 | 400.00 | |
| | Osteo | 1 tablet | 175 | 300.00 | |
| | Sleep | 4 tablets | 250 | 150.00 | |
| | Womens Master-Multi | 1 packet | 585 | 400.00 | |
| | Transition indictor main | . packet | 000 | 100.00 | |
| | | | 1 | 1 | 1 |

| AN | Active Womans Formula | 3 tablets | 400 | 400.00 | 1 |
|---|---|---|---|---|---|
| | Prenatal Plus | 4 tablets | 800 | 400.00 | |
| Anselmo | Super Multis | 3 tablets | 105 | 800.00 | |
| Atkins | Basic 3 | 3 tablets | 50 | 200.00 | |
| Atkilis | Dasic 3 | 3 tablets | 30 | 200.00 | |
| | Barefoot Coral Calcium Plus | 3 tablets | 250 | 400.00 | |
| | | | | | RX |
| Azur Pharm | Natalle-ez | 1 tablet | 100 | 400.00 | only |
| _ | | 0.11.1 | 222 | 100.00 | |
| Bayer | Citracal Plus Bone Density Builder | 2 tablets | 600 | 400.00 | |
| | Citracal Plus Heart Health | 1 tablet | 315 | 250.00 | |
| | Citracal UltraDense Calcium Citrate Petites | 2 caplets | 630 | 400.00 | |
| | Citracal UltraDense Calcium Citrate | | | | |
| | Tablets | 2 tablets | 400 | 400.00 | |
| | Citracal UltraDense Calcium Citrate | | | | |
| | Plus with Magnesium | 2 tablets | 500 | 250.00 | |
| | | 4 | 100 | 100.00 | |
| Belvedere | Healthy Day Multi | 1 tablet | 100 | 400.00 | |
| | One a Day | 1 tablet | 20 | 200.00 | |
| Diamatuusa | A diverse d Mars Mills | 6 | 400 | 400.00 | |
| Bionatures | Advanced Mega Multi | capsules<br>3 | 400 | 400.00 | |
| | Bone Support | capsules | 500 | 200.00 | |
| | Coral Calcium Plus - 1000mg | 1 tablet | 715 | 200.00 | |
| | Corai Calcium Fius - Tooomg | 1 tablet | 7 13 | 200.00 | |
| Biotics | Aqueous Multi-Plus | 1 tablet | 25 | 400.00 | |
| Diotioo | Bio-Multi Plus (all types) | 3 tablets | 200 | 400.00 | |
| | Bio Wali Flas (all types) | O tableto | 200 | 400.00 | |
| BodyTech | Tech X Lite | 1 packet | 300 | 240.00 | |
| | Tech X Mass Gainer | 1 packet | 500 | 200.00 | |
| | Tooli y made damer | 1 paonot | | 200.00 | |
| Breckenridge | Multifol Tablets | 1 tablet | 125 | 400.00 | |
| | | 1 10.00.0 | | | RX |
| | Vinate GT | 1 tablet | 200 | 400.00 | only |
| | | | | | RX |
| | Vinate II | 1 tablet | 200 | 400.00 | only |
| | | $\Box$ | | | RX |
| | Vinate-M | 1 tablet | 200 | 400.00 | only |
| | Vineta Calaiuss | 4 4-6-1-4 | 405 | 400.00 | RX |
| | Vinate Calcium | 1 tablet | 125 | 400.00 | only<br>RX |
| | Multifol Plus | 1 tablet | 100 | 400.00 | only |
| | Widition Flug | i tablet | 100 | 400.00 | Offiny |
| Bronson | | | | | |
| Laboratories | Calcium 600mg with Vitamin D | 4 tablets | 125 | 500.00 | |
| | Therapeutic Vitamin & Mineral | | .20 | 220.00 | |
| | Formula | 1 tablet | 100 | 400.00 | |

| Brookstone | BP Prenate | 1 tablet | 100 | 425.00 | RX<br>only |
|---|---|---|---|---|---|
| Canopy<br>Roads<br>Pharmaceutic | CDNIstel | 4 toblet | 100 | 425.00 | RX |
| als | CRNatal | 1 tablet | 100 | 425.00 | only |
| Carlson | Cardi-Rite | 4 tablets | 400 | 400.00 | |
| | Kids Chewable Vitamins with Minerals | 1 tablet | 50 | 400.00 | |
| | Liquid Cal Mag | 1 gelcap | 200 | 500.00 | |
| | Mini-Gel Vitamins & Minerals | 6 gelcaps | 1000 | 1200.00 | |
| | Mini-Multi Vitamins & Minerals | 1 tablet | 20 | 400.00 | |
| | Super-1-Daily Vitamins & Minerals | 1 tablet | 50 | 400.00 | |
| | Super-2-Daily Vitamins & Minerals | 2 tablets | 50 | 600.00 | |
| Centrum | Regular | 1 tablet | 200 | 400.00 | |
| | Performance | 1 tablet | 100 | 400.00 | |
| | Silver | 1 tablet | 200 | 400.00 | |
| | Women's Silver | 1 tablet | 500 | 800.00 | |
| | Men's Silver | 1 tablet | 250 | 600.00 | |
| | Chewable | 1 tablet | 108 | 400.00 | |
| | Cardio | 1 tablet | 54 | 200.00 | |
| | Advanced | 1 tablet | 162 | 400.00 | |
| | Ultra Men's Formula | 1 tablet | 210 | 600.00 | |
| | Ultra Women's Formula | 1 tablet | 500 | 800.00 | |
| | Kids Complete Chewable (various) | 1 tablet | 108 | 400.00 | |
| 0 1 1 1 | | 0 ( | 400 | 100.00 | |
| Country Life | Chewable Adult Multi | 8 wafers | 480 | 400.00 | |
| | Daily Total One | 2 wafers | 40 | 400.00 | |
| | Life Essential Lfe Caps | 8 caps | 320 | 400.00 | |
| | Max for Men | 4 tablets | 200 | 400.00 | |
| | Daily Multi Sorb | 2 tablets | 50 | 400.00 | |
| | Liquid Multi | 30ml | 50 | 400.00 | |
| | Life Superior Multiple | 3 wafers | 200 | 100.00 | |
| Cyclin | VITa-PMS Plus | 1 tablet | 167 | 17.00 | |
| Cypress | Calcium 600 with D | 1 tablet | 600 | 200.00 | |
| | Calvite P & D | 1 tablet | | 120.00 | |
| | Prenatal AD | 1 tablet | 200 | 400.00 | RX<br>only |
| | Prenatabs CBF | 1 tablet | 200 | 400.00 | RX<br>only |
| | Prenatab FA | 1 tablet | 200 | 400.00 | RX<br>only |
| | Prenatal 19 (Regular & Chewable) | 1 tablet | 200 | 400.00 | RX<br>only |
| | Prenatabs OBN | 1 tablet | 200 | 400.00 | RX<br>only |
| | Trinate | 1 tablet | 200 | 400.00 | RX |

| | | | | | only |
|---|---|---|---|---|---|
| | PrenaFirst | 1 tablet | 200 | 400.00 | RX<br>only |
| Cytosport | Cytogainer (all flaviors) | 6 scoops | 500 | 200.00 | |
| Сугозрогг | Muscle Milk (all flavors) | 240ml | 1000 | 600.00 | |
| | | | 0.70 | | |
| Douglas Labs | FM Support Pack Pro-PCA Fuel | 1 packet | 250 | 50.00 | |
| | Pro-PCA Fuei | 4 scoops | 250 | 200.00 | |
| | Ulta-Ostivone | capsules | 600 | 200.00 | |
| ETHEX | NutriSpire Tablets | 1 tablet | 200 | 400.00 | |
| | Prenatal MR 90 FE | 1 tablet | 250 | 400.00 | RX<br>only |
| | | | | 400.00 | RX |
| | NatalCare PIC Forte | 1 tablet | 250 | 400.00 | only<br>RX |
| | Advanced NatalCare | 1 tablet | 200 | 400.00 | only |
| | Ultra NatalCare | 1 tablet | 200 | 400.00 | RX<br>only |
| | | | 200 | | RX |
| | NatalCare GlossTabs | 1 tablet | 200 | 400.00 | only<br>RX |
| | Advanced-RF NatalCare | 1 tablet | 200 | 400.00 | only |
| | Prenatal Z Advance formula | 1 tablet | 200 | 400.00 | RX<br>only |
| | Prenatal RX 1 | 1 tablet | 200 | 400.00 | RX<br>only |
| | NataTab CFe | 1 tablet | 200 | 400.00 | RX<br>only |
| | NataTab FA | 1 tablet | 200 | 400.00 | RX<br>only |
| | CareNatal DHA | 1 tablet | 200 | 400.00 | RX only |
| | NatalCare Three | 1 tablet | 200 | 400.00 | RX<br>only |
| | Prenatal MTR with Selenium | 1 tablet | 200 | 400.00 | RX |
| | | | | | only<br>RX |
| | NatalCare Plus | 1 tablet | 200 | 400.00 | only<br>RX |
| | NatalCare PIC | 1 tablet | 125 | 400.00 | only<br>RX |
| | Cal-Nate | 1 tablet | 125 | 400.00 | only |
| | NatalCare RX | 1 tablet | 100 | 200.00 | RX<br>only |
| Everett | Vitafol Caplets | 1 caplet | 125 | 400.00 | |
| | Vitafol-PN Caplets | 1 caplet | 125 | 400.00 | |
| | Vitafol-OB Caplets | 1 caplet | 125 | 400.00 | |
| | Calcifolic-D Wafers | 1 wafer | 125 | 300.00 | D |
| | Vitafol-OB+DHA | 1 tablet | 100 | 400.00 | Rx |

| Freeda | Yelets Teenage Formula | 1 tablet | 60 | 400.00 |
|---|---|---|---|---|
| | Monocaps | 1 tablet | 50 | 400.00 |
| | Vitalets Chewables | 1 tablet | 80 | 200.00 |
| | Quintabs-M | 1 tablet | 30 | 400.00 |
| | Ultra-Freeda with Iron | 1 tablet | 83 | 133.00 |
| | Ultra-Freeda | 1 tablet | 83 | 133.00 |
| | Fem-Cal | 1 tablet | 80 | 100.00 |
| | Fem-Cal Citrate | 1 tablet | 60 | 80.00 |
| | KPN Prenatal with Extra Calcium | 1 tablet | 333 | 133.00 |
| | A-Free Prenatal | 1 tablet | 333 | 133.00 |
| Future | | | | |
| Biotics | Calcium Essentials | 6 caps | 900 | 100.00 |
| | Hair Skin and Nails | 6 tablets | 1200 | 400.00 |
| | | 3 | | |
| | MV Teen | capsules | 100 | 400.00 |
| | PMSharmony | 8 tablets | 600 | 200.00 |
| | Pressure Lo | 4 tablets | 1000 | 300.00 |
| | Vegetarian Super Multi | 6 tablets | 400 | 400.00 |
| | Vitomegamen | 3 tablets | 100 | 400.00 |
| | Vitomegawomen | 3 tablets | 100 | 400.00 |
| GNC | ActiveCal | 2 tablets | 1000 | 200.00 |
| | Calcimate Plus 800mg | 4 caps | 800 | 800.00 |
| | Calcium Citrate Plus 800 | 2 caps | 400 | 400.00 |
| | Chewable Calcium 600 | 1 tablet | 600 | 200.00 |
| | | 4 | | |
| | Coral Calcium | capsules | 800 | 400.00 |
| | Kids Multibite Plus minerals Chewable | 2 tablets | 30 | 400.00 |
| | Kids Vitamin Chews | 1 tablet | 150 | 400.00 |
| | | 4 | | |
| | Mega Men Sport | capsules | 400 | 400.00 |
| | Mega Teen | 3 tablets | 100 | 400.00 |
| | Mens Mega Men | 4 tablets | 400 | 400.00 |
| | | 2 | | |
| | Mens Mega Men 50 PLUS | capsules | 200 | 400.00 |
| | Men's Mega Multi Time Release | 2 tablets | 200 | 1600.00 |
| | Multi Mega Minerals | 2 tablets | 1000 | 400.00 |
| | Multi-Gel | 2 gelcaps | 200 | 400.00 |
| | Natural Brand Fantastic Fiber | 10gm | 250 | 400.00 |
| | Preventron | 4 tablets | 60 | 400.00 |
| | Solotron (with or without) | 1 tablet | 60 | 400.00 |
| | Solotron Platinum | 2 tablets | 200 | 400.00 |
| | Teen Chewable Mega Teen | 2 tablets | 100 | 400.00 |
| | Ultra Mega Gold (with or without iron) | 2 tablets | 100 | 400.00 |
| | ( | 2 | | |
| | Ultra Mega Green | capsules | 50 | 400.00 |
| | Ultra Mega Timed Release | 2 tablets | 100 | 400.00 |
| | Ultra Mega Two Timed Release (with | | | |
| | or without iron) | 2 tablets | 50 | 400.00 |
| | Women's Mega Multi Time Release | 2 tablets | 200 | 1600.00 |

| | Women's Prenatal without Iron | 2 tablets | 500 | 400.00 | |
|---|---|---|---|---|---|
| | Womens Ultra Mega | 2<br>capsules | 500 | 400.00 | |
| Garden of<br>Life | Living Calcium Advanced | 3 capsules | 500 | 300.00 | |
| | Living Multi Optimal Womens formula | 6 capsules | 400 | 200.00 | |
| | Vitamin Code 50 & Wiser Women | 4 capsules | 50 | 1000.00 | |
| | Vitamin Code Men | 4<br>capsules | 20 | 400.00 | |
| GlaxoSmithKl | | | | | |
| ine | Geritol Complete | 1 tablet | 148 | 400.00 | |
| | Fiber Choice Chewable | 1 tablet | 100 | 50.00 | |
| | Os-Cal Ultra | 1 caplet | 600 | 500.00 | |
| | Os-Cal Chewable | 1 caplet | 500 | 600.00 | |
| | Oscal-D | 1 caplet | 500 | 200.00 | |
| | Oscal Extra D | 1 caplet | 500 | 600.00 | |
| | Oscal Extra B | 1 tablet or | 300 | 000.00 | |
| | Oscal 500 + D | chewable | 500 | 400.00 | |
| Goldline | Therapeutic Tablets | 1 tablet | 400 | 400.00 | |
| | Calcarb 600 with Vitmain D | 1 tablet | 600 | 200.00 | |
| | Oyst-Cal-D | 1 tablet | 200 | 125.00 | |
| | Health HNS Fat Cutter | 4 tabs | 600 | 400.00 | |
| | Healthy N Fit Nutri Pack | 1 tablet | 1000 | 400.00 | |
| Hawthorne | ICAR Prenatal Therapy | 1 tablet | 600 | 200.00 | RX<br>only |
| Health Sense | Once Daily | 1 tablet | 400 | 400.00 | |
| Tieaitii Jeiise | Complete Senior | 1 tablet | 200 | 400.00 | |
| Hero<br>Nutritionals | Vegetarian Calcium with Vitamin D | 1 gummie | 125 | 100.00 | |
| Integrative<br>Therapeutics | Vitaline Total Formula 3 | 1 tablet | 500 | 400.00 | |
| Integrity | Stuart Prenatal | 1 tablet | 200 | 400.00 | RX<br>only |
| Irwin Naturals | Kids Supervitamin | 1<br>softchew | 150 | 400.00 | |
| | Super Calcium | capsules | 1000 | 400.00 | |
| | Mens Living Green Lig-Gel Multi | 3 gelcaps | 50 | 400.00 | |
|---|---|---|---|---|---|
| | Liqui-Gel Multi | 4<br>capsules | 100 | 200.00 | |
| | Elqui-Ger Walti | capsuics | 100 | 200.00 | |
| Ivax | Certagen Tablets | 1 tablet | 162 | 400.00 | |
| 17 4.21 | One-Tablet-Daily with Minerals | 1 tablet | 162 | 400.00 | |
| | Generix-T | 1 tablet | 58 | 400.00 | |
| | Prenatal S | 1 tablet | 200 | 400.00 | |
| Jarrow | All Canada Haalth Dale | 4 | 500 | 000.00 | |
| Formulas | All Capsule Health Pak | 1 packet | 500 | 200.00 | |
| | Bone-Up | capsules | 1000 | 400.00 | |
| | Вопе-ор | capsuics | 1000 | 400.00 | |
| KAL | Enhanced energy | 3 tablets | 300 | 400.00 | |
| | Amino-Max | 2 tablets | 1000 | 200.00 | |
| | Beyond Calcium Ipriflavone | 5 tablets | 1000 | 400.00 | |
| | Bone Meal | 4 tablets | 1000 | 400.00 | |
| | Cal Citrate Plus | 4 tablets | 1000 | 400.00 | |
| | Enhanced Energy Teen Complete | 1 tablet | 100 | 400.00 | |
| | | 2 | | | |
| | High Potency Soft Multiple | capsules | 200 | 400.00 | |
| | Mega Vita-Min | 1 tablet | 50 | 400.00 | |
| | Multi-Four Plus | 4 tablets | 500 | 400.00 | |
| | Multi-Max 1 | 1 tablet | 50 | 400.00 | |
| | Multiple Energy | 4 tablets | 500 | 400.00 | |
| | MultiSaurus DinoSours | 1 packet | 50 | 200.00 | |
| | Vita Mom Advanced | 3 tablets | 600 | 200.00 | |
| Kenwood/Bra | | + | | | |
| dley | Kenwood Therapeutic Liquid | 5ml | 250 | 133.00 | |
| dicy | rtenwood merupeatio Eiquid | Onn | 200 | 100.00 | |
| Kirkland | | | | | |
| Signature | Calcium 500mg + D | 2 tablets | 1000 | 400.00 | |
| | Calcium Chews 500mg + D + K | 2 chews | 1000 | 400.00 | |
| | Calcium Citrate, vitamin D, | | | | |
| | Magnesium & Zinc | 2 tablets | 500 | 250.00 | |
| | Childrens Chewable Multivitamin | 1 tablet | 200 | 400.00 | |
| | Daily Multivitamin Pack with Energy | | 4655 | 402.22 | |
| | Boosting Nutrients | 1 pack | 1200 | 400.00 | |
| | Daily Multivitamin with Lutein | 1 tablet | 162 | 400.00 | |
| | Mature Multi Vitamins & Minerals | 1 tablet | 200 | 400.00 | |
| | Premium Performance Multivitamin | 1 toblet | 165 | 400.00 | |
| | with Lycopene & Lutein | 1 tablet | 165 | 400.00 | |
| | | + | | | RX |
| Laser | Lactocal-F | 1 tablet | 200 | 400.00 | only |
| | | 1 | | | 1, |
| Leiner | One Daily Mens Health Formula | 1 tablet | 210 | 400.00 | |

| Life | | 1 | 1 | 1 | 1 |
|---|---|---|---|---|---|
| Enhancement | 3-way Calcium complex (Womens | 2 | | | |
| S | Health) | capsules | 500 | 400.00 | |
| | Troditi') | 4 | 000 | 100.00 | |
| | BioEnhance with DNAble | capsules | 1000 | 50.00 | |
| | | • | | | |
| Life | | | | | |
| Extension | Childrens Formula Life Extension Mix | 2 tablets | 100 | 400.00 | |
| | Mix with Extra Niacin Without Copper | 4 tablets | 100 | 400.00 | |
| | LifePlus Daily Biobasics | 1 scoop | 500 | 300.00 | |
| | Lie inia Or Mar 7in | 4.051 | 1000 | 400.00 | |
| | Liquimins Ca; Mag Zinc | 1.25ml | 1200 | 400.00 | |
| | | | | + | |
| | Longs Womnes | | | | |
| | Multivitamin/Multimineral.Herbs | 2 tablets | 500 | 400.00 | |
| | Waltavitariiii/Waltariiiierai.i ieroo | Z tablets | 000 | 400.00 | |
| | | 2 | | | |
| | MD Select Advanced Breast support | capsules | 225 | 400.00 | |
| Major | Certavite with Lutein | 1 tablet | 162 | 400.00 | |
| | Certavite with Lutein | 1 tablet | 160 | 400.00 | |
| | High Potency | 1 tablet | 60 | 400.00 | |
| | Thera Calcium 600-D | 1 tablet | 400 | 400.00 | |
| | | 1 tablet | 600 | 200.00 | |
| | Oyster Shell Calcium 500 + D Oyster Shell Calcium with D | 1 tablet<br>1 tablet | 500<br>400 | 200.00<br>125.00 | |
| | Prenatal Plus | 1 tablet | 200 | 400.00 | + |
| | r Terratar Flus | 1 tablet | 200 | 400.00 | |
| | | | | | RX |
| Marmel | Marnatal-F Plus | 1 tablet | 250 | 400.00 | only |
| | | | · | | |
| McNeil | Viactiv | 1 caplet | 200 | 400.00 | |
| | Viactiv for Teens | 1 tablet | 500 | 200.00 | |
| | Viactiv Calcium plus Vitamin D and K | 1 chew | 500 | 100.00 | |
| | Viactiv Flavor Glides | 1 glide | 500 | 100.00 | |
| | Viactiv Multi Vitamin Flavor Glides | 1 glide | 200 | 400.00 | |
| | Viactiv Multivitamin Chocolate Milk | 8oz | 200 | 400.00 | |
| <del></del> | | | | | |
| Michaels | Childrene Chewahles | 1 wofers | 200 | 400.00 | |
| Neuropathic | Childrens Chewables JUST ONE Multivitamin | 4 wafers<br>1 tablet | 200 | 400.00<br>400.00 | |
| | Vision Factors | 6 tablets | 50<br>150 | 100.00 | |
| | VISION FACIOIS | U labiels | 100 | 100.00 | |
| Miller | Rague | 1 tablet | 102 | 133.00 | |
| Miller | Ragus<br>Complere | 1 tablet | 193<br>150 | 133.00<br>133.00 | |

| | Theramill Plus | 1 tablet | 67 | 33.00 | 1 |
|---|---|---|---|---|---|
| | Theramill Forte | 1 capsule | 67 | 33.00 | |
| Mission | Calcet Plus | 1 tablet | 160 | 400.00 | |
| | Fosfree | 1 tablet | 175 | 150.00 | |
| | Citracal | 1 caplet | 315 | 200.00 | |
| | Citracal Plus | 1 caplet | 300 | 125.00 | |
| | Calcet | 1 tablet | 200 | 100.00 | |
| | Citracal Prenatal 90 + DHA | 1 tablet | 200 | 400.00 | RX<br>only |
| | CitraNatal 90 DHA | 1 tablet | 200 | 400.00 | RX<br>only |
| | Citracal Prenatal + DHA | 1 tablet | 125 | 400.00 | RX<br>only |
| | CitraNatal DHA | 1 tablet | 125 | 400.00 | RX<br>only |
| | CitraNatal Rx | 1 tablet | 125 | 400.00 | RX<br>only |
| | Prenatal F.A | 1 tablet | 50 | 400.00 | |
| | Prenatal HP | 1 tablet | 50 | 400.00 | |
| | Prenatal | 1 tablet | 50 | 400.00 | |
| | 14.5 | 44.11.4 | 222 | 100.00 | |
| Natrol | My Favorite Multiple | 4 tablets | 200 | 400.00 | |
| | My Favorite Multiple with Coral Calcium and Zeanthin | 2 capsules | 250 | 400.00 | |
| Naturade | Head Start Nutritional Breakfast drink | 240ml | 200 | 100.00 | |
| | Power Shake | 1 scoop | 280 | 400.00 | |
| | Ribo-tein Vital | 1 scoop | 280 | 400.00 | |
| | Super Weight Gain | 4 scoops | 30 | 200.00 | |
| Natural | Big Friends Childrens Chewable | | | | |
| Factors | (various flavors) | 1 tablet | 65 | 400.00 | |
| | Calcium & Magnesiuim Citrate with D | 4 tablets | 1000 | 400.00 | |
| | Mens 50 Plus MultiStart | 4 tablets | 400 | 200.00 | |
| | Mens MultiStart | 4 tablets | 400 | 100.00 | |
| | MulitFactors Womens 50 Plus | 3<br>Capsules | 200 | 1000.00 | |
| | MultiStart prenatal | 3 capsules | 500 | 50.00 | |
| | Super Multi Iron Free | 1 tablet | 125 | 400.00 | |
| | Ultra Multi Plus | 1 tablet | 125 | 400.00 | |
| | Womens MultiStart | 3 tablets | 500 | 200.00 | |
| | Womens Plus MultiStart | 3 tablets | 500 | 200.00 | |
| Nature Made | Women's Multi for Her | 1 tablet | 250 | 1000.00 | |
| - I I I I I I I I I I I I I I I I I I I | Men's Multi for Him | 1 tablet | 162 | 1000.00 | |
| | Women's Multi for Her 50+ | 1 tablet | 250 | 1000.00 | |
| | Men's Multi for Him 50+ | 1 tablet | 162 | 1000.00 | |
| | Advanced High Absorption Calcium with 100mg Phytonutrients | 2 tablets | 500 | 200.00 | |

| | Calcium Magnesium Zinc with Vitamin | 1 1 | | ĺ |
|---|---|---|---|---|
| | D | 1 tablet | 333 | 200.00 |
| | Calcium Plus soy | 1 tablet | 500 | 200.00 |
| | Calcium with Vitamin D | 1 tablet | 600 | 200.00 |
| | Diabetes Health Pack | 1 packet | 200 | 400.00 |
| | Essential 50+ | 1 tablet | 200 | 400.00 |
| | Essential Balance Compete Multi | | | |
| | Vitamin/Mineral | 1 tablet | 100 | 400.00 |
| | Essentail Daily | 1 tablet | 450 | 400.00 |
| | Essential Man 50+ | 1 tablet | 450 | 400.00 |
| | Essential multi Plus Energy | 1 tablet | 50 | 200.00 |
| | Essential Woman 50+ | 1 tablet | 250 | 400.00 |
| | Man with Lycopene | 1 tablet | 100 | 400.00 |
| | Maximin Pack | 1 packet | 850 | 800.00 |
| | Mens Pack | 1 packet | 350 | 400.00 |
| | Multi Complete with Iron & Calcium | 1 softgel | 100 | 1000.00 |
| | Multi for Her with Iron & Calcium | 1 softgel | 100 | 1000.00 |
| | Multi Prenatal Premium | 1 tablet | 200 | 400.00 |
| | man i onata i formani | , tablet | 200 | 700.00 |
| | Disney Princess Complete | | | |
| NatureSmart | Multivitamin Chewable Tablet | 1 tablet | 100 | 400.00 |
| rtatar o o mart | Winnie the Pooh Chewables | 1 tablet | 100 | 400.00 |
| | Gummies (Finding Nemo, Winnie the | 1 | 100 | 100.00 |
| | Pooh, etc) | gummies | 100 | 400.00 |
| | 1. 3311, 3337 | gammee | | 100.00 |
| Natures Best | Hardcore Pack | 1 packet | 1100 | 400.00 |
| | Zero Carb Isopure | 1 scoop | 300 | 100.00 |
| Nature's | | | | |
| Bounty | Theravim-M | 1 tablet | 40 | 400.00 |
| • | Multi-Day plus Minerals | 1 tablet | 162 | 400.00 |
| | Mega VM-80 | 1 tablet | 19 | 400.00 |
| | Absorbable Calcium 1220 + D | 2 softgels | 1200 | 200.00 |
| | Calcium 500mg with Vitamin D | 4 tablets | 120 | 500.00 |
| | Calcium 600 + Vitamin D with Soy | | - | |
| | Isoflavones | 2 tablets | 100 | 400.00 |
| | Chewable Calcium Wafers Plus | | | |
| | Vitamin D | 2 wafers | 200 | 200.00 |
| | Coral Calcium 1000mg Plus Vitamin D | | | |
| | and Magnesium | 2 tablets | 370 | 400.00 |
| | Green Source | 3 tablets | 250 | 400.00 |
| | Hair Skin and Nails Formula | 3 tablets | 830 | 100.00 |
| | High Potency Vitamin D 1000IU | 1 tablet | 120 | 1000.00 |
| | Multi-Day Weight Trim with Green Tea EGCG | 1 tablet | 300 | 400.00 |
| | Oystercal-D Calcium 500mg with | 1 100101 | | .00.00 |
| | Vitamin D3 | 1 tablet | 500 | 400.00 |
| | Pre-Natal Formula | 1 tablet | 200 | 400.00 |
| | Prescriptive Formulas Optimal Mens | 1 packet | 712 | 200.00 |
| | Prescriptive Formulas Optimal Prescriptive Formulas Optimal | ι ρασκει | 112 | 200.00 |
| | Womens Optimal | 1 packet | 975 | 525.00 |

| | Soy Protein shake Powder | 30gm | 900 | 40.00 |
|---|---|---|---|---|
| | Ultra Man Time Release | 2 tablets | 200 | 200.00 |
| | Ultra Vita-Min | 1 tablet | 60 | 400.00 |
| | Ultra Woman | 2 tablets | 500 | 400.00 |
| | Vitmain D 2000IU | 1 tablet | 1500 | 2000.00 |
| Natures Life | Antioxidant Soft Multi | 2 sofgels | 200 | 400.00 |
| | Great Greens | 3 tablets | 250 | 800.00 |
| | Green Pro-96 Multi | 1 tablet | 50 | 200.00 |
| | One Daily Vegetarian Multiple | 1 capsule | 20 | 400.00 |
| | | 6 | | |
| | Prenatal Multiple | capsules | 1000 | 200.00 |
| | Soft Gelatin Multiple | 2 softgels | 200 | 400.00 |
| | Stress Soft Multi | 2 softgels | 200 | 400.00 |
| | Ultra Mega Vite Multi | 1 tablet | 100 | 400.00 |
| | A L H OL LL MA HOTEL | | | |
| Natures Plus | Adults Chewable MultiVitamin and Minerals | 1 tablet | 10 | 400.00 |
| Natures Flus | | | 80 | |
| | Adults Chewable Vitamin D3 1000IU | 1 tablet | 80 | 1000.00 |
| | Adults Dental Care Probiotic Lozenges | lozenges | 150 | 400.00 |
| | Adults Multi-Vitamin Chewable | 1 tablet | 10 | 400.00 |
| | Childrens Chewable Dental Probiotic | i tablet | 10 | 400.00 |
| | (various flavors) | 2 tablets | 300 | 400.00 |
| | Bone Power - Calcium with Boron | 4 softgels | 1000 | 200.00 |
| | Dyno Vites Sustained Release | 2 tablets | 50 | 1000.00 |
| | Golden Years | 6 tablets | 300 | 400.00 |
| | Especially Yours Women's Multiple | 3 tablets | 150 | 400.00 |
| | Liquid Bone Power | 15ml | 1000 | 200.00 |
| | Liquid Calcium | 15ml | 1000 | 40.00 |
| | Love Bites Childrens Chewable | 1 tablet | 20 | 400.00 |
| | Mega Force Tablets for Men Only | 3 tablets | 25 | 400.00 |
| | Nutri-Genic Softgels for Sensitive | o tablete | 20 | 100.00 |
| | People | 2 softgels | 50 | 400.00 |
| | Nutri-Genic Tablets for Sensitive | | | |
| | People | 2 tablets | 50 | 400.00 |
| | Power Teen for Her Chewable | 2 tablets | 100 | 500.00 |
| | Power Teen for Him Chewable | 2 tablets | 50 | 500.00 |
| | Power-Plex sustained release | | | |
| | MultiVitamin and Mineral | 1 tablet | 26 | 400.00 |
| | Regeneration Liquid Sunshine | 60ml | 200 | 400.00 |
| | Regeneration Multivitamin and mineral | | | |
| | Softgels | 3 softgels | 100 | 400.00 |
| | Source of Life Adults Chewable Multi | 2 wafers | 100 | 400.00 |
| | Source of Life Animal Parade Liquid | 30ml | 20 | 200.00 |
| | Source of Life GOLD Mini-Tablets | 3 tablets | 250 | 400.00 |
| | Source of Life Gold tablets | 3 tablets | 250 | 400.00 |
| | Source of Life Gold Vcaps (Vegan) | 9 caps | 250 | 1000.00 |
| Natures | womens Whole Body Daily | | | |
| Secret | Multivitamin | 2 softgels | 100 | 400.00 |

| | | 1 1 | 1 | | 1 1 |
|---|---|---|---|---|---|
| Natures | Super Supplemental Vitamins and | | | | |
| Sunshine | Minerals without Iron | 4 tablets | 400 | 600.00 | |
| Natures Way | Alice Iron-Free Multivitamin | 3 tablets | 250 | 400.00 | |
| | Alive Mens Multivitamin & Mineral | 3 tablets | 250 | 800.00 | |
| | Alive Womens Multivitamin & Mineral | 3 tablets | 500 | 1000.00 | |
| | BoneSoy | 2 tablets | 400 | 133.00 | |
| | | 3 | | | |
| | Coral Calcium | capsules | 600 | 200.00 | |
| | Natures Way Alive | 3 tablets | 250 | 400.00 | |
| | Once Daily Women's 50 +Ultra | | | | |
| | Potency | 1 tablet | 500 | 1000.00 | |
| | Once Daily Men's 50 +Ultra Potency | 1 tablet | 100 | 1000.00 | |
| | Alive Once Daily Energy 50 + | 1 tablet | 100 | 1000.00 | |
| Nam Objects | Firem Warrana Da'' | 4 += -1 | 40 | 400.00 | - |
| New Chapter | Every Womans Daily | 1 tablet | 10 | 400.00 | |
| | Bone Strength Take Care | 3 tablets | 680 | 800.00 | |
| | Every Man | 3 tablets | 8 | 400.00 | |
| | Every Woman | 3 tablets | 25 | 400.00 | |
| | Every Woman II | 6 tablets | 75<br>2 | 400.00 | |
| | Only One Perfect Prenatal | 1 tablet | | 400.00 | |
| | | 3 tablets | 30<br>5 | 400.00 | |
| | Unbound Energy | 3 tablets | 5 | 1000.00 | |
| | | 4 | | | |
| New Phase | Complete Menopause Support | capslets | 800 | 400.00 | |
| Nnodum | | | | | |
| Pharmaceutic | | | | | RX |
| als | Inatal Advance | 1 tablet | 200 | 400.00 | only |
| | | | | | RX |
| | Inatal Ultra | 1 tablet | 200 | 400.00 | only |
| No de Ora | Della Defense Di e | 3 | 000 | 000.00 | |
| North Star | Daily Defense Plus | capsules | 200 | 200.00 | |
| | Ultimate Bionic Plus | 1 packet | 500 | 400.00 | |
| Novato | Multivitamin Plus | 1 tablet | 200 | 400.00 | |
| NOVALO | Widilivitailiii Fius | 2 | 200 | 400.00 | |
| | Super Multivitamins | capsules | 50 | 400.00 | |
| Now Foods | Full Spectrum Minerals | 2 tablets | 1000 | 200.00 | 1 |
| | | 3 | | | |
| | ADAM Superior | capsules | 350 | 400.00 | <u> </u> |
| | Bone Calcium | 4 tablets | 1000 | 200.00 | |
| | Daily Vits Vitamin | 1 tablet | 150 | 100.00 | |
| | Calcium Citrate | 2 tablets | 600 | 100.00 | |
| | | 2 | | | |
| | Eco-Green Multi Vitamin | capsules | 50 | 100.00 | |
| | Full Spectrum Minerals | 2 tablets | 1000 | 200.00 | |
| | Kids Vit Chewable (various flavors) | 2 tablets | 40 | 200.00 | |

| | Liquid Cal Mag | 15ml | 500 | 400.00 | Ī |
|---|---|---|---|---|---|
| | Liquid Multi Gels | 2 gelcaps | 100 | 400.00 | |
| | Magnesium & Calcium | 3 tablets | 400 | 200.00 | |
| | Magnesium & Calcium | 3 tablets | 700 | 200.00 | |
| | | 6 | | | |
| NSI | Prenatal Plus | capsules | 1300 | 400.00 | |
| | | 2 | | | |
| | Synergy Basic Multi Vitamin Version 2 | capsules | 20 | 700.00 | |
| | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 8 | 50 | 700.00 | |
| | Synergy Mens Multi Vitamin Version 2 | capsules<br>6 | 50 | 700.00 | |
| | Synergy Multi Vitamin Version 10 | capsules | 500 | 1000.00 | |
| Nutrilite | Col Mag D | 4 tablets | 1000 | 400.00 | |
| Nutrille | Cal Mag D | | 1000 | 400.00 | |
| | Daily Multivitamin and Multimineral | 1 tablet | 200 | 400.00 | |
| | | 1 | | | |
| <b>Nutrition Now</b> | Calcium Soft Chews | softchew | 500 | 100.00 | |
| | Rhino Beanie Vites | 2 tablets | 4 | 100.00 | |
| | Rhino Calcium | 1 tablet | 250 | 100.00 | |
| | Rhino Wigglers | 1 wiggler | 2 | 400.00 | |
| One A Day | Essential Multi | 1 tablet | 45 | 400.00 | |
| _ | Men's Health | 1 tablet | 210 | 400.00 | |
| | Men's 50+ | 1 tablet | 120 | 400.00 | |
| | Women's | 1 tablet | 450 | 800.00 | |
| | Maximum | 1 tablet | 162 | 400.00 | |
| | Complete Chewable (Flintstones, | | | | |
| | Bugs Bunny, Scooby Doo, etc | 1 tablet | 100 | 400.00 | |
| | Gummies (Flintstones, Bugs Bunnies, | | | | |
| | etc | 1 gummie | 100 | 400.00 | |
| | Energy | 1 tablet | 250 | 400.00 | |
| | Active | 1 tablet | 110 | 400.00 | |
| | Cholesterol Plus | 1 tablet | 200 | 400.00 | |
| | Daily Multivitamin Vital Body and Cells | 4 (-11-4 | 222 | 400.05 | |
| | Formula | 1 tablet | 200 | 400.00 | |
| | Joint and Bone Vitality | 1 tablet | 250 | 67.00 | |
| | Men's Pro Edge | 1 tablet | 200 | 800.00 | |
| | Menopause Formula | 1 tablet | 300 | 800.00 | |
| | Women's Prenatal | 1 tablet | 300 | 400.00 | |
| | Women's Active Mind & Body | 1 tablet | 300 | 800.00 | |
| | Women's Active Metabolism | 1 tablet | 300 | 800.00 | |
| | Weight Smart | 1 tablet | 300 | 400.00 | |
| | Carb Smart | 1 tablet | 200 | 400.00 | |
| | Today Science Daily | 1 tablet | 240 | 400.00 | |
| | , | 1 tablet | 250 | 400.00 | - |
| | Nutrilite Toop Advantage for Her | 1 tablet | 200 | 400.00 | |
| | Teen Advantage for Her | 1 tablet | 300 | 800.00 | |
| | Teen Advantage for Him | 1 tablet | 200 | 400.00 | |
| Optimox | Gynovite Plus | 1 tablet | 83 | 67.00 | |

| Optimum | 1 | | 1 | ĺ | ĺ |
|---|---|---|---|---|---|
| Nutrition | OptiMen | 3 tablets | 200 | 300.00 | |
| | | 2 | | 300.00 | |
| | OptiWomen | capsules | 150 | 600.00 | |
| | Nutrition Serious Mass | 2 scoops | 590 | 200.00 | |
| | | ' | | | |
| Perque | Life Guard | 2 tablets | 50 | 400.00 | |
| • | | 4 | | | |
| | Bone Guard Forte 20 | capsules | 500 | 400.00 | |
| | | 1 | | | |
| | Life Guard Chewables | chewable | 50 | 200.00 | |
| | Mito Guard 100 Plus | 1 tablet | 50 | 200.00 | |
| Pfizer | Myadec | 1 tablet | 162 | 400.00 | |
| | | 2 tablets | | | |
| | | or | | | |
| | Caltrate 600-D | softchews | 1200 | 800.00 | |
| | | 2 tablets | | | |
| | | or | | | |
| | Caltrate 600-D Plus minerals | softchews | 1200 | 800.00 | |
| Pharmanex | Bone Formula | 2 tablets | 250 | 50.00 | |
| | Life Essentials | 1 tablet | 100 | 200.00 | |
| | LifePak Kosher | 1 packet | 250 | 200.00 | |
| | LifePak Prenatal | 1 packet | 325 | 200.00 | |
| | LifePak Prime Anti Aging Formula | 1 packet | 500 | 300.00 | |
| | LifePak Teen | 1 capsule | 250 | 200.00 | |
| | LifePak Women | 1 packet | 500 | 200.00 | |
| | | 1 | | | |
| | Nutrimmune chews | chewtab | 250 | 50.00 | |
| | | 2 | | | |
| | Vitox | capsules | 250 | 200.00 | |
| Pharmaton | Ginsana Gold Formula | 2 softgels | 200 | 400.00 | |
| | | | | | RX |
| Pharmics | O-Cal FA | 1 tablet | 200 | 400.00 | only |
| PhysioLogics | MultiLogics Iron-Free Once Daily | 1 capsule | 92 | 400.00 | |
| | OsteoLogic Pro | 2 tablets | 400 | 150.00 | |
| | Phytotality Daily Multivitamin + | | | | |
| | Minerals | 3 tablets | 252 | 400.00 | |
| | Ultra MultiLogics for Men High | | | 400.00 | |
| | Potency | 2 tablets | 200 | 400.00 | |
| | Ultra Multillogics for Women High | | | | |
| | Potency | 2 tablets | 500 | 600.00 | |
| Precision | Mills and Eng Destate D | 4 | 000 | 440.00 | |
| Engineered | Milk and Egg Protein Powder | 1 scoop | 600 | 140.00 | |
| | Muscle Weight Gainer | 5 tbs | 1100 | 200.00 | |
| | ProtoPlex Deluxe | 3 scoops | 600 | 200.00 | |

| | Age-Defying Multivitamin & Mineral for | | | |
|---|---|---|---|---|
| Prevention | Men 50 Plus | 2 tablets | 250 | 400.00 |
| | Diabetic Support MultiNutrient | 2 tablets | 240 | 400.00 |
| | High Potency Multivitamin & Mineral | | | |
| | for Women | 1 tablet | 250 | 400.00 |
| Prime | | | | |
| Marketing | Thera-M with Minerals | 1 tablet | 40 | 400.00 |
| | Complete Tablets | 1 tablet | 162 | 400.00 |
| | Prenatal | 1 tablet | 200 | 400.00 |
| Pure | | 6 | | |
| Encapsulatio ns | Nutrient 950 (various formulations) | 6 | 300 | 800.00 |
| 115 | PureBears | capsules<br>2 tablets | | |
| | PureBears | 3 | 100 | 400.00 |
| | Daily Multi | capsules | 200 | 200.00 |
| | Daily Walti | capsules | 200 | 200.00 |
| Puritans | ABC PLUS SENIOR with Lutein & | + | + | |
| Pride | Lycopene | 1 tablet | 200 | 400.00 |
| 11140 | Lycoponic | 2 | 200 | 100.00 |
| | Absorbable Calcium with Vitamin D | capsules | 1000 | 100.00 |
| | | 1 | | 100100 |
| | Adult Chewable Multi-Vitamin | chewtab | 10 | 400.00 |
| | Calcium Magnesium with D | 3 tablets | 1000 | 400.00 |
| | Childrens Chewable Animal Chews | 1 | | |
| | (various formaltions) | chewtab | 125 | 200.00 |
| | | 1 | | |
| | Childrens Chewable Multivitamin | chewtab | 50 | 400.00 |
| | Complete One | 1 tablet | 54 | 400.00 |
| | Daily 3 Multiple with Cholesterol | 3 | | |
| | Regulators | capsules | 106 | 800.00 |
| | Formula 100 with Beta Carotene | 1 tableet | 100 | 400.00 |
| | Green Source | 3 tablets | 750 | 400.00 |
| | High Potency Calcium 600 + Vitamin | | | |
| | D | 2 tablets | 1200 | 400.00 |
| | Iron Free green Source | 3 tablets | 252 | 400.00 |
| | Mega Vita Gel | 2 softgels | 200 | 400.00 |
| | Mega Vita Min for Seniors | 2 tablets | 200 | 400.00 |
| | Mega Vita Min for Women | 2 tablets | 500 | 400.00 |
| | Mega Vita min for Women Timed | 0.4-1-1-1 | F 4 0 | 400.00 |
| | Release | 2 tablets | 510 | 400.00 |
| | Mega Vita Min | 1 capsule | 15 | 400.00 |
| | Multi-Day Plus Minerals | 1 tablet | 162 | 400.00 |
| | Multi-Day Take One Green Tea | 4 40 61 - 4 | 200 | 400.00 |
| | Formula | 1 tablet | 300 | 400.00 |
| | Potent 75 Super VM | 1 tablet | 50 | 400.00 |
| | Propostal Compley | 4 | 1200 | 400.00 |
| | Prenatal Complex Puritron | capsules<br>6 tablets | 1300 | 400.00<br>400.00 |
| | | | 800 | |
| | Super All Day Nutricom Powder | 15gm | 500 | 400.00 |
| | Ultra Vita-Mam Time Release for Men | 2 tablets | 200 | 200.00 |

| | Ultra Vita-Min VM-33 | 1 tablet | 60 | 400.00 |
|---|---|---|---|---|
| | Vita-min Complete Formula 1 | 6 tablets | 800 | 200.00 |
| | · | 3 | | |
| | Whole Food Concentrate | capsules | 500 | 400.00 |
| Quantum | Mega 1 Daily Iron Free | 1 capsule | 25 | 200.00 |
| 40.00.110.111 | Natures Daily Multi Vitamin | 1 tablet | 50 | 400.00 |
| | Complete Super Vitamin Multi | 1 tablet | 50 | 400.00 |
| Radiance | Absorbable Calcium with Vitamin D | 2 softgels | 1000 | 100.00 |
| - Tuurun - O | Calcium 600 + Vitamin D | 2 tablets | 1200 | 250.00 |
| | Coral Calcium 500 Plus | 2 capsules | 370 | 400.00 |
| | Green Source Multivitamins and | capsules | 370 | 400.00 |
| | minerals | 3 tablets | 250 | 400.00 |
| | Mega Vita Gel | 2 softgels | 200 | 400.00 |
| | Mega Vita Min for women | 2 tablets | 500 | 400.00 |
| | Mega Vita Min High Potency 9 time | | | |
| | Release | 2 tablets | 500 | 400.00 |
| | Prenatal Vitamin | 1 tablet | 200 | 400.00 |
| | Skin, Hair & Nails Formula | 3 tablets | 834 | 100.00 |
| | Ultra Vita Man High Potency Timed | | | |
| | Release | 2 tablets | 200 | 200.00 |
| | Vanilla Soy Protein shake | 30gm | 200 | 200.00 |
| Rainbow | | | | |
| Light | Active Health Teen Multi | 3 tablets | 200 | 100.00 |
| | Active Senior Multivitamin | 1 tablet | 200 | 400.00 |
| | Advanced Nutritional System | 6 tablets | 240 | 400.00 |
| | Complete Menopause Support | 4 tablets | 1000 | 400.00 |
| | Everyday Calcium with Enzymes | 4 tablets | 1200 | 200.00 |
| | Just Once Iron Free Safe Guard | | | |
| | multivitamin | 1 tablet | 30 | 400.00 |
| | Just Once Food Based Calcium | 1 tablet | 500 | 200.00 |
| | Mens One Multivitamin | 1 tablet | 50 | 400.00 |
| | Nutritional Systems NutriStars | 2 tablets | 40 | 50.00 |
| | Prenatal One Multivitamin | 1 tablet | 200 | 400.00 |
| | Womens Nutritional System | 6 tablets | 1000 | 400.00 |
| | Womens One Multivitamin | 1 tablet | 200 | 400.00 |
| | Womens Whole Nutrition Liquid Multi | 2 softgels | 100 | 400.00 |
| | Mens Whole Nutrition Liqiud Multi | 2 softgels | 100 | 400.00 |
| Reliv | RelivClassic | 2 scoops | 1000 | 400.00 |
| | RelivNow for kids | 2 scoops | 1000 | 400.00 |
| | Simplicity | 1 scoop | 500 | 200.00 |
| | Cimplicity | | | |
| Rexall- | | . 33336 | | |
| Rexall-<br>Sundown | | · | 162 | 400.00 |
| | Complete Daily with Lutein SunVite | 1 tablet | | |
| | Complete Daily with Lutein | 1 tablet | 162 | 400.00 |

| Vitamins to Go Maximum | 1 tablet | 777 | 525.00 | |
|---|---|---|---|---|
| Osteo Bi-Flex Plus Calcium With | | - | | |
| Vitamins C and D | 3 caplets | 500 | 400.00 | |
| | 4 4-6-1-4 | 405 | 400.00 | |
| Multivitamin/Mineral | | 165 | 400.00 | |
| Calcium Soft Chows | • | 500 | 100.00 | |
| Ochilai Vite | Tablet | 102 | 30.00 | |
| | | | | RX |
| VitaPhil | 1 tablet | 100 | 400.00 | only |
| , | | | | |
| Prenavite | 1 tablet | 200 | 400.00 | |
| | · . | | | |
| | chewtab | 20 | 200.00 | |
| | 0.1-1-1-1- | 4000 | 400.00 | |
| Prime Years Multi Vitamin | | 100 | 400.00 | |
| Prostrato Health | | 20 | 400.00 | |
| | 2 surigers | 1200 | 400.00 | |
| | 1 tablet | 25 | 400.00 | |
| | 2 | | | |
| Carotene | capsules | 200 | 400.00 | |
| Vita Loa Iran Farmula High Potonov | | | | |
| | 2 tablets | 450 | 200.00 | |
| Waltivitariiii & Willerai | | 700 | 200.00 | |
| OsteoMatrix | capsules | 1000 | 400.00 | |
| Vita-Lea Gold Vitamin K Formula high | | | | |
| Potency Multivitamin & Mineral | 2 tablets | 450 | 400.00 | |
| | 4 | T | | |
| Chewable Cal Mag Plus | chewtabs | 1000 | 200.00 | |
| Cinch 3-in-1 Inch Loss Plan Boost | 3 tablets | 300 | 260.00 | |
| + | | | | RX |
| OptiNate | 1 tablet | 200 | 400.00 | only |
| + · r ··· · | | | | |
| | | 1 | I | |
| | Whole Source Mature Adult Multivitamin/Mineral Calcium Soft Chews 600mg Calcium Plus Vitamin D Central Vite VitaPhil Advance Formula Cerovite Cerovite Jr. Chewables VITa-PMS Calcium 600-D Oysco 500 + D Oysco D Prenavite Childrens chewables Guided Minerals Multi Minerals Complex Hair, Skin and Nails with MSM Prime Years Multi Vitamin Prostrate Health Single Day Antioxidant Rich Super Calcium 1200 with Vitamin D Sustained Release Single Day Multi Vitamin Vegetarian Multiple with Beta Carotene Vita-Lea Iron Formula High Potency Multivitamin & Mineral OsteoMatrix Vita-Lea Gold Vitamin K Formula high Potency Multivitamin & Mineral | Daily Multi 50+ Osteo Bi-Flex Plus Calcium With Vitamins C and D Whole Source Mature Adult Multivitamin/Mineral Calcium Soft Chews 600mg Calcium Plus Vitamin D Central Vite 1 tablet VitaPhil 1 tablet Advance Formula Cerovite Cerovite Jr. Chewables VITa-PMS 1 tablet Calcium 600-D 1 tablet Oysco 500 + D Oysco D 1 tablet Childrens chewables Guided Minerals Multi Minerals Complex Hair, Skin and Nails with MSM Prime Years Multi Vitamin Vegetarian Multiple with Beta Carotene Vita-Lea Iron Formula High Potency Multivitamin & Mineral Vita-Lea Gold Vitamin K Formula high Potency Multivitamin & Mineral Chewable Cal Mag Plus Cinch 3-in-1 Inch Loss Plan Boost 1 tablets 1 tablets 2 tablets 4 chewables 4 chewtabs Chewable Cal Mag Plus Cinch 3-in-1 Inch Loss Plan Boost 3 tablets 4 chewtabs | Daily Multi 50+ | Daily Multi 50+ |

| | | capsules | | 1 | 1 |
|---|---|---|---|---|---|
| | | 3 | | | |
| | Mens Golden Multi-Vita-Min | capsules | 75 | 400.00 | |
| | | 4 | | | |
| | Multi-Vita Mega-Mineral Multi-Vita-Min | capsules | 420 | 400.00 | |
| | Once Daily High Energy Multi-Vita-Min | 1 capsule | 10 | 400.00 | |
| | Once Daily Softgel with Lutein Multi- | _ | | | |
| | Vita-Min | 1 softgel | 25 | 400.00 | |
| | Provide Multi-Vita-Min | 2 softgels | 200 | 400.00 | |
| | | 4 | | | |
| | Spectro 50 Plus Multi-Vita-Min | capsules | 200 | 800.00 | |
| | | 4 | 0.50 | 222.22 | |
| | Spectro Energy Multi-Vita-Min | capsules | 250 | 800.00 | |
| | Spectro Kid Multi-Vitamin | 2 tablets | 200 | 400.00 | |
| | | 4 | | | |
| | Spectro Man Multi-Vita-Min | capsules | 200 | 400.00 | |
| | | 4 | | | |
| | Spectro Woman Multi-Vita-Min | capsules | 400 | 800.00 | |
| | T . B . M | 2 | | 400.00 | |
| | Twice Daily Multi-Vita-Min | capsules | 200 | 400.00 | |
| | Manatarian Operator NA III NOS NA | 6 | 500 | 400.00 | |
| | Vegetarian Spectro Multi-Vita-Min | capsules | 500 | 400.00 | |
| | | 4 | 400 | | |
| | VitaPrime for Men Multi-Vita_min | capsules | 400 | 400.00 | |
| | VitaPrime for Women Multivitamin and | 4 | | | |
| | Multimneral | capsules | 400 | 400.00 | |
| | | 3 | | | |
| | Womens Golden Multi-Vita-min | capsules | 75 | 400.00 | |
| | YumAid Multi-Vita-Min Punch | 1tsp | 50 | 400.00 | |
| _ | | 2 | | | |
| Solgar | Adv Proanthocyanidin Complex | capsules | 170 | 800.00 | |
| | Calcium Magnesium with Vitamin D | 5 tablets | 1000 | 400.00 | |
| | Earth Source Multi-Nutrient | 3 tablets | 250 | 400.00 | |
| | Female Multiple | 3 tablets | 400 | 400.00 | |
| | Formula V VM-75 Multivitamin with | 2 | | | |
| | Chelated Minerals | capsules | 20 | 400.00 | |
| | Formula VM-2000 | 2 tablets | 50 | 400.00 | |
| | Formula VM-Prime for Adults 50 Plus | | | | |
| | Iron Free | 1 tablet | 20 | 400.00 | |
| | Iron Free Formula VM-75 | 1 tablet | 20 | 400.00 | |
| | Kangavites Complete Childrens | | | | |
| | Formula | 2 tablets | 128 | 200.00 | |
| | Male Multiple | 3 tablets | 400 | 400.00 | |
| | Omnium Multiple Vintamin and Mineral | 2 | | | |
| | Formula Iron Free | tabletws | 25 | 200.00 | |
| | Prenatal Nutrients | 4 tablets | 1300 | 400.00 | |
| | 1 Total Hamonia | TIGNICIS | 1000 | 700.00 | |
| Contro | Advanced One Multiple (with and | 1 | | | |
| Source | Advanced One Multiple (witn and | 1 tablet | 50 | 400.00 | |
| Naturals | without Iron) | 1 tablet | 50 | 400.00 | |
| | Advanced Triple Boron with Calcium | 2 | F00 | 400.00 | |
| | 1000mg | capsules | 500 | 400.00 | |
| | Calcium & Magnesium 300mg | 1 tablet | 200 | 500.00 | |

| | Calcium Hydroxyapatite | 2 tablets | 600 | 500.00 | Ī |
|---|---|---|---|---|---|
| | Calcium Night 150mg | 2 tablets | 300 | 100.00 | |
| | Calcium 200mg | 1 tablet | 200 | 500.00 | |
| | Elan Vital Multiple | 6 tablets | 200 | 400.00 | |
| | Life Defense | 4 tablets | 95 | 200.00 | |
| | Ello Belefice | 4 | 33 | 200.00 | |
| | Life Force | capsules | 100 | 1000.00 | |
| | Mega Kid | 1 wafer | 20 | 200.00 | |
| | Mens Life Force | 3 tablets | 100 | 400.00 | |
| | Mothers Choice | 4 tablets | 615 | 400.00 | |
| | Spirulina | 2 tablets | 106 | 400.00 | |
| | Ultra | 6 tablets | 125 | 400.00 | |
| | Womens Life Force | 3 tablets | 200 | 400.00 | |
| Sundown | Advanced SunVite | 1 tablet | 162 | 400.00 | |
| | Calcium 600 + D | 1 capsule | 600 | 200.00 | |
| | Calcium Oyster Shell 1000mg | 3 tablets | 1000 | 400.00 | |
| | Complete Daily with Lutein | 1 caplet | 162 | 400.00 | |
| | Daily Multi & Min | 1 caplet | 162 | 400.00 | |
| | Daily Multiple 50+ Iron Free with | | | | |
| | Lutein & Lycopene | 1 caplet | 200 | 400.00 | |
| | Multiple Complete Womens | 1 caplet | 250 | 400.00 | |
| | Naturals Prenatal Formula | 1 tablet | 200 | 400.00 | |
| | One Daily Multiple for Women | 1 caplet | 400 | 400.00 | |
| | Prenatal Vitamin and Mineral Formula | 1 tablet | 200 | 400.00 | |
| | Vitamins to Go Womens | 1 packet | 660 | 125.00 | |
| Super | | | | | |
| Nutrition | Calcium Blend | 3 tablets | 1000 | 1000.00 | |
| | Longevity | 1 tablet | 68 | 400.00 | |
| | Menopause Multiple Blend | 8 tablets | 750 | 500.00 | |
| | Mens Blend | 3 tablets | 300 | 500.00 | |
| | Simply One Prenatal | 1 tablet | 210 | 500.00 | |
| | Simply One - One Per Day | 1 tablet | 33 | 400.00 | |
| | Simply Perfect Kids | 4 tablets | 120 | 400.00 | |
| | Super Blend | 4 tablets | 500 | 500.00 | |
| The DV | Daine a Coura Coffee I | 4 | 400 | 400.00 | RX |
| Ther-RX | PrimaCare Softgel | 1 softgel | 400 | 400.00 | only |
| | PrimaCare Advantage | 1 softgel | 250 | 230.00 | RX<br>only |
| | | 1 | | | RX |
| | PrimaCare ONE | capsules | 150 | 170.00 | only |
| Thompson | Adult Plex | 3 tablets | 300 | 400.00 | |
| mompson | All in One Multivitamin Iron Free | 1 capsule | 100 | 400.00 | |
| | Coachs Formula with Enzymes | 2 tablets | 333 | 133.00 | |
| | Mega 80 | 1 tablet | 45 | 600.00 | |
| | wega oo | 2 | 40 | 000.00 | |
| | Multi Formula for Women | capsules | 300 | 200.00 | |
| | Multi Vitamins with Minerals | 2 tablets | 170 | 200.00 | |
| | Nuplex with Iron | 1 tablet | 120 | 400.00 | |

| | Prenatal Formula | 2 tablets | 68 | 610.00 | |
|---|---|---|---|---|---|
| | Teenplex Multivitamin | 2 tablets | 200 | 400.00 | |
| | ' | | | | |
| TwinLab | Daily One Caps (with or without Iron) | 1 capsule | 25 | 400.00 | |
| | Dr. Greene Childrens (various flavors) | 1 tablet | 100 | 400.00 | |
| | Dr. Greene Healthy Bone Formula | 1 tablet | 500 | 200.00 | |
| | , | 2 | | | |
| | Dr. Greene Pre-Natal formula | capsules | 500 | 400.00 | |
| | Dualtabs Mega Vitamin and Mineral | | | | |
| | formula | 2 tablets | 500 | 200.00 | |
| | | 2 | | | |
| | Allergy Multi Caps | capsules | 333 | 133.00 | |
| | Animal Friends Kids Chewable | 1 | | | |
| | (various flavors) | chewable | 100 | 400.00 | |
| | Bone Support with Ostivone | 4 tablets | 1500 | 800.00 | |
| | Cal Quick Liquid | 5ml | 500 | 100.00 | |
| | Calcium 500 with Magnesium & | | | | |
| | Vitamin D | 1 tablet | 500 | 200.00 | |
| | Calcium Citrate Chewable | 4 wafers | 1000 | 400.00 | |
| | | 2 | | | |
| | Pre-Natal Care | capsules | 400 | 400.00 | |
| | | 4 | | | |
| | Womens Ultra Daily | capsules | 510 | 400.00 | |
| Usana | Active Calcium | 4 tablets | 800 | 400.00 | |
| | | 4 | | | |
| | Body Rox Active Calcium Chewable | chewtabs | 800 | 400.00 | |
| | Essentials Usanimals | 1 tablet | 75 | 100.00 | |
| | HealthPak | 1 packet | 335 | 1000.00 | |
| VegLife | MultiVeg Energy | 4 tablets | 34 | 400.00 | |
| | | 3 | | | |
| | MultiVeg Energy with Lutein and Iron | capsules | 50 | 800.00 | |
| | SpectroVeg High Energy | 6 tablets | 500 | 400.00 | |
| | Vegan Cal-Mag Citrate Plus Vitamin D | 3 tablets | 500 | 200.00 | |
| | Vegan Kids | 2 tablets | 30 | 400.00 | |
| | Vegan One Multi with Iron | 1 tablet | 50 | 400.00 | |
| | | 2 | | | |
| | Vital Teen Boys | capsules | 150 | 800.00 | |
| | | 2 | | | |
| | Vital Teen Girls | capsules | 150 | 1000.00 | |
| Vitabase | Active Mans Formula | 1 tablet | 50 | 400.00 | |
| | Childrens Multiple Liquid | 30ml | 200 | 220.00 | |
| | Coral Calcium 1000mg | 1 capsule | 250 | 200.00 | |
| | | 3 | | | |
| | Hair, Skin & Nails Liquid | liquicaps | 300 | 200.00 | 1 |
| | | 2 | | | |
| | Kids Chewable Calcium | chewtabs | 200 | 200.00 | 1 |
| | PreNatal Plus | 4 tablets | 800 | 400.00 | |
| | Super Calcium & Magnesium | 3 tablets | 1000 | 200.00 | |
| | Super Softgel Formula | 2 softgels | 200 | 400.00 | |

| Vitaline | Total Formula | 1 tablet | 100 | 400.00 | |
|---|---|---|---|---|---|
| | Total Formula 2 | 1 tablet | 100 | 400.00 | |
| | Maximum Red | 1 tablet | 83 | 67.00 | |
| Vitamin | | | | | |
| Shoppe | 1 Daily | 1 tablet | 100 | 400.00 | |
| Спорро | Ultimate Man | 2 tablets | 200 | 1000.00 | |
| | Ultimate Woman | 2 tablets | 500 | 1000.00 | |
| | Calcium Citrate | 2 tablets | 333 | 204.00 | |
| Vitamin | | | | | |
| World | Bone Reinforcer with Hydroxyapatite | 4 tablets | 1200 | 400.00 | |
| | Calcium Magnesiun with D | 3 tablets | 1000 | 400.00 | |
| | Canal Calaires 500 as Blue Vitarain D | 2 | 270 | 400.00 | |
| | Coral Calcium 500mg Plus Vitamin D | capsules | 370 | 400.00 | |
| | Daily 3 Multiple with Chloesterol Regulators | 3 | 106 | 800.00 | |
| | Green Source | capsules<br>3 tablets | 250 | 400.00 | |
| | Spirulina Soy protein Drink | 1 scoop | 300 | 400.00 | |
| | Thervim M | 1 tablet | 40 | 400.00 | |
| | Ultra Vita Man timed release | 2 tablets | 200 | 200.00 | |
| | Cal Mag Calaium & Magnasium | | | | |
| Whole Health | Cal-Mag Calcium & Magnesium Citrates 1400mg | 4 tablets | 1000 | 400.00 | |
| Wilole Health | Citiates 1400mg | 2 | 1000 | 400.00 | |
| | Childrens Chewable Multivitamin | chewtabs | 55 | 400.00 | |
| | Children's Chewasie Malaytaniin | 2 | | 100.00 | |
| | GreenHealth Natural Multi | capsules | 50 | 100.00 | |
| | | 4 | | | |
| | HerHealth | capsules | 780 | 600.00 | |
| | | 3 | | | |
| | HisHealth | capsules | 272 | 400.00 | |
| | Prenatal Health | 4 tablets | 1000 | 220.00 | |
| | Super Multi Plus | 3 tablets | 400 | 400.00 | |
| 140 | | | | | |
| Whole | Matura Adulta Multi Minaral with Llarba | 1 toblet | 165 | 400.00 | |
| Source | Mature Adults Multi Mineral with Herbs | 1 tablet | 165 | 400.00 | |
| | Ezcal 2000 + D (regular tablets & | | | | |
| Windmill | chewables) | 1 tablet | 1000 | 400.00 | |
| William | CiteWables) | i tablet | 1000 | 400.00 | |
| Women's | | | | | |
| Health | | | | | |
| America | ProCycle Gold | 1 tablet | | 100.00 | |
| | Mulitvitamin/Multimineral with Beta | | | | |
| Wonder Labs | Carotene & Lycopene | 1 tablet | 162 | 400.00 | |
| | | 3 | | | |
| | Pure coral Calcium 2500mg | capsules | 2500 | 200.00 | |
| | 2 (20) | | | 455.55 | |
| Xanodyne | Duet DHA | 1 tablet | 200 | 400.00 | RX |

| | | | | only | / |
|---------------|----------|-----|--------|------|---|
| | | | | RX | |
| Duet Chewable | 1 tablet | 100 | 400.00 | only | / |

Questionnaire adapted from Rapid Vit D data from USDA database from NDS

INSTRUCTIONS

Use the excel spreadsheet to calculate the average daily dietary intake of calcium and vitamin D from food.

Please ask the participant to recall food items eaten over the last 3 days.

Ask the participant about each food item in column "B" and record how many servings (size of each serving detailed in spreadsheet) he/she ate over the last 3 days bent the participant about each food item in column "B" and record how many servings (size of each serving detailed in spreadsheet) he/she ate over the last 3 days. Enter the number of servings in column "C". The total amount of calcium and vitamin D from that food item will be automatically calculated in the spreadsheet and di The total DAILY intake of calcium and vitamin D (an average of the 3 day intake) will be automatically calculated and displayed in row 65; these are the numbers to I Upload the spreadsheet using the File Exchange Utility located on the FSTRF website (www.fstrf.org)

| Food | servings | Calcium/serving (IVitD/serving (mcg) CA Total (mg) D Total (IU) | (mcg) CA To | tal (mg) D Total | (D) |
|---|---|---|---|---|---|
| Milk/yogurt/cheese | | | | | |
| cheese (1 oz or 6 tbsp) | | 200 | 60.0 | 0 | 0 |
| cottage cheese (1/2cup) | | 20 | 0.03 | 0 | 0 |
| custard, pudding, cream pie (1/2 cup) | | 150 | 1.43 | 0 | 0 |
| ice cream, frozen yogurt, milkshake (1 cup) | | 200 | 1.26 | 0 | 0 |
| yogurt (1 cup) | | 388 | 0.03 | 0 | 0 |
| butter (1 tbsp) | | 100 | 0.20 | 0 | 0 |
| milk (1 cup) | | 300 | 2.50 | 0 | 0 |
| latte or mocha latte (1 cup) | | 220 | 2.00 | 0 | 0 |
| café au lait (1 cup) | | 66 | 2.00 | 0 | 0 |
| cappucchino (1 cup) | | 250 | 2.00 | 0 | 0 |
| Fortified orange juice (1 cup) | | 350 | 2.50 | 0 | 0 |
| soy milk, unfortified (1 cup) | | 10 | 0.00 | 0 | 0 |
| soy milk, fortified (1 cup) | | 300 | 2.50 | 0 | 0 |
| cream soup/sauce (1 cup) | | 200 | 0.18 | 0 | 0 |
| macaroni and cheese (1 cup) | | 250 | 0.23 | 0 | 0 |
| pizza (1 slice) | | 250 | 0.03 | 0 | 0 |
| quiche (1 slice) | | 250 | 1.01 | 0 | 0 |
| Fruits/Vegetable | | | | 0 | 0 |
| broccoli or cooked greens (1/2 cup) | | 100 | 0.00 | 0 | 0 |
| other vegetables (1/2 cup) | | 30 | 00.0 | 0 | 0 |
| fruit (1/2 cup or 1 small) | | 30 | 00.0 | 0 | 0 |
| Bread/Cereal/Rice/Pasta | | | | 0 | 0 |
| bread (1 slice) | | 20 | 00.0 | 0 | 0 |
| calcium enriched bread (1 slice) | | 102 | 0.00 | 0 | 0 |
| cereal (1 oz) | | 20 | 0.94 | 0 | 0 |

| smoked eel (1oz) | | 0.89 | 0 | _ |
|--------------------------------------|---|-------|---|---|
| herring (1oz) | _ | 1.54 | 0 | _ |
| canned salmon with bones (3oz) 150 | | 9.91 | 0 | _ |
| canned sardines with bones (3oz) 400 | | 3.91 | 0 | _ |
| shrimp (3oz) 100 | | 3.04 | 0 | _ |
| oysters (7-9) 100 | | 9.36 | 0 | _ |
| tofu (2.5x2.5x1 inch) 100 | | 00:00 | 0 | _ |
| peanuts (1/2 cup) 30 | | 00:0 | 0 | _ |
| 699 (1) | | 0.56 | 0 | _ |
| Fat/Sugar/Alcohol | | | 0 | _ |
| cake (1 slice) 40 | | 0.12 | 0 | _ |
| beer (12 oz) 10 | | 00.0 | 0 | _ |
| cola (12 oz) 10 | | 00.00 | 0 | _ |
| chocolate (1 oz) 50 | | 0.00 | 0 | _ |